## Statistical Analysis Plan

# Plexxikon Inc. PLX121-01

A Phase 1b and 2a Study to Assess Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PLX9486 as a Single Agent and in Combination with PLX3397 or Sunitinib (Sutent®) in Patients with Advanced Solid Tumors and Patients with Locally Advanced, Unresectable, or Metastatic Gastrointestinal Stromal Tumor (GIST) Who Have Been Previously Treated with Imatinib Mesylate/KIT-Directed Tyrosine Kinase Inhibitor (TKI) Therapy

Protocol Version: 23 July 2019 / Amendment 7

**Sponsor:** Plexxikon Inc.

91 Bolivar Dr.

Berkeley, CA 94710, USA

Prepared by:

**Synteract** 

430 Davis Drive, Suite 500 Morrisville, NC 27560, USA

Version 1.0 July 19, 2018

**Version 2.0 October 4, 2018** 

**Version 3.0 October 11, 2018** 

Version 4.0 December 4, 2018

Version 5.0 June 19, 2019

Version 6.0 August 30, 2019

Version 7.0 September 13, 2019

Version 8.0 December 3, 2019

Version 9.0 July 1, 2020

Date

Date

Plexxikon Inc.
PLX121-01

Authors

Electronically signed by:
Fleason: I am the author of this document
Date: Jul 1, 2020 11:06 CDT

Statistical Analysis Plan
01Jul2020

Synteract

430 Davis Drive, Suite 500, Morrisville, NC 27560, USA



Plexxikon Inc.

91 Bolivar Dr.Berkeley, CA 94710, USA

## TABLE OF CONTENTS

| LIS | T OF | ABBREVIATIONS | 5 |
|---|---|---|---|
| DE | FINIT | TIONS | 6 |
| 1. | INTI | RODUCTION | 7 |
| 2. | STU | DY OBJECTIVES | 7 |
| | 2.1 | PART 1 (DOSE-EVALUATION COHORT) OBJECTIVES | |
| | | PRIMARY OBJECTIVES | |
| | | SECONDARY OBJECTIVES | |
| | | EXPLORATORY OBJECTIVES | |
| | 2.2 | PART 2 (EXTENSION COHORTS: PARTS 2B AND 2E) OBJECTIVES | 8 |
| | | PRIMARY OBJECTIVES | |
| | | SECONDARY OBJECTIVES | |
| | | EXPLORATORY OBJECTIVES | |
| <b>3.</b> | STU | DY DESIGN AND PLAN | 8 |
| | 3.1 | DOSE LIMITING TOXICITIES | 10 |
| | 3.2 | SCHEDULE OF EVENTS | 12 |
| 4. | DET | ERMINATION OF SAMPLE SIZE | 12 |
| 5. | GEN | IERAL ANALYSIS CONSIDERATIONS | 12 |
| | 5.1 | Data Summaries | |
| | 5.2 | DATA HANDLING | |
| | 0.2 | 5.2.1 Baseline Values | |
| | | 5.2.2 Conventions | |
| 6. | ANA | LYSIS POPULATIONS | 14 |
| 7. | | DY POPULATION | |
| ′• | 7.1 | PATIENT DISPOSITION | |
| | 7.1 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 14 |
| | 7.3 | MEDICAL HISTORY | |
| | 7.4 | CONCOMITANT MEDICATIONS (AND PROCEDURES) | |
| 8. | | ICACY ANALYSES | |
| ٠. | 8.1 | TUMOR RESPONSE | |
| | 0.1 | 8.1.1 Overall Timepoint Response | |
| | | 8.1.2 Best Response | |
| | | 8.1.3 Best Overall Response | |
| | 8.2 | EFFICACY VARIABLES | |
| | 8.3 | ADJUSTMENTS FOR COVARIATES | |
| | 8.4 | HANDLING OF DROPOUTS OR MISSING DATA | 21 |
| | 8.5 | INTERIM ANALYSIS AND DATA MONITORING | |
| | 8.6 | EXAMINATION OF SUBGROUPS | |
| | 8.7 | MULTIPLE COMPARISON/MULTIPLICITY | |
| | 8.8<br>8.9 | MULTICENTER STUDIES | |
| 9. | | RMACOKINETIC ANALYSES | |
| | | RMACODYNAMIC ANALYSES | |
| 11. | SAF | ETY ANALYSES | 22 |
| | 11.1 | EXTENT OF EXPOSURE | 22 |
| | 11.2 | ADVERSE EVENTS | 22 |

| Plexxikon Inc.<br>PLX121-01 | | Statistical Analysis Plar<br>29Jun2020 |
|---|---|---|
| 11.3 | CLINICAL LABORATORY EVALUATION | 24 |
| 11.4 | VITAL SIGNS | |
| | PHYSICAL EXAMINATION | |
| 11.6 | ELECTROCARDIOGRAM | 25 |
| 11.7 | EASTERN COOPERATIVE ONCOLOGY GROUP (ECOG) | 26 |
| 12. CHA | NGES TO PROTOCOL-SPECIFIED ANALYSES | 20 |

#### LIST OF ABBREVIATIONS

AE Adverse event BID Twice daily

ATC Anatomical Therapeutic Chemical

BMI Body Mass Index
CI Confidence interval
CR Complete response
CRF Case report form
CSR Clinical study report

CTCAE Common Terminology Criteria for Adverse Events

CxDy Cycle x Day y

DLT Dose limiting toxicity
DOR Duration of response
ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

GIST Gastrointestinal stromal tumor

MedDRA Medical Dictionary for Regulatory Activities

MTD Maximum tolerated dose

NE Not evaluable

ORR Overall Response Rate
PD Progressive disease

PFS Progression-free survival

PK Pharmacokinetic
PR Partial Response
QD Once a day

QTcF Heart-rate-corrected QT interval (Fridericia's formula)

RECIST Response Evaluation Criteria In Solid Tumors

RP2D Recommended phase 2 dose

SAE Serious adverse event

SD Stable disease

TEAE Treatment-emergent adverse event

TKI Tyrosine Kinase Inhibitor WHO World Health Organization

#### **DEFINITIONS**

Adverse Event (AE) An adverse event (AE) is any untoward medical

> occurrence in a patient administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (e.g., including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not it is considered to be study drug related. This includes any newly occurring event or previous condition that has increased in severity or frequency

since the administration of study drug.

Dose Limiting Toxicities (DLTs) are defined as AEs Dose Limiting occurring during the first 28 days of study drug Toxicity (DLT)

administration that are classified as possibly or probably related to the study drug, and meet one of the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria listed in Section 3.1 of the SAP.

Safety Population The Safety Population will include all patients treated

with at least one dose of study drug.

Efficacy Evaluable The Efficacy Evaluable Population will include all

> patients who have taken at least 1 dose of study drug and have had at least 1 post-baseline tumor assessment or discontinue study medication due to disease progression

or death.

Pharmacokinetic (PK) All patients who have adequate pharmacokinetic (PK)

**Population** data.

Serious AE (SAE) A serious AE (SAE) is an AE occurring at any dose that:

results in death; is a life-threatening experience; requires inpatient hospitalization longer than 24 hours or

prolongation of an existing hospitalization; results in a persistent or significant disability/incapacity; is a congenital anomaly or birth defect, or is an important

medical event.

Treatment-emergent AE

**Population** 

A treatment-emergent AE (TEAE) is an AE that started (TEAE) or worsened in severity on or after the date of the initial

dose of study drug.

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of Plexxikon Protocol Number PLX121-01 "A Phase 1b and 2a Study to Assess Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PLX9486 as a Single Agent and in Combination with PLX3397 or Sunitinib (Sutent®) in Patients with Advanced Solid Tumors and Patients with Locally Advanced, Unresectable, or Metastatic Gastrointestinal Stromal Tumor (GIST) Who Have Been Previously Treated with Imatinib Mesylate/KIT-Directed Tyrosine Kinase Inhibitor (TKI) Therapy" Amendment 7 dated 23 July, 2019.

This study is designed in 7 parts. Part 1 will establish the maximum tolerated dose/recommended Phase 2 dose of PLX9486 in patients with advanced solid tumors (including GIST) as well as evaluate the efficacy of PLX9486 in solid tumors. Parts 2 will assess safety, tolerability, and efficacy of PLX9486 as a single agent or in combination with PLX3397 or sunitinib in patients advanced solid tumors (including GIST) or patients with advanced solid tumors/advanced solid tumor with KIT mutations.

The purpose of this analysis plan is to provide specific guidelines from which the analysis of Part 1, Part 2b and Part 2e will proceed. Any deviations from these guidelines will be documented in the clinical study report (CSR).

Details of the pharmacokinetic (PK) statistical analysis plan will be outlined in a separate document and a formal PK report will be written for inclusion in the final study report.

### 2. STUDY OBJECTIVES

## 2.1 Part 1 (Dose-Evaluation Cohort) Objectives

## 2.1.1 Primary Objectives

The primary objectives of Part 1 of this study are:

- To evaluate safety and pharmacokinetics (PK) of orally administered PLX9486 as single and as multiple doses
- To establish the maximum tolerated dose/recommended Phase 2 dose (MTD/RP2D) in patients with advanced solid tumors (including GIST).

## 2.1.2 Secondary Objectives

The secondary objective of Part 1 of this study is to evaluate the efficacy of PLX9486 in solid tumors as measured by Overall Response Rate (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, Duration of Response (DOR), and Progression-Free Survival (PFS).

## 2.1.3 Exploratory Objectives

The exploratory objective of Part 1 of this study is to assess biomarkers in peripheral blood, archival tumor tissue, and available tumor biopsies.

## 2.2 Part 2 (Extension Cohorts: Parts 2b and 2e) Objectives

## 2.2.1 Primary Objectives

The primary objectives of Part 2b and Part 2e of this study are:

- Part 2b: To assess the safety and tolerability of the combination of PLX9486 and PLX3397 and to establish an RP2D of PLX9486 in combination with PLX3397 in patients with advanced solid tumors (including GIST).
- Part 2e: To assess the safety and tolerability of the combination of PLX9486 and sunitinib and to establish an RP2D of PLX9486 in combination with sunitinib in patients with advanced solid tumors (including GIST)

## 2.2.2 Secondary Objectives

The secondary objectives of Part 2b and Part 2e are:

- To determine the pharmacokinetics (PK) of PLX9486 as a single agent and in combination with PLX3397 (Part 2b) or sunitinib (Part 2e).
- To estimate the following: ORR (using RECIST 1.1), clinical benefit rate (CBR), Overall Survival (OS) and 12-month OS rate, PFS and 6-month PFS rate, and DOR.

## 2.2.3 Exploratory Objectives

The exploratory objective of Part 2 of this study is to assess biomarkers in peripheral blood and in archival tumor tissue.

### 3. STUDY DESIGN AND PLAN

This Phase 1b and 2a, open-label, multicenter study includes a dose-evaluation portion (Part 1) in which the safety profile and RP2D of PLX9486 as a single oral agent, administered daily in 28-day dosing cycles will be evaluated in patients with solid tumors (including GIST), followed by signal-seeking expansion cohorts (Part 2, consisting of Part 2b, 2e and as described in the protocol). This document covers the analysis plan for Part 1 Dose Escalation of PLX9486, Part 2b and Part 2e only that were planned in the protocol as follows:

Part 1 (dose escalation) will enroll approximately 30 solid tumor patients in a standard "3+3" design. Additional patients may be required depending on the number of cohorts and evaluable patients needed.

Part 2b will be the open-label, sequential cohort dose-finding study of PLX9486 combined with PLX3397 in up to approximately 30 patients with solid tumors (including GIST) in a 3+3 design.

Part 2e will be the open-label, sequential cohort dose-finding study of PLX9486 combined with sunitinib in up to approximately 30 patients with solid tumors (including GIST) in a 3+3 design.

Figure 1 provides an overview of the study design.

Figure 1: Overview of Study PLX121-01



In the absence of Grade ≥2 toxicity that is considered "possibly" or "probably" related to the study agent or dose-limiting toxicity (DLT) and in conjunction with review of the pharmacokinetic data, dose escalation in each study part (Part 1, 2b and 2e) is planned to occur as shown in the table below.

PLX9486 Administration in Part 1: Initial and Potential Dose- escalation Cohorts

| Cohort Number | PLX9486 Dose Level (mg/day) <sup>a</sup> | Number and Unit Strength |
|---|---|---|
| 4 | 1000 | 20 x 50 mg |
| 5 | 500 (BID) | 10 x 50 mg (BID) |
| 6 | 1500 | 30 x 50 mg |
| 7 | 2000 | 40 x 50 mg |

<sup>&</sup>lt;sup>a</sup>Dosing interval/frequency will be QD unless otherwise specified (e.g., BID dosing).

## PLX9486 and PLX3397 Administration in Part 2b: Initial and Potential Dose-escalation Cohorts

| Cohort<br>Number | PLX9486 Dose Level (mg/day) <sup>a</sup> | PLX3397 Dose Level (mg/day) |
|---|---|---|
| 1 | Approximately 50% of Part 1 RP2D | 600<br>(200 mg in AM and 400 mg in PM) |

| 2 | Approximately 100% of Part 1 RP2D | 600<br>(200 mg in AM and 400 mg in PM) |
|---|---|---|
| 3 | 100% of Part 1 RP2D | 400 mg QD (Cycles 1 and 2) |
| 3 | | 600 mg QD (Cycle 3 +) <sup>b</sup> |
| 4 + | TBD° | TBDc |

RP2D = recommended phase 2 dose; TBD = to be determined

- <sup>a</sup> PLX9486 administered once-daily (QD) or for higher total daily doses, as split doses (e.g., twice-daily [BID]).
- At the discretion of the investigator and in the absence of clinically significant drug-related toxicity (Section 9.3 in the protocol) during Cycles 1 and 2.
- Based on a review of the data by the Study Committee.

## PLX9486 and Sunitinib Administration in Part 2e: Initial and Potential Dose-escalation Cohorts

| Cohort Number | PLX9486 Dose Level (mg/day) <sup>a</sup> | Sunitinib Dose Level (mg/day) |
|---|---|---|
| 1 | Approximately 50% of Part 1 RP2D | 25 |
| 2 | 100% of Part 1 RP2D | 25 |
| 3 | 100% of Part 1 RP2D | 37.5 |

RP2D = recommended phase 2 dose

Patients who are considered in dose-escalation decisions are not allowed dose reductions during the DLT assessment window. Patients who withdraw from the study prior to completing Cycle 1 for any reason other than a DLT will be replaced. A patient who experiences a DLT may remain in the trial and continue receiving study drug at a lower dose per the investigator's decision in consultation with the Medical Monitor. Further dose escalation and de-escalation rules can be found in the protocol Section 9.2.

The screening period for the study will be 21 days with the exception of tumor burden assessment [i.e., CT scan], which may be performed within 28 days of dosing. The treatment period will occur in 28-day ( $\pm$  7 days) cycles until patient discontinuation or withdrawal or study termination. Patients will be monitored throughout the study for adverse reactions to the drug formulation and/or study procedures. Safety and tolerability assessments will include physical examinations, vital signs, 12-lead electrocardiograms (ECGs), ECOG score, adverse events (AEs), hematology, complete chemistry panel, coagulation, and urinalysis.

An end of study visit must occur ≥30 days after the last dose of PLX9486 and prior to starting any new anti-cancer therapy. A post-study follow-up contact by phone by site staff will be conducted every 3 months during Year 1, then every 6 months thereafter to obtain information on any new anti-cancer therapy received, response, and survival status.

For more information on scheduled assessments and procedures, see Trial Flow Charts (Table 1, Table 3, and Table 6 in the protocol).

## 3.1 Dose Limiting Toxicities

For Part 1, 2b and 2e, in the absence of a DLT, patients must complete the first cycle of treatment (28 days) in order to be considered evaluable for DLT. Patients who discontinue for

Dosing interval/frequency will be QD unless otherwise specified (e.g., BID dosing).

any reason other than a DLT or Grade ≥2 toxicity and have received less than 21 of 28 days of dosing will not be considered evaluable for DLT and will be replaced; however, their data will be reviewed by the study committee and a decision will be made based on their review.

Dose Limiting Toxicities (DLTs) are defined as AEs occurring during the first 28 days of study drug administration (Cycle 1) that are classified as possibly or probably related to the study drug, and meet one of the following Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria.

## Hematologic Toxicities

- Grade 4 neutropenia lasting >7 days
- Grade  $\geq$  3 neutropenia with fever
- Grade 4 thrombocytopenia
- Grade ≥ 3 thrombocytopenia lasting more than 7 days or associated with clinically significant bleeding
- Grade 4 anemia

## Other Toxicities

Any  $\geq$  Grade 3 (AE or laboratory) toxicity despite adequate supportive care <u>except for the following</u>.

- Grade ≥ 3 nausea, vomiting, or diarrhea that resolves to Grade ≤ 2 within 72 hours, with or without medical intervention or prophylaxis because this would not be considered treatment-limiting in an oncology population
- Grade 3 fatigue that resolves to ≤ Grade 2 within 14 days because this would not be considered treatment-limiting in an oncology population
- Grade ≥ 3 asymptomatic changes in alkaline phosphatase, hypomagnesemia, hyperglycemia, or hypophosphatemia that are felt by the investigator to be clinically insignificant
- Grade 3 asymptomatic increases in transaminases (AST, ALT) confirmed upon repeat testing which resolves to ≤Grade 2 within <5 days

Any other Grade  $\geq 3$  toxicity (except those noted above) for which either the Principal Investigator or Sponsor deems further dose escalation inappropriate

Dose escalation will continue unless there are dose-limiting toxicities in ≥2 of at least 6 patients (i.e., 33%) in one cohort within the first 28 days. In the absence of a DLT, patients must complete the first cycle of treatment (28 days) in order to be considered evaluable for DLT. Patients who discontinue for any reason other than a DLT or Grade ≥2 toxicity and have received less than 21 of 28 days of dosing will not be considered evaluable for DLT and will be replaced. Further dose escalation or de-escalation may be considered depending upon safety and PK findings and discussion between the Sponsor and the investigators. If no DLT is observed, the recommended dose for further evaluation may be established based on toxicity, PK, and convenience of dosing in approximately 3-6 patients treated at that dose.

#### 3.2 Schedule of Events

The Schedules of Events can be found in the corresponding Trial Flow Charts in the protocol (Table 1 for Part 1, Table 3 for Part 2b, and Table 6 for Part 2e).

#### 4. DETERMINATION OF SAMPLE SIZE

The sample sizes of the different parts of the study are based on clinical rather than statistical considerations. The dose escalation cohorts (Part 1 and Parts 2b and 2e) follow a typical 3 + 3 design.

The following table shows the probability of escalating to the next higher dose—after either 3 or 6 patients—given the true DLT incidence rate.

| True Incidence of DLTs | 10% | 20% | 30% | 40% | 50% | 60% | 70% |
|---|---|---|---|---|---|---|---|
| <b>Probability of Escalating Dose</b> | 0.91 | 0.71 | 0.49 | 0.31 | 0.17 | 0.08 | 0.03 |

From the table we see that, when the likelihood of a DLT is low (e.g., if the true DLT incidence rate is 10% or less), the probability of escalating to the next higher dose is high (> 90%), However, when the likelihood of a DLT is high (e.g., if the true DLT incidence rate is 60% or higher), the probability (or risk) of escalating to the next higher dose is low (< 10%).

#### 5. GENERAL ANALYSIS CONSIDERATIONS

#### 5.1 Data Summaries

The statistical analyses will be reported using summary tables, figures, and data listings. The International Conference on Harmonisation numbering convention will be used for all tables, listings, and figures. All statistical testing will be two-sided and will be performed at the 0.05 significance level. All confidence intervals (CIs) will be constructed at the two-sided, 95% confidence level. If there is intra-patient dose escalation, summary for these patients will be presented under their original cohorts.

Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums. Categorical variables will be summarized by counts and by percentages of patients in corresponding categories. Time-to-event variables will be summarized using the Kaplan-Meier method. All summary tables will be presented by study part, dose cohorts, and overall. Baseline summaries will also include a total summary column.

Individual patient data obtained from the case report forms (CRFs), PK data, and pharmacodynamics data, will be presented by cohort, patient, and time point (if applicable) in data listings. Data from all assessments, whether scheduled or unscheduled, will be included in the listing. Listings will present the dates in their original format (without any imputation).

Some patients in Part 1b were given a low dose of PLX9486 at study day -10 for use in the PK analysis. For the purposes of safety analyses this dose will be considered the date of first dose. For the purposes of efficacy analyses the date of first dose will be considered C1D1.

The analyses described in this plan are considered a priori, in that they are defined prior to database lock. Post-hoc analyses will be identified in the CSR.

All analyses and tabulations will be performed using SAS® v9.4 on a SAS server platform. Tables and listings will be presented in rich text format. Upon completion, all SAS programs will be validated by an independent programmer. In addition, all program output will undergo two independent statistical reviews, one of which is a senior level statistical review. The validation process will be used to confirm that statistically valid methods have been implemented and that all data manipulations and calculations are accurate. Checks will be made to ensure accuracy, consistency with this plan, consistency within tables, and consistency between tables and corresponding data listings. Upon completion of validation and quality review procedures, all documentation will be collected and filed by the project statistician or designee.

## 5.2 Data Handling

#### 5.2.1 Baseline Values

Unless otherwise specified, the baseline value is defined as the last non-missing value obtained prior to the first dose of any study drug (PLX9486 for Part 1, PLX9486 or PLX3397 for Part 2b, and PLX9486 or sunitinib for Part 2e). Post-baseline values are defined as values obtained after the first dose of any study drug. Change from baseline is defined as a post-baseline value minus the baseline value.

Baseline weight is defined as the value obtained at Cycle 1 Day 1 (C1D1), if this value is missing the last value obtained before the date and time of the first dose of any study drug will be used.

#### 5.2.2 Conventions

Percentages are routinely based on the total category count excluding missing values if not otherwise mentioned. Percentages showing a rate relative to the total number of patients in this group are given in special tables (e.g., AE tables). Table footnotes will specify the basis for percentages.

The precision of the original measurements will be maintained in summaries and listings, when possible. Generally, means, medians and standard deviations will be presented with an increased level of precision; means and medians will be presented to one more decimal place than the raw data, and the standard deviations will be presented to two more decimal places than the raw data.

Summaries of continuous variables that have some values recorded using approximate values (e.g. < or >) will use imputed values. That is, approximate values will be imputed using the closest exact value for that measurement. Listings will present the data in the original format.

For tables where rounding is required, rounding will be done to the nearest round-off unit. For example, if the round-off unit is the ones place (i.e., integers), values  $\geq XX.5$  will be rounded up to XX+1 while values  $\leq XX.5$  will be rounded down to XX.

Conventions for handling partial dates for AEs and prior and concomitant medications are given in Appendix 1.

Listings will present the dates in their original format (without any imputation). In listings, durations of AEs and concomitant medications will not be derived using imputed dates but, rather, be set to missing when an event has a partially or completely missing start date or end date.

For frequency counts of categorical variables, categories whose counts are zero will be displayed for the sake of completeness. For example, if none of the patients discontinue due to "lost to follow-up," this reason will be included in the table with a count of 0. Categories with zero counts will not have zero percentages displayed.

#### 6. ANALYSIS POPULATIONS

The Efficacy Evaluable population will include all patients who have taken at least one dose of study drug and have had at least one post-baseline tumor assessment or discontinue study medication early due to disease progression or death.

The Safety population will include all patients treated with at least one dose of any study drug.

The PK and PD analysis populations will consist of all patients who have adequate PK and PD data.

#### 7. STUDY POPULATION

## 7.1 Patient Disposition

Patient disposition information will be summarized by study part, dose cohort and overall. Summaries will include the number of enrolled patients, the number of patients in each analysis population, and the primary reason for discontinuation.

## 7.2 Demographic and Baseline Characteristics

Demographic variables include age, gender, ethnicity, and race.

Descriptive statistics will be presented for age. Frequency counts and percentages will be presented for gender, ethnicity, and race. Demographic and baseline characteristics will be summarized by study part and overall. All demographic and baseline characteristics will be presented in a data listing.

## 7.3 Medical History

The number and percentage of patients will be summarized by study part, dose cohort and overall for each body system.

Primary Cancer History and Prior Treatment for Primary Malignancy will be listed.

## 7.4 Concomitant Medications (and Procedures)

Verbatim terms on CRFs will be mapped to Anatomical Therapeutic Chemical (ATC) class and Generic Drug Names using the World Health Organization (WHO) Drug Dictionary Enhanced B2 format, March 1, 2015 release.

Prior medications are those that begin prior to the administration of study drug\_which have a stop date prior to the date of first dose. Concomitant medications are those which are taken at any time between the date of first dose and the date of last dose of any study medication. See Appendix 1 for handling of partial dates for medications. In cases where it is not possible to determine if a medication is concomitant, the medication will be classified as concomitant.

Prior and concomitant medications will be summarized separately, by WHO ATC class and generic drug name for the Safety Population. Summaries will be presented for each study part, dose cohort, and overall. The number and percentage of patients using each medication will be presented. Patients may have more than one medication per ATC class and generic drug name. At each level of patient summarization, a patient is counted once if he/she reported one or more medications at that level. Each summary will be ordered by descending order of incidence of ATC class and generic drug name within each ATC class.

#### 7.5 Protocol Deviations

A listing of protocol deviations will be provided.

## 8. EFFICACY ANALYSES

Several efficacy variables will be derived based on the collected data and will be summarized. All efficacy summaries (or analyses) will be based on Efficacy Evaluable population. This study will utilize the definition of tumor response as described in RECIST 1.1.

## 8.1 Tumor Response

## 8.1.1 Overall Timepoint Response

The investigator's assessment of a patient's target lesion response, non-target lesion response, and appearance of new lesions (collected from the CRF) will be used to determine the overall tumor response at each time point as shown in Table 1 (for patients with target lesions (with or without non-target lesions)) and Table 2 (for patients with non-target lesions only).

The possible overall tumor responses at a time point, from best to worst, are as follows.

- Complete Response (CR)
- Partial Response (PR)
- Stable Disease (SD)
- Progressive Disease (PD)

If no assessment was done or a response cannot be determined, overall timepoint response is designated as Not Evaluable (NE).

Plexxikon Inc. PLX121-01 Statistical Analysis Plan 01Jul2020

Table 1. Time Point Response: Patients with Target (+/- Non-Target) Disease

| Target Lesion | Non-Target Lesions | New Lesions | Overall<br>(Time point)<br>Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

Table 2. Time Point Response: Patients with Non-Target Disease Only

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------------------|
| CR | No | CR |
| Non-CR/Non-PD | No | Non-CR/non-PD <sup>[1]</sup> |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

CR = Complete Response; PR = Partial Response; SD = Stable Disease; PD = Progressive Disease; NE = Not Evaluable.

Note: 'Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as endpoint for assessment of efficacy in some trials so to assign this category when no lesions can be measured is not advised.

The date of the assessment of tumor response for a time point is the earliest date of target, non-target or new lesion assessment dates. If all of these dates are missing, the date of tumor response assessment is used.

## 8.1.2 Best Response

The best responses for pairs of time point responses (when confirmation of CR and PR are required) are determined as shown in Table 3. Table 3 is an extended version of the corresponding RECIST table. The additional discussion provided here clarify how Best Responses for individual pairs of Overall Time Point Responses, i.e., paired by sequential time points, are determined. The Best Responses will then be used to determine Best Overall Response (Section 8.1.3).

In Table 3, the first and subsequent time points referenced in the column headers refer to an arbitrary pair of sequential time points. Also, as indicated in the table and in the table notes, special rules may apply when the first time point of the pair is the very first (post-treatment) assessment time point or when there is only one assessment.

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

Table 3. Best Response When Confirmation of CR and PR are Required

| | Overall<br>Response<br>First<br>Time Point | Overall<br>Response<br>Subsequent<br>Time Point | Best Response for the Pair |
|---|---|---|---|
| 1 | CR | CR | CR (if minimum criteria for CR duration is met), otherwise Best Response = NE. |
| 2 | CR | PR | If the first time point is truly CR, any worsening at a subsequent time point—even disease meeting the PR criteria—makes the disease PD at that subsequent time point. Then <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met at the first time point; otherwise <b>Best Response</b> = <b>PD</b> . However, sometimes 'CR' may still be claimed when subsequent scans suggest small lesions that were likely present and in fact, the patient had PR, not CR, at the first time point. Under these circumstances, the original CR should be changed to PR; see <b>Row 6 for Best Response criteria</b> . |
| 3 | CR | SD | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met by the second time point; otherwise <b>Best Response</b> = <b>PD</b> . |
| 4 | CR, PR, SD | PD | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met at the first time point; otherwise <b>Best Response</b> = <b>PD</b> . |
| 5 | CR, PR | NE | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met at the first time point; otherwise <b>Best Response</b> = <b>NE</b> . |
| 6 | PR | CR, PR | <b>Best Response</b> = <b>PR</b> provided minimum criteria for PR duration is met; otherwise, <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met by the second time point; otherwise <b>Best Response</b> = <b>NE</b> . |
| 7 | PR | SD | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met by the second time point; otherwise <b>Best Response</b> = <b>NE</b> . |
| 8 | SD | SD, CR, PR | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met by the second time point; otherwise <b>Best Response</b> = <b>NE</b> . |
| 9 | SD | NE | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met at the first time point; otherwise <b>Best Response</b> = <b>NE</b> . |
| 10 | SD | PD | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met at the first time point; otherwise <b>Best Response</b> = <b>PD</b> . |
| 11 | PD | CR, PR, SD,<br>PD, NE | Best Response = PD. |
| 12 | NE | CR, PR, SD, NE | Best Response = NE. |
| 13 | NE | PD | Best Response = PD. |
| 14 | CR, PR, SD | No 2 <sup>nd</sup> visit | <b>Best Response</b> = <b>SD</b> provided minimum criteria for SD duration is met at first time point; otherwise <b>Best Response</b> = <b>NE</b> . |
| 15 | PD | No 2 <sup>nd</sup> visit | Best Response = PD. |
| 16 | NE | No 2 <sup>nd</sup> visit | Best Response = NE. |

CR = complete response, PR = partial response, SD = stable disease, PD = progressive disease, NE = not evaluable.

Note: If response = SD, CR, or PR at the initial post-treatment assessment then, in meeting the minimum criteria for SD duration (only SD, not CR or PR), duration is measured from the treatment start date rather than the date of the assessment.

Note: In some situations, it may be necessary to check across more than two sequential time points in order to determine whether or not a minimum duration criteria has been met. The same logic as used for the pairs of time points should be applied. For example, for the triplet SD CR SD, duration is calculated from the first assessment date (or from the treatment start date if these are the initial assessments) to the third assessment date, if needed, to determine whether the minimum criteria for SD duration has been met.

Per the RECIST guidance and as indicated in the first table note, for patients with SD at the first time point: in determining whether the minimum criteria for SD duration is met, duration is measured from the treatment start date to that first assessment date. Then, if the duration meets the minimum interval requirement for SD, **Best Response** = **SD**, otherwise **Best Response** = **NE**. Further, as indicated in the note, this same rule is also applied to patients with a response better than SD at the first time point.

In some situations, it may be necessary to check across more than two sequential time points in order to determine whether or not a minimum duration criteria has been met. The same logic as used for the pairs of time points should be applied. For example, note the following examples.

- For the triplet SD CR/PR/SD SD, duration is calculated from the first assessment date (or from the treatment start date if these are the initial assessments) to the third assessment date, if needed, to determine whether the minimum criteria for SD duration has been met. If it is met, then **Best Response** = **SD**. Otherwise, **Best Response** = **NE**.
- For the triplet CR NE CR, if the minimum criteria for CR duration is met for the interval between the two CR assessments, then **Best Response** = **CR**. Otherwise **Best Response** = **NE**.
- For the triplet PR NE PR, if the minimum interval criteria for PR is met for the interval between the two PR assessments, then Best Response = PR. Otherwise Best Response = NE.
- For the triplet SD NE SD, **Best Response** = **NE**.

The minimum interval for confirmation of CR and PR is 4 weeks—the minimum of the range suggested in RECIST. The minimum interval for duration of SD is 8 weeks (i.e. 49 days taking visit window of +/-7 days into consideration).

#### 8.1.3 Best Overall Response

A Best Response is determined for each sequential pair of post-treatment time points (and in some cases, triplets of sequential time points) as indicated in the previous section, Section 8.1.2. Then, the Best Overall Response for a patient (when confirmation of CR and PR are required) is the best of these Best Responses.

## 8.2 Efficacy Variables

The efficacy variables for Part 1, Part 2b, and Part 2e are as follows.

• Response to treatment according to RECIST version 1.1.

- Best Overall Response is the best of the best responses (with confirmation), as detailed in the previous section
- ORR, defined as the number of patients who have a Best Overall Response of CR or PR divided by the total number of patients in the efficacy evaluable population.
- Progression-free Survival (PFS), defined as the number of days from the first day of treatment (C1D1) to the first documented PI assessment using RECIST criteria of disease progression/relapse or date of death prior to discontinuing treatment of PLX9486, whichever occurs first. The date of disease progression is earliest overall timepoint response of PI assessed PD as defined in Section 8.1.1. Patients without an assessment of disease progression/relapse who discontinue PLX9486 or discontinue from the study and indicate progressive disease or clinical progression as the primary reason for ending PLX9486 or study discontinuation will be counted as having progressed on their last dose date (if primary reason for ending treatment is progressive disease or clinical progression or death) or on their study exit date (if the primary reason for study exit is progressive disease or clinical progression or death). Patients who discontinue from the trial without having a post-baseline scan will be censored at study day 2. If disease progression/relapse/death does not occur and the patient does not discontinue PLX9486 due to clinical progression, PFS is censored as of the date of patient's last imaging exam of target or non-target lesions. See Figure 1 for a decision flowchart.
- 6-month PFS rate, defined as the number of patients with PFS of at least 180 days divided by the total number of patients in the efficacy evaluable population.
- DOR is calculated for every patient with a response to therapy and is defined as the number of days from the date of first response (PR or CR confirmed at least 28 days later) to the date of first documented disease progression/relapse or death, whichever occurs first. For the date of disease progression and the date censored, the same rules described as above for PFS are used.
- Clinical Benefit Rate: Patients are considered to experience clinical benefit if they have a Best Overall Response of SD that lasted for at least 16 weeks, or confirmed Best Overall Response of PR or CR. The Clinical Benefit Rate (CBR) is defined as the number of patients who have CBR divided by the total number of patients in the efficacy evaluable population.
- Overall Survival (OS), defined as the number of days from the first day of treatment (C1D1) until the date of death. If a patient is lost to follow-up, OS is censored at the date of last contact. Date of last contact is the latest dates among the visit dates recorded in the following CRF forms: Hematology, Chemistry, Coagulation, Urinalysis, Vital Signs, ECG, Physical Exam, Tumor Assessments (Target, Non-Target), and study drug dosing logs (PLX9486, PX3397, Sunitinib), Study Exit Status, Phone Interview where patient status is recorded as alive.
- 12-month OS rate, defined as the number of patients alive at 12 months (365 days) divided by the total number of patients in the efficacy evaluable population.
- Biomarkers in peripheral blood, in archival tumor tissue and in available tumor biopsies

Biomarker descriptive statistics is not in the scope of this SAP, except for the summary of tumor markers.

Figure 1 – PFS Decision Flowchart



 $PFS = Progression \ free \ survival; \ PI = Primary \ investigator; \ PD = Progressive \ disease.$ 

Red boxes indicate PFS decision events. Magenta boxes indicate censored decision events.

<sup>&</sup>lt;sup>a</sup> For events using a minimum date, the minimum of the dates of PD, withdrawal from PLX9486, and the death date if they exist is used as the date of the event.

### 8.3 Adjustments for Covariates

No adjustments for covariates are planned.

## 8.4 Handling of Dropouts or Missing Data

No imputations will be made for missing values except as noted in considering a NE response for determining timepoint response and Best Overall Response.

## 8.5 Interim Analysis and Data Monitoring

There are no planned interim analyses.

## 8.6 Examination of Subgroups

There are no planned subgroup efficacy analyses.

## 8.7 Multiple Comparison/Multiplicity

No adjustments for multiplicity or multiple testing will be made.

## 8.8 Multicenter Studies

There are no analyses planned to compare differences in response by site.

## 8.9 Methods of Efficacy Analysis

Patients' target lesion response, non-target lesion response, and appearance of new lesions at each time point, the overall tumor response at each time point and the Best Overall Response will be shown in listings. The target lesion assessment listing will also include change and percent change from baseline of the sum of the longest diameter from the target lesions. Nadir (the smallest sum of longest diameters of target lesions recorded since treatment started), change from nadir and the percent change from nadir will also be provided in this listing.

The number and percent of patients in each category of best overall response (CR, PR, SD, PD, and NE) will be summarized along with the ORR and CBR. Exact two-sided binomial 95% confidence intervals (CIs) will be provided for each category response and the ORR and CBR. 6-month PFS rate and 12-month OS rates will be summarized by dose cohorts and overall and the two-sided, exact binomial 95% confidence interval for these rates will be provided.

OS, PFS and DOR (in days) will be estimated using Kaplan-Meier method. The number and percentages of patients who progressed or died and who did not, will be summarized by cohort and overall. The Kaplan-Meier estimate of the 25<sup>th</sup>, median and 75<sup>th</sup> percentiles and their two-sided 95% confidence intervals will be presented by study part, dose cohort and overall. Range of DOR and PFS for all patients and for patients who progressed or died will also be presented by study part, dose cohort and overall.

Cox proportional hazards regression may be used to perform exploratory post-hoc analyses to investigate the contributions of various factors to OS, PFS and DOR.

A figure of PFS by Study Part and Cohort will also be provided.

## 9. PHARMACOKINETIC ANALYSES

A separate formal PK report will be written for inclusion in the final study report. Synteract is not responsible for PK analysis.

#### 10. PHARMACODYNAMIC ANALYSES

Exploratory PD parameters will be analyzed appropriately (if samples are available). No formal statistical analysis of pharmacodynamics endpoints will be performed.

The exploratory PD endpoints of Part 1, Part 2b, and Part 2e of this study includes biomarkers in peripheral blood, in archival tumor tissue, and in available tumor biopsies. Patients with collected tumor marker sample will be listed by cohort and patient and display the collection date, collection time, test type, and result (in units).

Synteract is not responsible for PD analysis.

#### 11. SAFETY ANALYSES

All safety analyses will be based on the safety population and summarized for each dose escalation cohort Safety variables to be assessed will include AEs, laboratory test results (hematology, serum chemistry, and urinalysis), ECGs, weight, and vital signs.

#### 11.1 Extent of Exposure

Summary of duration for each study drug and total dose taken (mg) will be summarized by study part, cohort, and overall. Duration of treatment for each study drug (PLX9486, PLX3397 and sunitinib) is defined as the last dose date of that study drug minus the first dose date of that study drug plus 1. The overall duration of treatment is defined as the last dose date of any study drug (PLX9486, PLX3397, sunitinib) minus the first dose date of any study drug (PLX9486, PLX3397, sunitinib) plus 1.

Drug administration and accountability will be presented in data listings.

#### 11.2 Adverse Events

An adverse event (AE) is any untoward medical occurrence in a patient administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. An AE can be any unfavorable and unintended sign (e.g., including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not it is considered to be study drug related. This includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. An AE includes, but is not limited to, the following:

• Any clinically significant worsening of a preexisting condition.

- An AE occurring from overdose (i.e., a dose higher than that indicated in the protocol) of a test article, whether accidental or intentional.
- An AE occurring from abuse (e.g., use for nonclinical reasons) of a study drug.
- An AE that has been associated with the discontinuation of the use of a study drug.

A serious adverse event (SAE) is an AE that:

- Results in death.
- Is life-threatening.
- Requires inpatient hospitalization longer than 24 hours or prolongation of existing hospitalization (see clarification in the protocol on planned hospitalizations). An emergency room visit without hospitalization is not considered a hospitalization.
- Results in persistent or significant disability or incapacity. Disability is defined as a substantial disruption of a person's ability to conduct normal life functions.
- Is a congenital anomaly or birth defect.
- Is an important medical event. An important medical event is an event that may not result in death, be life-threatening, or require hospitalization but may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in the definitions for SAEs.

All AE summaries will be restricted to TEAEs, which are defined as those AEs that occurred on or after dosing, and those existing AEs that worsened during the study. Furthermore, an AE is not considered treatment emergent if it is not treatment related and its onset is more than 28 days after the last dose of study drug. If it cannot be determined whether the AE is treatment emergent due to a partial onset date then it will be counted as such. See Appendix 1 for handling of partial dates for AEs. Verbatim terms on case report forms will be mapped to preferred terms and system organ classes using the Medical Dictionary for Regulatory Activities (MedDRA) v18.0.

Each AE summary will be displayed by cohort and overall. Summaries that are displayed by system organ class and preferred terms will be ordered by descending order of incidence of system organ class and preferred term within each system organ class. Summaries of the following types will be presented.

Summaries of treatment-related TEAEs include all events reported as "Possibly Related" or "Probably Related" to any of Study Treatment (PLX9486, PLX3397, and sunitinib). At each level of patient summarization, a patient is classified according to the closest relationship if the patient reported one or more events. AEs with a missing relationship are not included.

For summaries of TEAEs by highest severity, at each level of patient summarization a patient is classified according to the highest severity if the patient reported one or more events. AEs with missing severity are not included.

Summary tables will be produced for the following:

- Overall Summary of TEAEs, including summaries of total number of TEAEs, number of
  patients with at least one TEAE, number of patients with at least one treatment-emergent
  SAE, number of patients with at least one related TEAE, number of patients with at least
  one treatment-emergent related SAE, and number of patients with at least one TEAE
  leading to permanent withdrawal of study product (any of PLX9486, PLX3397, and
  sunitinib) or discontinuation from the study.
- Patient incidence of TEAEs by MedDRA system organ class and preferred term.
- Patient incidence of TEAEs by preferred term and highest severity grade orderd by descending order of the overall count of TEAEs
- Patient incidence of treatment-related TEAEs by preferred term and highest severity grade.
- Patient incidence of PLX9486-Related TEAEs by preferred term (Safety Population) and highest severity grade.
- Patient incidence of PLX3397-Related TEAEs by preferred term (Safety Population) and highest severity grade.
- Patient incidence of Sunitinib-Related TEAEs by preferred term (Safety Population) and highest severity grade.

AEs leading to permanent withdrawal of study drug or discontinuation from the study are defined as those having an action of "Drug Withdrawn" for any of study drugs (PLX9486, PLX3397, and sunitinib), or primary AEs associated with records from the CRF forms 'End of Treatment' or 'Study Exit Status' where the reason for end of treatment or for study exit is 'Adverse Event'. Listings of all AEs, SAEs, AEs leading to changes in study treatment, AEs leading to death, and dose limiting toxicity will be provided. Summary listing of deaths will also be provided.

## 11.3 Clinical Laboratory Evaluation

Laboratory results (hematology and coagulation tests, serum chemistry) will be summarized by study part, cohort and overall using descriptive statistics at baseline and at each scheduled post-baseline time point. Changes from baseline of laboratory results will also be summarized by study part, cohort and overall.

Select laboratory analytes will be graded according to National Cancer Institute CTCAE as shown in Appendix 2. The worst scheduled post-baseline CTCAE grade for each analyte will be summarized by study part, cohort and overall in shift tables to assess changes from baseline for applicable hematology and coagulation analytes (WBC, hemoglobin, lymphocytes, platelets, ANC, aPTT and INR) and applicable chemistry analytes (ALT, AST, alkaline phosphatase, direct bilirubin, total bilirubin, creatinine and phosphorus). In the hematology shift table, the following analytes will have a shift table for high and low grading: WBC, hemoglobin, and lymphocytes. Laboratory results (hematology, serum chemistry, urinalysis, and coagulation tests) will be presented in data listings. Abnormal values will be flagged as high or low relative to the local lab normal ranges, where applicable. Values that are deemed as abnormal, clinically significant (as collected on the CRF) will also be flagged. CTCAE v4.03 grades are included in these listings where applicable. In addition, listings of hematology results and chemistry results with CTCAE grade 3 or higher will be provided.

## 11.4 Vital Signs

The baseline value is defined as the last non-missing value obtained before the date and time of the first dose of any study drug or on pre-dose timepoint of the first dose date of any study drug.

Vital signs (heart rate, respiratory rate, blood pressure, temperature and weight) will be summarized by cohort using descriptive statistics at baseline and at each scheduled post-baseline time point. Changes from baseline will also be summarized.

A listing of vital signs will be provided.

## 11.5 Physical Examination

Physical examination findings will be included in a data listing only.

## 11.6 Electrocardiogram

The ECG data analysis will be conducted based on methodology recommended in the International Conference on Harmonization E14 guidance, The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-antiarrhymic Drugs [2].

To compensate for the effect of heart rate on QT interval, heart rate corrections will be computed for each observed QT interval using Fridericia's correction (QTcF) and will be included in the data listings. QT is the unadjusted QT interval in milliseconds and RR is the RR interval in milliseconds. The RR interval will be calculated from heart rate using the following formula:

• RR (milliseconds) = 60\*1000 / [heart rate in beats per minute]

Then, the definitions of the heart-rate corrected QT intervals (in milliseconds) are:

• QTcF = QT /  $[(RR/1000)^{1/3}]$  or, equivalently, QT /  $[(60/heart rate)^{1/3}]$ 

where, again, heart rate is in beats per minute.

Triplicate ECG measurements are collected. The average value of the ECG triplicates for ECG parameters (heart rate, pulse rate, RR, QRS, QT, and QTcF) will be summarized using descriptive statistics at baseline and at each scheduled post-baseline time point. Changes from baseline of the average values of the ECG triplicates will also be summarized. The derived RR and QTcF will be used in this summary. A one-sided upper 95% CI will be included for each change from baseline time point for QTcF.

The derived RR and QTcF values and the collected values in the eCRF for other ECG parameters will be displayed in a data listing. In addition, change from baseline in the derived QTcF will also be included in this listing. Outlier QTc values are those that meet at least one of the following criteria: (1) QTcF  $\geq$  450 msec (for males) or  $\geq$  470 msec (for females) or (2) increase from baseline in QTcF >30 msec. A summary of the number and percentage of patients who experience outlier QTc values will be summarized by cohort. The individual patient QTc data meeting the outlier criteria described above flagged in the data listing.

## 11.7 Eastern Cooperative Oncology Group (ECOG)

Eastern Cooperative Oncology Group (ECOG) performance data will be summarized using a shift table to assess changes from baseline for each cohort. ECOG data will be presented in a patient listing for all patients.

## 11.8 Other Collected Samples

Other selected disease related samples which were collected will be slisted including circulating DNA samples, tumor marker samples, archival tumor tissue collection, and optional paired tumor biopsy collection

## 8. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

The Efficacy Evaluable population will include patients that discontinued treatment due to disease progression or died prior to having a post-baseline assessment.

Analyses for the exploratory objective to assess tumor response in the Part 2 cohorts by Choi's criteria will not be conducted.

PK and PD analyses (including the specification of window timing of PK and PD measurements) are not covered in this document.

The RR value derived from heart rate will be used in any derivations (eg, in the derivation of QTcF) rather than the value collected on the eCRF. Further, the derived QTcB and QTcF values rather than the QTcB and QTcF values collected in the eCRF will be used for all analyses.

## **REFERENCES**

- 1. National Cancer Institute Common Terminology Criteria for Adverse Events v4.03, NCI, NIH, DHHS, June 14, 2010, NIH publication # 09-7473.
- 2. Guidance for Industry E14 The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-antiarrhythmic Drugs, U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), October 2005.

## **APPENDIX 1: PARTIAL DATE CONVENTIONS**

Imputed dates will NOT be presented in the listings.

Algorithm for Treatment Emergence of Adverse Events

| Start Date | Stop Date | Action |
|---|---|---|
| Known | Known/Partial/Missing | If start date $\leq$ study med start date, then not TEAE;<br>If start date $\geq$ study med start date and (start date $\leq$ (study med end date $+$ 28) or related), then TEAE. |
| | 1 | 1 |
| Partial, but known components show that it cannot be on or | W /Dankin 1/0 dinning | N. A. T.E. A. E. |
| after study med start date | Known/Partial/Missing | Not TEAE |
| Partial, could be on or after study med start date | Known | If stop date < study med start date, then not TEAE;<br>If stop date ≥ study med start date, then TEAE. |
| | | Impute stop date as latest possible date (i.e. last day of month if day is unknown or 31 December if day and month are unknown), then: If stop date < study med start date, then not TEAE; |
| | Partial | If stop date \geq study med start date, then not TEAE, If stop date \geq study med start date, then TEAE. |
| | Missing | Assumed TEAE |
| | 1 | |
| Missing | Known | If stop date < study med start date, then not TEAE;<br>If stop date ≥ study med start date, then TEAE. |
| | | Impute stop date as latest possible date (i.e. last day of month if day is unknown or 31 December if day and month are unknown), then: |
| | Partial | If stop date < study med start date, then not TEAE;<br>If stop date ≥ study med start date, then TEAE. |
| | Missing | Assumed TEAE |

## Algorithm for Prior/Concomitant Medications

| Start<br>Date | Stop Date | Action |
|---|---|---|
| Known | Known/Partial/Missing | If start date < study med start date, then assign as prior; If start date ≥ study med start date and start date ≤ end of treatment (latest last dose of any study medication), then assign as concomitant |
| Partial | Known/Partial/Missing | Impute start date as earliest possible date (i.e. first day of month if day is unknown or 1st January if day and month are unknown), then: If start date < study med start date, then assign as prior; If start date ≥ study med start date and start date ≤ end of treatment, then assign as concomitant |
| | 1 | |
| Missing | Known | If stop date < study med start date, then assign as prior;<br>If stop date ≥ study med start date, then assign as concomitant |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day is unknown or 31 December if day and month are unknown), then: If stop date < study med start date, then assign as prior; If stop date ≥ study med start date, then assign as concomitant |
| | Missing | Assign as concomitant |

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

## APPENDIX 2: CTCAE TOXICITY GRADES FOR LABORATORY ANALYTES

## CTCAE Toxicity Grades: Hematology and Coagulation

| Analyte | Standard<br>Unit | Directional Change | Toxicity Grades (CTCAE v4.03) |
|---|---|---|---|
| Hemoglobin <sup>[1]</sup> | g/dL | Decrease | Grade 1: $<$ LLN $-$ 10.0 g/dL |
| | | | Grade 2: $< 10.0 - 8.0 \text{ g/dL}$ |
| | | | Grade 3: < 8.0 |
| | | | Grade 4: Not defined |
| | | Increase | Grade 1: $> ULN - (2+ULN) g/dL$ |
| | | | Grade 2: $> (2+ULN) - (4+ULN) g/dL$ |
| | | | Grade 3: $> 4+ULN g/dL$ |
| | | | Grade 4: Not defined |
| ANC | x10^9/L | Decrease | Grade 1: $< LLN - 1.5 \times 10^{9}/L$ |
| | | | Grade 2: $< 1.5 - 1.0 \times 10^{9}$ L |
| | | | Grade 3: $< 1.0 - 0.5 \times 10^{9}$ L |
| | | | Grade 4: $< 0.5 \text{ x} 10^{9}/\text{L}$ |
| Platelets | x10^9/L | Decrease | Grade 1: < LLN – 75.0 x10^9/L |
| | | | Grade 2: $< 75.0 - 50.0 \times 10^{9}$ L |
| | | | Grade 3: $< 50.0 - 25.0 \times 10^{9}$ L |
| | | | Grade 4: $< 25.0 \text{ x} 10^{9}/\text{L}$ |
| WBC | x10^9/L | Decrease | Grade 1: $<$ LLN $- 3.0 \times 10^{9}$ /L |
| | | | Grade 2: $< 3.0 - 2.0 \times 10^{9}/L$ |
| | | | Grade 3: $< 2.0 - 1.0 \times 10^{9}/L$ |
| | | | Grade 4: $< 1.0 \text{ x} 10^9/\text{L}$ |
| | | Increase | Grade 1: Not defined |
| | | | Grade 2: Not defined |
| | | | Grade 3: $>100 \times 10^{9}$ L |
| | | | Grade 4: Not defined |
| Lymphocytes | x10^9/L | Decrease | Grade 1: $<$ LLN $-$ 0.8 x10^9/L |
| | | | Grade 2: $< 0.8 - 0.5 \times 10^{9}$ L |
| | | | Grade 3: $< 0.5 - 0.2 \times 10^{9}/L$ |
| | | | Grade 4: $< 0.2 \times 10^9/L$ |
| | x10^9/L | Increase | Grade 1: Not defined |
| | | | Grade 2: $>4.0 - 20.0 \text{ x} 10^9/\text{L}$ |
| | | | Grade 3: $>20.0 \times 10^{9}/L$ |
| | | | Grade 4: Not defined |
| aPTT | sec | Increase | Grade 1: >ULN − 1.5 x ULN |
| | | | Grade 2: $>1.5 - 2.5 \times ULN$ |
| | | | Grade 3: >2.5 x ULN |
| | | | Grade 4: Not defined |
| INR | No units | Increase | Grade 1: >ULN – 1.5 x ULN |
| | | | Grade 2: $>1.5 - 2.5 \times ULN$ |
| | | | Grade 3: >2.5 x ULN |
| | | | Grade 4: Not defined |

LLN=lower limit of normal; ULN=upper limit of normal. The LLN and ULN for each analyte will be determined from the normal range of each local laboratory.

| Analyte | Standard<br>Unit | Directional Change | Toxicity Grades (CTCAE v4.03) |
|---|---|---|---|
| [1] For increased hemoglobin results, if the baseline value is above the ULN, the baseline value will be used instead of the ULN to assess grades 1, 2, and 3. | | | |

## CTCAE Toxicity Grades: Serum Chemistry

| Analyte | Standard<br>Unit | Directional<br>Change | Toxicity Grades (CTCAE v4.03) |
|---|---|---|---|
| Albumin | g/dL | Decrease | Grade 1: < LLN – 3.0 g/dL |
| | Ü | | Grade 2: $< 3.0 - 2.0 \text{ g/dL}$ |
| | | | Grade 3: < 2.0 g/dL |
| | | | Grade 4: Not defined |
| Alkaline Phosphatase | U/L | Increase | Grade 1: > ULN − 2.5 x ULN |
| • | | | Grade 2: $> 2.5 - 5.0 \text{ x ULN}$ |
| | | | Grade 3: $> 5.0 - 20.0 \text{ x ULN}$ |
| | | | Grade 4: $> 20.0 \text{ x ULN}$ |
| ALT (SGPT) | U/L | Increase | Grade 1: $>$ ULN $-$ 3.0 x ULN |
| | | | Grade 2: $> 3.0 - 5.0 \text{ x ULN}$ |
| | | | Grade 3: $> 5.0 - 20.0 \text{ x ULN}$ |
| | | | Grade 4: $> 20.0 \times ULN$ |
| AST (SGOT) | U/L | Increase | Grade 1: $>$ ULN $-$ 3.0 x ULN |
| | | | Grade 2: $> 3.0 - 5.0 \text{ x ULN}$ |
| | | | Grade 3: $> 5.0 - 20.0 \text{ x ULN}$ |
| | | | Grade 4: $> 20.0 \text{ x ULN}$ |
| Calcium | mg/dL | Decrease | Grade 1: $<$ LLN $-$ 8.0 mg/dL |
| | | | Grade 2: $< 8.0 - 7.0 \text{ mg/dL}$ |
| | | | Grade 3: $< 7.0 - 6.0 \text{ mg/dL}$ |
| | | | Grade 4: $< 6.0 \text{ mg/dL}$ |
| | | Increase | Grade 1: >ULN – 11.5 mg/dL |
| | | | Grade 2: >11.5 – 12.5 mg/dL |
| | | | Grade 3: >12.5 – 13.5 mg/dL |
| | | | Grade 4: >13.5 mg/dL |
| Creatinine | mg/dL | Increase | Grade 1: $>$ ULN $-$ 1.5 x ULN |
| | | | Grade 2: $> 1.5 - 3.0 \text{ x ULN}$ |
| | | | Grade 3: $> 3.0 - 6.0 \text{ x ULN}$ |
| | | | Grade 4: $> 6.0 \text{ x ULN}$ |
| Creatine | | | |
| Phosphokinase (CPK) | U/L | Increase | Grade 1: $>$ ULN - 2.5 x ULN |
| | | | Grade 2: $>2.5 \times ULN - 5 \times ULN$ |
| | | | Grade 3: $>5$ x ULN - $10$ x ULN |
| | | | Grade 4: $>10 \times ULN$ |
| Direct Bilirubin | mg/dL | Increase | Grade 1: $>$ ULN $-$ 1.5 x ULN |
| | | | Grade 2: $>1.5 - 3.0 \text{ x ULN}$ |
| | | | Grade 3: $>3.0 - 10.0 \text{ x ULN}$ |
| | | | Grade 4: >10.0 x ULN |
| Total Bilirubin | mg/dL | Increase | Grade 1: $>$ ULN $-$ 1.5 x ULN |
| | | | Grade 2: $>1.5 - 3.0 \text{ x ULN}$ |
| | | | Grade 3: $>3.0 - 10.0 \text{ x ULN}$ |
| | | | Grade 4: >10.0 x ULN |
| Glucose | mg/dL | Decrease | Grade 1: $<$ LLN $-$ 55 mg/dL |
| | | | Grade 2: $< 55 - 40 \text{ mg/dL}$ |
| | | | Grade 3: $< 40 - 30 \text{ mg/dL}$ |

| Analyte | Standard<br>Unit | Directional<br>Change | Toxicity Grades<br>(CTCAE v4.03) |
|---|---|---|---|
| | | | Grade 4: < 30 mg/dL |
| | | Increase | Grade 1: $>$ ULN $-$ 160 mg/dL |
| | | | Grade 2: $> 160 - 250 \text{ mg/dL}$ |
| | | | Grade 3: $> 250 - 500 \text{ mg/dL}$ |
| | | | Grade 4: > 500 mg/dL |
| Magnesium | mg/dL | Decrease | Grade 1: <lln -="" 1.2="" dl<="" mg="" td=""></lln> |
| | | | Grade 2: <1.2 - 0.9 mg/dL |
| | | | Grade 3: <0.9 - 0.7 mg/dL |
| | | | Grade 4: <0.7 mg/dL; |
| | | Increase | Grade 1: >ULN - 3.0 mg/dL |
| | | | Grade 2: Not defined |
| | | | Grade 3: >3.0 - 8.0 mg/dL |
| | | | Grade 4: >8.0 mg/dL |
| Phosphorus | mg/dL | Decrease | Grade 1: $<$ LLN $-$ 2.5 mg/dL |
| | | | Grade 2: $< 2.5 - 2.0 \text{ mg/dL}$ |
| | | | Grade 3: $< 2.0 - 1.0 \text{ mg/dL}$ |
| | | | Grade 4: < 1.0 mg/dL |
| Potassium | mmol/L | Decrease | Grade 1: < LLN – 3.0 mmol/L |
| | | | Grade 2: Not defined |
| | | | Grade 3: $< 3.0 - 2.5 \text{ mmol/L}$ |
| | | | Grade 4: < 2.5 mmol/L |
| | mmol/L | Increase | Grade 1: $> ULN - 5.5 \text{ mmol/L}$ |
| | | | Grade 2: $> 5.5 - 6.0 \text{ mmol/L}$ |
| | | | Grade 3: $> 6.0 - 7.0 \text{ mmol/L}$ |
| | | | Grade 4: > 7.0 mmol/L |
| Sodium | mmol/L | Decrease | Grade 1: < LLN – 130 mmol/L |
| | | | Grade 2: Not defined |
| | | | Grade 3: < 130 – 120 mmol/L |
| | | | Grade 4: < 120 mmol/L |
| | | Increase | Grade 1: > ULN – 150 mmol/L |
| | | | Grade 2: > 150 – 155 mmol/L |
| | | | Grade 3: > 155 – 160 mmol/L |
| | | | Grade 4: > 160 mmol/L |
| Uric Acid | mg/dL | Increase | Grade 1: >ULN - 10 mg/dL |
| | | | Grade 2: Not defined |
| | | | Grade 3: Not defined |
| | | | Grade 4: >10 mg/dL |

LLN=lower limit of normal; ULN=upper limit of normal. The LLN and ULN for each analyte will be determined from the normal range of each local laboratory.

## **APPENDICES**

## Appendix A: List of Tables, Figures, and Listings

### List of Tables

| List of Table ICH Heading | Table Number | Table Description |
|---|---|---|
| 14.1 | Table Number | Demographics |
| 14.1 | 14.1.1 | Summary of Patient Disposition (All Patients) |
| | 14.1.2 | Summary of Demographic and Baseline Characteristics (Safety Population) |
| | 14.1.3 | Summary of Medical History (Safety Population) |
| | 14.1.4 | Summary of Prior Medications (Safety Population) |
| | 14.1.5 | Summary of Concomitant Medications (Safety Population) |
| 14.2 | 14.1.3 | Efficacy |
| 17,2 | 14.2.1 | Best Overall Tumor Response (Efficacy Evaluable Population) |
| | 14.2.2 | Duration of Response (Efficacy Evaluable Population) |
| | 14.2.3 | Progression-Free Survival (Efficacy Evaluable Population) |
| | 14.2.4 | Overall Survival (Efficacy Evaluable Population) |
| 14.3 | 14.2.4 | Safety |
| 14.3.1 | | Adverse Events |
| 14.3.1 | 14211 | |
| | 14.3.1.1 | Overall Summary of Treatment-Emergent Adverse Events (Safety Population) |
| | 14.3.1.2 | Summary of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term (Safety Population) |
| | 14.3.1.3 | Summary of Treatment-Emergent Adverse Events by System Organ Class and Severity Grade (Safety Population) |
| | 14.3.1.4.1 | Summary of Any Drug-Related Treatment-Emergent Adverse Events by Preferred Term and Severity Grade (Safety Population) |
| | 14.3.1.4.2 | Summary of PLX9486-Related Treatment-Emergent Adverse Events by Preferred Term and Severity Grade (Safety Population) |
| | 14.3.1.4.3 | Summary of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Relatedness (Safety Population) |
| 14.3.2 | | Listings of Deaths, Other Serious and Significant Adverse Events |
| | 14.3.2.1 | Summary Listing of Deaths |
| | 14.3.2.2 | Summary Listing of Serious Adverse Events (Safety Population) |
| Other Safety | | Laboratory |
| , | 14.3.4.1.1 | Summary of Hematology and Coagulation by Cycle and Day (Safety Population) |
| | 14.3.4.1.2 | Summary of Hematology and Coagulation - CTCAE Shift from Baseline (Safety Population) |
| | 14.3.4.2.1 | Summary of Serum Chemistry by Cycle and Day (Safety Population) |
| | 14.3.4.2.2 | Summary of Serum Chemistry - CTCAE Shift from Baseline (Safety Population) |
| | | Exposure |
| | 14.3.5.1 | Summary of PLX9486 Exposure (Safety Population) |
| | 14.3.5.2 | Summary of PLX3397 Exposure (Safety Population) |
| | 14.3.5.3 | Summary of Sunitinib Exposure (Safety Population) |
| | | Other Data |
| | 14.3.6 | Summary of Vital Signs (Safety Population) |
| | 14.3.7.1 | Summary of Electrocardiogram (Safety Population) |
| | 14.3.7.2 | Summary of Electrocardiogram – Abnormal QTcF Results (Safety Population) |
| | 14.3.8 | Summary of ECOG – Shift from Baseline (Safety Population) |

## **List of Figures**

| ICH Heading | Table Number | Table Description |
|---|---|---|
| | 14.2.1 | Progression-Free Survival by Study Part – Study Part 1 (Efficacy Evaluable Population) |

Clinical Study Report PLX121-01

Plexxikon Inc.Statistical Analysis PlanPLX121-0130Jun2020

Listings

| ICH<br>Heading | Listing<br>Number | Listing Description | CRF Form(s) |
|---|---|---|---|
| 16.2 | | PATIENT DATA LISTINGS | |
| 16.2.1 | 1 Discontinued patients | | |
| | 16.2.1.1 | Patient Disposition | Study Exit Status, End of Treatment,<br>Demographics |
| 16.2.2 | | Demographics and Baseline Characteristics | |
| | 16.2.2.1 | Demographics and Baseline Characteristics | Demographics, Vital Signs |
| | 16.2.2.2 | Medical History | Medical History |
| | 16.2.2.3.1 | Primary Cancer History – Study Part 1 | Primary Cancer History |
| | 16.2.2.3.2 | Primary Cancer History – Study Part 2 | Primary Cancer History – Part 2 |
| | 16.2.2.4 | Prior Treatment for Primary Malignancy | Prior Treatment for Primary Malignancy |
| | 16.2.2.5 | Prior and Concomitant Medications | Concomitant Medications |
| | 16.2.2.6 | Major Protocol Deviations | |
| 16.2.3 | | Study Drug Exposure | |
| | 16.2.3.1.1 | PLX9486 Dosing Log | PLX9486 Study Drug Dosing Log |
| | 16.2.3.1.2 | PLX3397 Dosing Log | PLX3397 Study Drug Dosing Log |
| | 16.2.3.1.3 | Sunitinib Dosing Log | Sunitinib Study Drug Dosing Log |
| | 16.2.3.2 | Study Drug Accountability | Drug Accountability |
| | 16.2.3.3.1 | PLX9486 and Overall Exposure | Derived |
| | 16.2.3.3.2 | PLX3397 Exposure | Derived |
| | 16.2.3.3.3 | Sunitinib Exposure | Derived |
| 16.2.4 | | Individual efficacy response data | |
| | 16.2.4.1 | Tumor Assessment (Target Lesions) | Tumor Evaluation - Target Lesions |
| | 16.2.4.2 | Tumor Assessment (Non-Target Lesions) | Tumor Evaluation - Non-Target Lesions Baseline;<br>Tumor Evaluation - Non-Target Lesions |
| | 16.2.4.3 | Tumor Assessment (New Lesions) | Tumor Evaluation - New Lesions |
| | 16.2.4.4 | Tumor Response Assessment (Target and Non-Target Lesions) | Tumor Response Assessment |
| | 16.2.4.5 | Derived Efficacy Endpoints Based on Tumor<br>Response | Derived |
| 16.2.5 | | Adverse Events Listings | |
| | 16.2.5.1 | Adverse Events | Adverse Events |
| | 16.2.5.2 | Adverse Events Leading Changes in Study<br>Treatment | Adverse Events; Study Exit Status; End of Treatment |
| | 16.2.5.3 | Dose Limiting Toxicity | Dose Limiting Toxicity |
| | 16.2.5.4 | Adverse Events Leading to Death | Adverse Events; Death Detail |
| 16.2.6 | | Individual Laboratory Measurements | |
| | 16.2.6.1.1 | Hematology | Hematology |
| | 16.2.6.1.2 | Hematology – Other Tests | Hematology |
| | 16.2.6.1.3 | Hematology Laboratory Results - Grade 3 or Higher | Hematology |
| | 16.2.6.2.1 | Chemistry | Chemistry |
| | 16.2.6.2.2 | Chemistry – Other Tests | Chemistry |
| | 16.2.6.2.3 | Chemistry Laboratory Results - Grade 3 or Higher | Chemistry |
| | 16.2.6.3.1 | Urinalysis | Urinalysis |
| | 16.2.6.3.2 | Urinalysis – Other Tests | Urinalysis |
| | 16.2.6.4.1 | Coagulation | Coagulation |
| | 16.2.6.4.2 | Coagulation – Other Tests | Coagulation |
| 16.2.7 | | Other Data | |
| | 16.2.7.1 | Vital Signs | Vital Signs |
| | 16.2.7.2 | Physical Examination | Physical Examination |
#### Clinical Study Report PLX121-01

Plexxikon Inc.Statistical Analysis PlanPLX121-0130Jun2020

| | | 12-Lead ECG, Pre and Post Dose 12-Lead ECG, |
|---|---|---|
| | | Post Dose 12-Lead ECG, 12-Lead ECG – 3 |
| 16.2.7.3.1 | 12-Lead Electrocardiogram | Recordings, 12-Lead ECG (Pre/3hr Post Dose), 12- |
| | | Lead ECG (Pre/Post Dose), 12-Lead ECG |
| | | (Pre/3&6hr Post Dose) 3 Recordings |
| | | 12-Lead ECG, Pre and Post Dose 12-Lead ECG, |
| | Electrocardiogram - Patients with Outlier QTc | Post Dose 12-Lead ECG, 12-Lead ECG – 3 |
| 16.2.7.3.2 | Values | Recordings, 12-Lead ECG (Pre/3hr Post Dose), 12- |
| | values | Lead ECG (Pre/Post Dose), 12-Lead ECG |
| | | (Pre/3&6hr Post Dose) 3 Recordings |
| 16.2.7.4 | ECOG Performance Status Assessment | Physical Examination |
| 16.2.7.5 | Echocardiogram/MUGA Scan | Echocardiogram/MUGA Scan |
| 16.2.7.6 | Thyroid Stimulating Hormone (TSH) Level | Thyroid Stimulating Hormone (TSH) Level |
| 16.2.7.7 | Pregnancy Test | Pregnancy Test |
| 16.2.7.8.1 | Circulating DNA | Circulating DNA |
| 16.2.7.8.2 | Tumor Markers | Tumor Markers |
| 16.2.7.8.3 | Archival Tumor Tissue Collection | Archival Tumor Tissue Collection |
| 16.2.7.8.4 | Optional Paired Tumor Biopsy | Optional Paired Tumor Biopsy |

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan

### Appendix B: Table Layouts

### Notes to programmer:

specified otherwise in the mocks. For an example of a mock with all the study parts, see Table 14.1.1 – Summary of Patient Disposition. Study Parts to be presented Sponsor, protocol, and footnotes will appear on all pages of all Study Parts. For all tables, the mock shells outline layout for Study Part 1 – Dose Escalation Study Parts (Single-Agent PLX9486) if the layout is the same for all study parts. The remainder of the table will follow the same format for other Study Parts, unless

### Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486)

Column headers under Study Part 1 are: '250 mg QD PLX9486', '350 mg QD PLX9486', '500 mg QD PLX9486', '1000 mg QD PLX9486', '500 mg BID PLX9486', 'Total'

## Study Part 2b - Dose Extension Study Parts (PLX9486 Combined with PLX3397)

Column headers under Study Part 2b are:

500 mg QD PLX9486 + 600 mg PLX3397 fasting', '500 mg QD PLX9486 + 600 mg PLX3397 non-fasting', 'Total'

## Study Part 2e - Dose Extension Study Parts (PLX9486 Combined with Sunitinib)

Column headers under Study Part 2e are:

'500mg QD PLX9486 + 25mg Sunitinib', '1000mg PLX9486 + 25 mg Sunitinib', '1000mg PLX9486 + 37.5 mg Sunitinib', 'Total'

Overall (Study Part 1, 2b and 2e)

Column header under Overall is 'Total'

Note that the Overall part contains only 1 column, column 'Total'

- (2) To present the results of xx (xx.x), if the count is 0, do not include the percent information, i.e. only present 0.
  - (3) When the percentage is 100%, display the result as "100", no decimal place, e.g. xx (100)
- (4) Means and medians will be presented to one more decimal place than the raw data, and the standard deviations will be presented to two more decimal places than the raw data. (5) If a statistic is missing (e.g. standard deviation is missing when N=1 or 0, Imissing ower/upper bounds for confidence interval), display 'NA' for that statistics in the table and
  - add 'NA = Not Applicable' to the abbreviation footnote (i.e. the last footnote if there is an abbreviation in the table title or body)

PLX9486

Plexxikon Inc. PLX121-01

Protocol PLX121-01

Plexxikon Inc.

Statistical Analysis Plan


Clinical Study Report PLX121-01

Summary of Patient Disposition **Table 14.1.1** All Patients

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | 250 mg QD | | | | |
|---|---|---|---|---|---|
| | ADSL.COHORTN | 350 mg QD | 500 mg QD | : | $Total^{[2]}$ |
| | (N = xx) | (N = xx) | (N = xx) | (N = xx) | (N = xx) |
| Description | n (%) | n (%) | n (%) | n (%) | n (%) |
| Patients Enrolled(1,2) ADSL.ENRLFL=Y | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Safety Population[3] ADSL.SAFFL=Y | XX (XX.X) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| Efficacy Evaluable Population <sup>[4]</sup> ADSL.EEFL=Y | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| Primary Reason for Study Discontinuation[5] ADSL.DCTERM | | | | | |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Clinical Progression | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX)(XX) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XX)(XX) | XX (XX.X) |
| Non-Compliance with Study Treatment | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease (Per RECIST) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| Protocol Deviation | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX(XX.X) | XX(XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

30 patients were planned for Part 2b, Note: The following patients have missing primary reason for study discontinuation: patients ttt, zzz, [1] Per protocol amendment 7, 30 patients were planned for Part 1,

date 

time


<sup>30</sup> patients were planned for Part 2e Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column with reason for discontinuation based upon their second enrollment.

[3] All patients who received study medication.

<sup>[4]</sup> All patients who have taken at least 1 dose of study drug and have had at least 1 post-baseline tumor assessment or who discontinued study medication early due to Clinical Progression or

Progressive Disease (Per RECIST).

[5] Based on primary reason for study completion/discontinuation from Study Exit Status form. Reference: Listing 16.2.1.1.

PLX9486

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01


Protocol PLX121-01

Plexxikon Inc.

Summary of Patient Disposition **Table 14.1.1** All Patients

Study Part 2 ADSL.PARTN=3 and 6

| | | Part 2b <sup>[1]</sup> ADSL.PARTN=3 | |
|---|---|---|---|
| | 500 mg QD PLX9486 + 600 mg<br>PI Y3307 Easting | 500 mg QD PLX9486 + 600 mg 500 mg QD PLX9486 + 600 mg DI X3307 Eacting DI X3307 Man facting | Total[1] |
| | $S_{\text{min}}$ | (N = X) | (N = xx) |
| Description | n (%) ' | n (%) | n (%) |
| Patients Enrolled <sup>[1,2]</sup> ADSLENRLFL=Y | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Safety Population[3] ADSLSAFFI=Y | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Efficacy Evaluable Population <sup>[4]</sup> ADSLEEFL=Y | | | |
| | XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Primary Reason for Study Discontinuation <sup>[5]</sup> ADSL.DCTERM | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adverse Event | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Clinical Progression | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Non-Compliance with Study Treatment | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease (Per RECIST) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Protocol Deviation | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | xx (xx.x) | xx (xx.x) | XX (XX.X) |

30 patients were planned for Part 2b, Note: The following patients have missing primary reason for study discontinuation: patients ttt, zzz, [1] Per protocol amendment 7, 30 patients were planned for Part 1,

date 

time


<sup>&</sup>lt;sup>[2]</sup> Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column. 30 patients were planned for Part 2e

<sup>[3]</sup> All patients who received study medication.

<sup>[4]</sup> All patients who have taken at least 1 dose of study drug and have had at least 1 post-baseline tumor assessment or who discontinued study medication early due to Clinical Progression or Progressive Disease (Per RECIST).

[5] Based on primary reason for study completion/discontinuation from Study Exit Status form.

Reference: Listing 16.2.1.1.

PLX9486

Plexxikon Inc.

PLX121-01

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. Protocol PLX121-01


Clinical Study Report PLX121-01

PLX121-01

Table 14.1.1 Summary of Patient Disposition All Patients

Study Part 2 ADSL.PARTN=3 and 6

| | | Part 2e AD | Part 2e ADSL.PARTN=6 | |
|---|---|---|---|---|
| | 500 mg QD PLX9486 + 25 | 1000mg PLX9486 + 25 m | 500 mg QD PLX9486 + 25 1000mg PLX9486 + 25 mg 1000mg PLX9486 + 37.5 | |
| | mg Sunitinib | Sunitinib | mg Sunitinib [1] | $Total^{[1]}$ |
| | (N = xx) | (N = xx) | (N = xx) | (N = xx) |
| Description | n (%) | n (%) | n (%) | n (%) |
| V - 13 I A PRI ENDIEI - V | | ` | ` | ` |
| Patients Enrolled [142] Abstractor 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Safety Population <sup>[3]</sup> ADSL.SAFFI.=Y | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Efficacy Evaluable Population <sup>[4]</sup> ADSLEEFL=Y | | | | |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Primary Reason for Study Discontinuation <sup>[5]</sup> ADSL.DCTERM | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Adverse Event | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Clinical Progression | XX (XX.X) | xx(xx.x) | XX (XX.X) | XX (XX.X) |
| Death | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Non-Compliance with Study Treatment | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Physician Decision | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progressive Disease (Per RECIST) | XX (XX.X) | XX(XX.X) | XX (XX.X) | XX (XX.X) |
| Protocol Deviation | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| Other | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) |

Note: The following patients have missing primary reason for study discontinuation: patients ttt, zzz, [1] Per protocol amendment 7, 30 patients were planned for Part 1,

30 patients were planned for Part 2b,

30 patients were planned for Part 2e Part 1 Completed their initial enrollment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column.

[3] All patients who received study medication.

14] All patients who have taken at least 1 dose of study drug and have had at least 1 post-baseline tumor assessment or who discontinued study medication early due to Clinical Progression or Progressive Disease (Per RECIST).

[5] Based on primary reason for study completion/discontinuation from Study Exit Status form. Reference: Listing 16.2.1.1.

 
time


Plexxikon Inc. PLX121-01

Statistical Analysis Plan


Clinical Study Report PLX121-01

Summary of Patient Disposition

Plexxikon Inc. Protocol PLX121-01

**Table 14.1.1** All Patients

Overall (Study Parts 1, 2b and 2e) ADSL.PARTN=1,3,6

| | Total <sup>[1]</sup> |
|---|---|
| | $(\mathbf{x} = \mathbf{x})$ |
| Description | n (%) |
| Patients Enrolled <sup>[1,2]</sup> ADSL.ENRIFE=Y | XX (XX.X) |
| Safety Population <sup>[3]</sup> ADSL-SAFIL=Y | |
| Efficacy Evaluable Population <sup>[4]</sup> ADSL-EFFI.=Y | |
| | XX (XX.X) |
| Primary Reason for Study Discontinuation <sup>[5]</sup> ADSLDCTERM | |
| Adverse Event | XX (XX.X) |
| Clinical Progression | XX (XX.X) |
| Death | XX (XX.X) |
| Lost to Follow-up | XX (XX.X) |
| Non-Compliance with Study Treatment | XX (XX.X) |
| Physician Decision | XX (XX.X) |
| Progressive Disease (Per RECIST) | XX (XX.X) |
| Protocol Deviation | XX (XX.X) |
| Study Terminated by Sponsor | XX (XX.X) |
| Withdrawal by Patient | XX (XX.X) |
| Other | XX (XX.X) |

30 patients were planned for Part 2b, Note: The following patients have missing primary reason for study discontinuation: patients ttt, zzz, [1] Per protocol amendment 7, 30 patients were planned for Part 1, and 30 patients were planned for Part 2e

12 Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column. <sup>[3]</sup> All patients who received study medication.

[4] All patients who have taken at least 1 dose of study drug and have had at least 1 post-baseline tumor assessment or who discontinued study medication early due to Clinical Progression or

Progressive Disease (Per RECIST).

[5] Based on primary reason for study completion/discontinuation from Study Exit Status form. Reference: Listing 16.2.1.1.

date 

time


Statistical Analysis Plan 01Jul2020


Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01

Table 14.1.2
Summary of Demographic and Baseline Characteristics
Safety Population ADSL.SAFFL=Y

| ## ADSL_SEX Ints ADSL_ETHNIC Ints ADSL_ETHNIC IN | Description | Part I $(N = xx)$ $(n \%)$ | Part 2b $ (N = x) $ $ (n \%) $ | Part 2e $(N = xx)$ $(n \%)$ | Overall [3] $(N = xx)$ $(n %)$ | 1 |
|---|---|---|---|---|---|---|
| xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxxx) x | Mean Age of Patients (years) [1] ADSLAGE | XXX | XX.X | XX.X | XX.X | |
| SL.ETHNIC xx (xx.x) xx (xx.x) xx (xx.x) | Sex of Patients ADSL.SEX<br>Female | (X.XX) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| acific Islander | Male | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| T XX (XX.X) XX (XX.X) XX (XX.X) | Race of Patients [2] ADSL.RACE | | | | | |
| T | White | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) | |
| T | Black or African American | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) | |
| XX (XX.X) XX (XX.X) XX (XX.X) | Native Hawaiian or Other Pacific Islander | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) | Asian | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) xx (xx,x) | American Indian or Alaska Native | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | Multiple | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Unknown | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Ethnic Origin of Patients ADSL.ETHNIC | | | | | |
| xx(x.x) $xx(x.x)$ $xx(x.x)$ $xx(x.x)$ $xx(x.x)$ $xx(x.x)$ | Not Hispanic or Latino | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| xx(xx,x) $xx(xx,x)$ $xx(xx,x)$ | Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | |
| | Unavailable | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) | |

Note: N = the number of patients assigned to the cohort.
[1] Age is calculated as of the date the informed consent is signed as (Date informed consent signed minus the date of birth (in days) divided by 365.25) rounded down to the closest year.

[2] Patients could mark more than one race.

[3] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column.

Reference: Listing 16.2.2.1.

time

date 

Plexxikon Inc.

PLX121-01

Statistical Analysis Plan

Plexxikon Inc. Protocol PLX121-01


Safety Population ADSL.SAFFL=Y Summary of Medical History **Table 14.1.3** 

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | 4 | | | | |
|---|---|---|---|---|---|
| | 250 mg QD | | | | Ē |
| | ADSL.COHORTN | 350 mg QD | 500 mg QD | : | Total [1] |
| | (N = xx) | (N = xx) | (N = xx) | (N = xx) | (N = xx) |
| Body System ADMH.MHCAT | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ears/Nose/Throat | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cardiovascular | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Respiratory | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Dermatological | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Musculoskeletal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Gastrointestinal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Endocrine/Metabolic | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Hepatic | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Lymphatic | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Immunological | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Neurological | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Genitourinary/Reproductive | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Psychiatric | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) |

Note: Patients could mark more than one body system.

time

date

### Programming note:

- Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column. 1) Repeat for Study Part 2b, Study Part 2e, Overall (ADSL.PARTN=2, PARTN=3 for overall PARTN=1,3,6)
  2) Include index [2] on column hondore 500 mm PID in Dand 1 500 mm PID in CIP NEW 1.5.6)


<sup>&</sup>lt;sup>[1]</sup> Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column.

Reference: Listing 16.2.2.2

Clinical Study Report PLX121-01

Statistical Analysis Plan

Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01


#### Summary of Prior Medications ADCM.PRIORFL=Y Safety Population ADSL.SAFFL=Y **Table 14.1.4**

## Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| ATC Class /<br>Generic Drug Name | 250 mg QD ADSL.COHORTN (N = xx) n (%) | 350 mg QD<br>(N = xx)<br>n (%) | 500 mg QD<br>(N = xx)<br>n (%) | (xx = N) u (%) u | Total [1] $(N = xx)$ $n (\%)$ |
|---|---|---|---|---|---|
| Patients Receiving any Prior Medications ADCM.PMANYFL | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC Class 1 ADCM.PMATCFL Generic Drug Name 1 ADCM.PMGENFL Generic Drug Name 2 | XX (XX.X) | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| ATC Class 2 Generic Drug Name 1 Generic Drug Name 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Prior medications are those that begin prior to the administration of study drug, even if they continue after dosing.

[1] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the Note: Patients could report multiple medications; at each level of summation (overall, ATC class, generic drug name), patients reporting more than one medication are counted only once. cohorts they enrolled in; however, the patients are only counted once in the Overall column. Reference: Listing 16.2.2.5

date 

time

Programming note:

Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column. Repeat for Study Part 2b, Study Part 2e, Overall (ADSL\_PARTN=2, PARTN=3 for overall PARTN=1,3,6)
 Include index [2] on column headers 500 mg BID in Part 1. 500 mσ OD PLX948κ ± 600 mσ PI Y3307 ξ-...


Plexxikon Inc.


Clinical Study Report PLX121-01

Statistical Analysis Plan


Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01

Summary of Concomitant Medications ADCM.CONCOMFL=Y Safety Population ADSL.SAFFL=Y **Table 14.1.5** 

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| ATC Class ADCM.CMCLAS /<br>Generic Drug Name ADCM.CMDECOD | 250 mg QD ADSL.COHORTN ( $N = xx$ ) $n (\%)$ | 350 mg QD<br>(N = xx)<br>n (%) | 500 mg QD<br>(N = xx)<br>n (%) | (xx = N) (%) u | Total [1] (N = xx) n (%) |
|---|---|---|---|---|---|
| Patients Receiving any Concomitant Medications ADCM.CMANYFL | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| ATC Class 1 ADCM.CMATCFL Generic Drug Name 1 ADCM.CMGENFL Generic Drug Name 2 | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xxx) | xx (xx.x) |
| | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xxx) | xx (xx.x) |
| | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ATC Class 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Generic Drug Name 1 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Generic Drug Name 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Concomitant medications are those which are taken at any time between the date of first dose and the date of last dose of any study medication. In cases where it is not possible to determine if a medication is concomitant, the medication is classified as concomitant.

Note: Patients could report multiple medications; at each level of summation (overall, ATC class, generic drug name), patients reporting more than one medication are counted only once

Note: Concomitant medications are coded according to the 01 March, 2015 WHODrug Dictionary.

[1] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column. Reference: Listing 16.2.2.5

time

date 

### Programming note:

- Repeat for Study Part 2b, Study Part 2e, Overall (ADSL.PARTN=2, PARTN=3 for overall PARTN=1,3,6).
- Order by descending count of the Overall summary ATC and by descending count of generic drug name within ATC class in the Overall summary. Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column. 357


PLX9486

Statistical Analysis Plan

Plexxikon Inc. PLX121-01

Protocol PLX121-01 Plexxikon Inc.


### Best Overall Tumor Response ADRS.PARAMCD=CBEST Efficacy Evaluable Population ADSL.EEFL=Y **Table 14.2.1**

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | 250 mg QD ADSL.COHORTN (N = xx) $n (\%)$ Response Rate 95% ( | g QD<br>hHORTN<br>xx)<br>%0<br>95% C.I <sup>[3]</sup> | 350 mg QD $(N = xx)$ $n (\%)$ Response Rate 95 | g QD<br>: xx)<br>%)<br>95% C.I <sup>[3]</sup> | (N = xx) n (%) Response Rate | . xx)<br>%)<br>95% C.I <sup>[3]</sup> | Total[4] $(N = xx)$ $n (%)$ $n (%)$ Response Rate | 1[4]<br>xx)<br>%)<br>95% C.I [3] |
|---|---|---|---|---|---|---|---|---|
| Best Overall Tumor Response [1] | | | | | | | | |
| Complete Response (CR) | u (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | (%) u | xx.x%, xx.x% |
| Partial Response (PR) | n (%) | xx.x%, xx.x% | n (%) | XX.X%, XX.X% | n (%) | xx.x%, xx.x% | n (%) | XX.X%, XX.X% |
| Stable Disease (SD) | n (%) | XX.X%, XX.X% | n (%) | XX.X%, XX.X% | n (%) | xx.x%, xx.x% | n (%) | XX.X%, XX.X% |
| Progressive Disease (PD) | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% |
| Not Evaluable (NE) | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% |
| Not Done [2] | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% |
| Best Overall Response Rate (CR or PR) | n (%) | xx.x%, xx.x% | n (%) | xx.x%, xx.x% | (%) u | xx.x%, xx.x% | n (%) | xx.x%, xx.x% |
| Best Clinical Benefit Rate (CR, PR or SD at 16 weeks) | u (%) | xx.x%, xx.x% | u (%) | xx.x%, xx.x% | u (%) | xx.x%, xx.x% | u (%) | xx.x%, xx.x% |

<sup>[1]</sup> Response based on RECIST (Response Criteria Evaluation in Solid Tumors) guideline (version 1.1), with confirmation of CR and PR required.

time date

### Programming note:

- Repeat for Study Part 2b, Study Part 2e, Overall (ADSL.PARTN=2, PARTN=3 for overall PARTN=1,3,6)
- Include index [4] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column. 7 7
  - For the BOR analysis only include re-enrolled patients in the initial cohort they enrolled in. Do not include them in the Part 2e analysis or the Overall analysis.


<sup>&</sup>lt;sup>[2]</sup> Three patients withdrew from the trial due to clinical progression without having a post-baseline scan. They are included in this row. <sup>[3]</sup> The CI is the two-sided exact binomial 95% Confidence Interval.

<sup>[4]</sup> Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. BOR for re-enrolled patients is included in their initial cohort analysis and the Overall analysis but not in the Part 2e analysis. Reference: Listing 16.2.4.4

Clinical Study Report PLX121-01

Statistical Analysis Plan


Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01

Duration of Response ADTTE.PARAMCD=DOR **Table 14.2.2** 

Efficacy Evaluable Population ADSL.EEFL=Y

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

xxx [xxx, xxx] xxx [xxx, xxx] xxx [xxx, xxx] XX.X - XX.X $Total^{[2]}$ (X = XX)n (%) n (%) n (%) XXX [XXX, XXX] XXX [XXX, XXX] xxx [xxx, xxx] XX.X - XX.XXX.X - XX.X(N = xx)n (%) n (%) u (%) xxx [xxx, xxx] xxx [xxx, xxx] xxx [xxx, xxx] 500 mg QD XX.X - XX.X(N = xx)u (%) n (%) xxx [xxx, xxx] xxx [xxx, xxx] xxx [xxx, xxx] 350 mg QD XX.X - XX.X(N = xx)n (%) n (%) (%) u ADSL.COHORTN xxx [xxx, xxx] xxx [xxx, xxx] xxx [xxx, xxx] 250 mg QD XX.X - XX.XXX.X - XX.X(N = xx)n (%) n (%) n (%) Number of responders who progressed or died [ n (%)] Number of responders who did not progress or die (censored) [ n (%)] Range of DOR (All patients who Progressed or Died) Range of DOR (All patients with response) Percentiles [95% CI] of DOR (days)[1] Total number of responders [ n (%)] Median

Note: DOR is calculated for every patient with a response to therapy as the number of days from the date of initial response (PR or CR) to the date of first documented disease progression or death, whichever occurs first. If disease progression or death does not occur, DOR is censored as of the date of their last post-baseline tumor response evaluation. Patients without a tumor response Note: Responders are patients with best overall response of CR or PR. Response based on RECIST guideline (version 1.1), with confirmation of CR or PR required. evaluation after responding to therapy have their event censored on the day after response with a duration of one day.

[1] Kaplan-Meier product-limit estimates.

121 Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. DOR for re-enrolled patients is included in their initial cohort analysis and the Overall analysis but not in the Part 2e analysis.

CR = Complete Response; DOR = Duration of Response; N/A = Not Applicable; PR = Partial Response; NE = Not Estimable.

Reference: Table 14.3.2.1, Listings 16.2.4.5

date 

time

### Programming note:

- Repeat for Study Part 2b, Study Part 2e, Overall (ADSL.PARTN=2, PARTN=3 for overall PARTN=1,3,6) 7
- Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column.
  - For the DOR analysis only include re-enrolled patients in the initial cohort they enrolled in. Do not include them in the Part 2e analysis or the Overall analysis.


Plexxikon Inc.


Clinical Study Report PLX121-01

Statistical Analysis Plan

Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01


Progression-Free Survival ADTTE.PARAMCD=PFS Efficacy Evaluable Population ADSL.EEFL=Y **Table 14.2.3** 

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | 250 mg QD<br>ADSL.COHORTN<br>(N = xx) | 350 mg QD<br>(N = xx) | 500 mg QD<br>(N = xx) | <br>(X = N) | $Total^{[2]}$ $(N = xx)$ |
|---|---|---|---|---|---|
| Number of patients who progressed or died [n (%)] | n (%) | n (%) | n (%) | n (%) | n (%) |
| Number of patients who did not progress or die (censored) [n (%)] | n (%) | n (%) | n (%) | n (%) | n (%) |
| Percentiles [95% CI] of PFS (days) <sup>[1]</sup> 25th Median 75th | xxx [xxx, xxx] | XXX [XXX, XXX] | xxx [xxx, xxx] | XXX [XXX, XXX] | xxx [xxx, xxx] |
| | xxx [xxx, xxx] | XXX [XXX, XXX] | xxx [xxx, xxx] | XXX [XXX, XXX] | xxx [xxx, xxx] |
| | xxx [xxx, xxx] | XXX [XXX, XXX] | xxx [xxx, xxx] | XXX [XXX, XXX] | xxx [xxx, xxx] |
| Range of PFS for all patients (days) Range of PFS for patients who progressed or died (days) | XX.X - XX.X | XX.X — XX.X | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| | XX.X - XX.X | XX.X — XX.X | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| 6-month PFS <sup>[1]</sup> Percent [95% CI] CALCULATED FROM PROC LIFETEST ADTTE.PARAM="PFS" estimated at 6 months | xxx [xxx, xxx] | xxx [xxx, xxx] | xxx [xxx, xxx] | xxx [xxx, xxx] | xxx [xxx, xxx] |

Note: PFS is defined as the number of days from the start of therapy (i.e., CIDI) to the date of first documented disease progression/relapse or death, whichever occurs first. If disease progression/relapse/death does not occur, PFS is censored as of the date of their last evaluable tumor assessment.

<sup>[1]</sup> Kaplan-Meier product-limit estimates. The 6-month time point is defined as 180 days for this analysis.

[2] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. PFS for re-enrolled patients is included in their initial cohort analysis and the Overall analysis but not in the Part 2e analysis. Reference: Table 14.3.2.1, Listings 16.2.4.5

time

date Programming note:

- Repeat for Study Part 2b, Study Part 2e, Overall (ADSL.PARTN=2, PARTN=3 for overall PARTN=1,3,6).
- Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column.
  - For the PFS analysis only include re-enrolled patients in the initial cohort they enrolled in. Do not include them in the Part 2e analysis or the Overall analysis.


Plexxikon Inc.


| PLX9486 |
|---------|

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

Repeat Table 14.2.3 shell for:

## Table 14.2.4, Overall Survival, Efficacy Evaluable Population ADTTE.PARAM=SURV

### Programming note:

- Update footnote [1] to be "Kaplan-Meier product-limit estimates. The 12-month time point is defined as 365 days for this analysis.".
  Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Replace 6-month PFS with 12-month OS, CALCULATED FROM PROC LIFETEST ADTTE.PARAM="SURV" estimated at 12 months.
   Update footnote [1] to be "Kaplan-Meier product-limit estimates. The 12-month time point is defined as 365 days for this analysis.".
   Include index [2] on column headers 500 mg RID in Part 1 500 mg Or DIVAGO.
- For the OS response re-enrolled patients will have their OS calculated only for their initial cohort, however OS will use the stop date from the second cohort as this is an indication of survival. OS for re-enrolled patients is included in their initial cohort analysis and the Overall analysis but not in the Part 2e analysis. Sunitinib and the Total columns in Part 2e, and the Overall column. 4

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

 Plexxikon Inc. Pa Protocol PLX121-01

Plexxikon Inc.

PLX121-01

### Overall Summary of Treatment-Emergent Adverse Events ADAE.TRTEMFL=Y Safety Population ADSL.SAFFL=Y Table 14.3.1.1

## Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| Adverse Event Category | 250 mg QD ADSL.COHORTN (N = xx) n (%) | 350 mg QD (N = xx) $n (\%)$ | 500 mg QD $(N = xx)$ $n (\%)$ | (N = xx) $n (%)$ | Total[2] $(N = xx)$ $n (%)$ |
|---|---|---|---|---|---|
| Total Number of TEAEs | X | XX | XX | XX | XX |
| Patients with at least one TEAE | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients with at least one TE SAE ADAE.AESER=Y | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients with at least one Related TEAE $^{[1]}$ ADAE.AREL | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients with at least one Related TE SAE <sup>[1]</sup> ADAE.AESER,ADAE.AREL | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patients with at lease one TEAE leading to any changes in study treatment ADAE.TEIRWFL | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients with at least one TEAE leading to permanent withdrawal of study product or discontinuation from the study ADAE.TEWDFL | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) |

Note: Patients could report multiple events; for each summation, patients reporting more than one event are counted only once.

Reference: Listing 16.2.5.1

time date 

Programming note:

1) Include index [1] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column.


SAE = Serious Adverse Event; TE = Treatment-Emergent; TEAE = Treatment-Emergent Adverse Event.

<sup>[1]</sup> Relatedness refers to any TEAEs reported as "Possibly Related" or "Probably Related" to any study treatment the patient received.

<sup>[2]</sup> Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column.

PLX9486

Plexxikon Inc.

PLX121-01

Statistical Analysis Plan


Protocol PLX121-01 Plexxikon Inc.

Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term ADAE.TRTEMFL=Y Safety Population ADSL.SAFFL=Y **Table 14.3.1.2** 

| | | | ADSL.P4 | ADSL.PARTN, COHORTN | RTN, COHORTN | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Part 1 | | | Pa | Part 2b | | Part 2e | | |
| Treatment-Emergent Adverse | | | | 1000 mg | | 500 mg QD<br>PLX9486 + 600 | 500 mg QD<br>PLX9486 + 600 | 500 mg QD 1<br>PLX9486 + | 1000 mg QD<br>PLX9486 + | 1000 mg QD<br>PLX9486 + | |
| Events <sup>[1]</sup> | 250 mg QD | 250 mg QD 350 mg QD | 500 mg QD | _<br>(D) | 500 mg BID | 7 | mg PLX3397 non- | 25 mg | 25 mg | 37.5 mg | |
| System Organ Class | PLX9486 | PLX9486 PLX9486 | PLX9486 | PLX9486 | $PLX9486^{[2]}$ | $fasting^{[2]}$ | fasting | Sunitinib | Sunitinib | Sunitinib <sup>[2]</sup> | Overall $^{[2]}$ |
| ADAE.AEBODSYS / | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) |
| Preferred Term ADAE.AEDECOD | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | u (%) | n (%) |
| Patients Reporting at Least One | (x.xx) xx (x.xx) xx | XX (XX.X) | XX (XX.X) | (x,x) | (XXX) XX | (XXX) XX | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | (XXX) XX |
| TEAE | | | | | | | | | | | |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: N = the number of patients assigned to the cohort.

Note: TEAEs are those with start dates on or after the treatment start date. Treatment start date is the earliest dose date of any of the study drugs (PLX9486, PLX3397, and sunitinib), including dose date of the run-in PK period. The TEAEs of patients who escalated to a higher dose are classified according to the patient's initial dose cohort.

Note: The denominator for the percentages is the number of patients (N) in the Safety Population.

Note: Adverse Events are coded using MedDRA v 23.0.

Note: System organ classes are listed in descending order based on the Total column; within each system organ class, preferred terms are listed in descending order based on the Total column. 111 At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once.

121 Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2b. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column.

MedDRA = Medical Dictionary for Regulatory Activities; TEAE = Treatment-Emergent Adverse Event. Reference: Listing 16.2.5.1

time date 

Programming note:

1) Sort by descending SOC and PT within PT.


Clinical Study Report PLX121-01

Statistical Analysis Plan

Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01


### Summary of Treatment-Emergent Adverse Events by Preferred Term and Severity Grade ADAE.TRTEMFL=Y Safety Population ADSL.SAFFL=Y Table 14.3.1.3

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | 250 mg QD | ďδ | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ADSL.COHOR | IORTN | 350 mg QD | g QD | 500 mg QD | g QD | 1000 mg QD | ıg QD | $500 \text{ mg BID}^{[2]}$ | $BID^{[2]}$ | $Total^{[2]}$ | [2] |
| | (N=1) | ) | (N = N) | = ) | (N=) | ( = | (N = 1) | = ) | (=N) | <u> </u> | (N = 1) | = ) |
| | | ADAE. | | | | | | | | | | |
| | | GK3ANYF<br>L=Y | | | | | | | | | | |
| | Any Grade | CTCAE | | CTCAE | | CTCAE | | CTCAE | | CTCAE | | CTCAE |
| Preferred Term [n (%)] ADAE.AEDECOD ADAE.ASEV Grade $\geq 3$ Any Grade $\geq 3$ Any Grade Grade $\geq 3$ Any Grade Grade $\geq 3$ Any Grade $\geq 3$ Any Grade Grade $\geq 3$ Any Grade $\geq 3$ Any Grade $\geq 3$ Any Grade $\geq 3$ Any Grade Grade $\geq 3$ Any | ADAE.ASEV | Grade $\geq 3$ | Any Grade | Grade $\geq 3$ | Any Grade | Grade $\geq 3$ | Any Grade | Grade $\geq 3$ | Any Grade | $Grade \ge 3$ | Any Grade | Grade $\geq 3$ |
| Patients Reporting at Least One TEAE | xx (xx.x) | XX (XX.X) | $xx\left(xx.x\right) xx\left(xx.x\right) xx\left$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| Preferred Term 1 | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) $xx(xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) $xx(xx.x)$ $xx(xx.x)$ $xx(xx.x)$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) xx(xx.x) | xx(xx.x) xx(xx.x) | xx (xx.x) | | xx(xx.x) xx(xx.x) | xx (xx.x) | xx (xx.x) |
| ::: | | | | | | | | | | | | |

Note: N = the number of patients assigned to the cohort.

Note: TEAEs are those with start dates on or after the treatment start date. Treatment start date is the earliest dose date of any of the study drugs (PLX9486, PLX3397, and sunitinib), including dose date of the run-in PK period. The TEAEs of patients who escalated to a higher dose are classified according to the patient's initial dose cohort.

Note: The denominator for the percentages is the number of patients (N) in the Safety Population.

Note: Adverse Events are coded using MedDRA v 23.0.

Note: Preferred terms are listed in descending order based on the Total column.

11] At each level of summation (overall and preferred term), patients reporting more than one adverse event are counted only once. cohorts they enrolled in; however, the patients are only counted once in the Overall column.

MedDRA = Medical Dictionary for Regulatory Activities; TEAE = Treatment-Emergent Adverse Event.

Reference: Listing 16.2.5.1

time date 


Clinical Study Report PLX121-01

Statistical Analysis Plan

Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01


### Summary of Treatment-Emergent Adverse Events by Preferred Term and Severity Grade Safety Population Table 14.3.1.3

## Study Part 2b - Dose Extension Study Parts (PLX9486 Combined with PLX3397) ADSL.PARTN=3

| | 500 mg QD PLX9486 + 600 mg | 9486 + 600 mg asting <sup>[2]</sup> | 500 mg QD PI<br>mg PLX3397 | .X9486 + 600<br>7 non-fasting | $Total^{[2]}$ | [2] |
|---|---|---|---|---|---|---|
| | (N = 1) | | (=N) | = | (N = N) | |
| | | CTCAE | | CTCAE | | CTCAE |
| Preferred Term [n (%)] | Any Grade | Grade $\geq 3$ | Any Grade | Any Grade $\Rightarrow 3$ | Any Grade $Grade \ge 3$ | Grade $\geq 3$ |
| Patients Reporting at Least One TEAE | xx (xx.x) | (xxx) xx | xx (xx.x) | (x.xx) xx | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| Preferred Term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term 4 | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: N =the number of patients assigned to the cohort.

Note: TEAEs are those with start dates on orafter the treatment start date. Treatment start date is the earliest dose date of any of the study drugs (PLX9486, PLX3397, and sunitinib), including dose date of the run-in PK period. The TEAEs of patients who escalated to a higher dose are classified according to the patient's initial dose cohort.

Note: The denominator for the percentages is the number of patients (N) in the Safety Population.

Note: Preferred terms are listed in descending order based on the Total column. Note: Adverse Events are coded using MedDRA v 23.0.

[1] At each level of summation (overall and preferred term), patients reporting more than one adverse event are counted only once.

[2] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column.

MedDRA = Medical Dictionary for Regulatory Activities; TEAE = Treatment-Emergent Adverse Event. Reference: Listing 16.2.5.1

time time date date 


Clinical Study Report PLX121-01

Statistical Analysis Plan

Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01


### Summary of Treatment-Emergent Adverse Events by Preferred Term and Severity Grade Safety Population Table 14.3.1.3

Study Part 2e - Dose Extension Study Parts (PLX9486 Combined with Sunitinib) ADAE.PARTN=6

| | $500\mathrm{m}$ | 500 mg QD | 1000 1 | 000 mg QD | 1000 | 000 mg QD | | |
|---|---|---|---|---|---|---|---|---|
| | + 25mg Sunitimi | Sunitinib | + 25mg | - 25mg Sunitinib | +37.5mg | + 37.5mg Sunitinib <sup>[2]</sup> | Total <sup>[2]</sup> | 1[2] |
| | N) | = ) | N) | N = J | (N | (N = ) | : N) | = ) |
| | | CTCAE | | CTCAE | | CTCAE | | CTCAE |
| Preferred Term [n (%)] | Any Grade | Grade $\geq 3$ | Any Grade | Grade $\geq 3$ | Any Grade | Grade $\geq 3$ | Any Grade | Grade $\geq 3$ |
| Patients Reporting at Least One TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | XX (XX.X) | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) |
| Preferred Term 2 | XX (XX.X) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term 3 | XX (XX.X) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Preferred Term 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: N = the number of patients assigned to the cohort.

Note: TEAEs are those with start dates on or after the treatment start date. Treatment start date is the earliest dose date of any of the study drugs (PLX9486, PLX3397, and sunitinib), including dose date of the run-in PK period. The TEAEs of patients who escalated to a higher dose are classified according to the patient's initial dose cohort.

Note: The denominator for the percentages is the number of patients (N) in the Safety Population.

Note: Preferred terms are listed in descending order based on the Total column. Note: Adverse Events are coded using MedDRA v 23.0.

[1] At each level of summation (overall and preferred term), patients reporting more than one adverse event are counted only once.

[2] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column.

MedDRA = Medical Dictionary for Regulatory Activities; TEAE = Treatment-Emergent Adverse Event.

Reference: Listing 16.2.5.1

date date 

time time


Plexxikon Inc.

Statistical Analysis Plan

Clinical Study Report PLX121-01

PLX121-01

Protocol PLX121-01 Plexxikon Inc.


### Table 14.3.1.3 Summary of Treatment-Emergent Adverse Events by Preferred Term and Severity Grade (Safety Population) Safety Population

### Overall (Study Part 1, 2b and 2e) ADSL.PARTN=1,3,6

| | Over | Overall <sup>[2]</sup> |
|--------------------------------------|-----------|------------------------|
| | (=N) | |
| | | CTCAE |
| Preferred Term [n (%)] | Any Grade | Grade $\geq 3$ |
| Patients Reporting at Least One TEAE | XX (XX.X) | xx (xx.x) |
| Preferred Term 1 | XX (XX.X) | XX (XX.X) |
| Preferred Term 2 | XX (XX.X) | XX (XX.X) |
| Preferred Term 3 | XX (XX.X) | XX (XX.X) |
| Preferred Term 4 | XX (XX.X) | xx (xx.x) |

Note: N = the number of patients assigned to the cohort.

Note: TEAEs are those with start dates on orafter the treatment start date. Treatment start date is the earliest dose date of any of the study drugs (PLX9486, PLX3397, and sunitinib), including dose date of the run-in PK period. The TEAEs of patients who escalated to a higher dose are classified according to the patient's initial dose cohort.

Note: The denominator for the percentages is the number of patients (N) in the Safety Population.

Note: Preferred terms are listed in descending order based on the Total column. Note: Adverse Events are coded using MedDRA v 23.0.

[1] At each level of summation (overall and preferred term), patients reporting more than one adverse event are counted only once.

[2] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the

cohorts they enrolled in; however, the patients are only counted once in the Overall column.

MedDRA = Medical Dictionary for Regulatory Activities; TEAE = Treatment-Emergent Adverse Event.

Reference: Listing 16.2.5.1

time time date date 


| thods | |
|------------------|-------|
| ical Me | |
| f Statisti | |
| ion of | |
| Documentation or | |
| 9 Docui | X9486 |
| 16.1.9 I | PLX |

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

Repeat Table 14.3.1.3 shell for:

Table 14.3.1.4.1 Summary of Any Drug-Related Treatment-Emergent Adverse Events by Preferred Term and Severity Grade, Safety Population INCLUDE AE IN TABLE IF EITHER ONE OF ADAE.AREL OR AREL2 OR AREL3 IS RELATED.

Programming note: I) Add the following note: Note: Relatedness refers to any TEAEs reported as "Possibly Related" or "Probably Related" to study treatment.

Table 14.3.1.4.2, Summary of PLX9486-Related Treatment-Emergent Adverse Events by Preferred Term and Severity Grade, Safety Population INCLUDE AE IN TABLE IF AREL=RELATED

### Programming note:

1) Add the following note: Note: Relatedness refers to any TEAEs reported as "Possibly Related" or "Probably Related" to study treatment.


PLX9486

Plexxikon Inc.

PLX121-01

Statistical Analysis Plan

Protocol PLX121-01 Plexxikon Inc.


Summary of Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Relatedness ADAE.TRTEMFL=Y
Safety Population ADSL.SAFFL=Y Table 14.3.1.4.3

ADSL.PARTN, ADSL.COHORTN

| Part 2e | 1000 mg QD PLX9486<br>+ 37 5 mg Sunitinih | (X = X) $(X)$ | Related to | xx (xx.x) | XX (XX.X) XX (XX | $xx(xx.x) \ xx(xx.x) \ xx(xx.x)$ |
|---|---|---|---|---|---|---|
| | 1000 + 35 | F | Related to 9486 | xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | XX (XX.X) |
| | 79486<br>pib | | Related to both | XX (XX.X) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x) |
| Part 2e | 1000 mg QD PLX9486<br>+ 25 mg Sunitinih | (X = X) | elated to Related to Related to 9486 sunitinib both | xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x) |
| | 1000 | F | Related to 9486 | xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x) |
| | .9486<br>nib | | Related to both | xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x) |
| Part 2e | 500 mg QD PLX9486<br>+ 25 mg Sunitinih | (X = X) $(X = X)$ | lated to Related to Related to 9486 sunitinib both ADAE.AR EL3 | xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x) |
| | 500 | ÷ | Related to 9486 | xx (xx.x) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | xx (xx.x) |
| | K9486 | non-rastmg | 3397 both | xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x) |
| Part 2b | 500 mg QD PLX9486<br>+ 600 mg PI X3307 non-fasting | (N = XX) | Related to 3397 | _ | | _ |
| | 500<br>+ 600 ms | 1000 F | Related to 9486 | xx (xx.x) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | xx (xx.x) |
| þ | 500 mg QD PLX9486<br>+ 600 mg PI X3307 fasting | x) | to Related to both A | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | XX (XXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXXX) XX (XXXXXX (XXXXXXX (XXXXXXXX | x) xx (xx) |
| Part 2b | 500 mg QD PLX9486 | (x = N) | Related to Related to 9486 3397 ADAE.A ADAE.A REL2 | .x) xx (xx. | (x) xx (xx.<br>(x) xx (xx.<br>(x) xx (xx. | (x.x) $xx$ $(x.x)$ $xx$ $(x.x)$ $xx$ |
| | _ | | Related 9486<br>ADAE | | | 2 xx (xx. |
| | System Organ Class | Preferred Term | ADAL ALDESON | Patients Reporting at<br>Least One TEAE | System Organ Class 1<br>Preferred Term 1<br>Preferred Term 2 | System Organ Class 2 xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) |

Note: Adverse Events are coded using MedDRA v 23.0.

Note: TEAEs are those with start dates on or after the treatment start date. Treatment start date is the earliest dose date of any of the study drugs (PLX9486, PLX3397, and sunitinib), including dose date of the run-in PK period. The TEAEs of patients who escalated to a higher dose are classified according to the patient's initial dose cohort.

Note: Patients could report multiple events. At each level of summation (overall, system organ class, preferred term), patients reporting more than one adverse event are counted only once. System organ classes are listed in descending order based on the total count; within each system organ class, preferred terms are listed in descending order based on the total count.

Note: The denominator for the percentages is the number of patients (N) in the Safety Population.

[1] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the Note: Relatedness refers to any TEAEs reported as "Possibly Related" or "Probably Related" to Study Treatment. cohorts they enrolled in.

MedDRA = Medical Dictionary for Regulatory Activities; TEAE = Treatment-Emergent Adverse Event. Reference: Listing 16.2.5.1

time

date

Programming note:

1) Split by study part if needed.


| <b>Methods</b> | |
|-----------------|---------|
| atistical 1 | |
| ion of Stati | |
| ocumentation of | |
| 6.1.9 Do | 7010X I |

PLX9486

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

PLX121-01

Plexxikon Inc.

Plexxikon Inc. Protocol PLX121-01


### Listing of Deaths ADSL.DTHDT or DTHCAUS IS NON MISSING Table 14.3.2.1

# DATASETS:ADSL, DD

| | | | DDATPERF DDDTHCRT Cause of Death DDPRCDTH, DDAENO Comments DDCOM | Disease for which Patient was given Study | | SAE: Primary AE number | | Other, Specify: xx |
|---|---|---|---|---|---|---|---|---|
| | | | Cause of | Disease for | Healineil | SAE: Prin | Unknown | Other, Sp |
| | Death Certificate | Obtained? | DDDTHCRT | | Yes/No | | | |
| | Autopsy | Performed? | DDATPERF | | Yes/No | | | |
| | Date of Last Dose | DTHDT/ of PLX9486/Study Performed? Obtained? | Day <sup>[2]</sup> Day | | 08/ | | | |
| | Date of Death | DTHDT/ | | | 88 | | | |
| | | | ARTN TRT01P USUBJID Death Period <sup>[1] DTTPC</sup> Study | During Chida/During Doct | Study Follow-up | | | |
| an | Patient | No. | <b>JSUBJID</b> | | XXXXX | | | |
| ALASEIS:ADSE, DD | Study Planned Patient | Dose | TRT01P ( | 250 mg | PLX9486 | | | |
| MINDE | Study | Part | PARTN | | 1 | | | |

<sup>[1]</sup> Patient Death Period: "During Study" if Death is the reason given for ending treatment on End of Treatment form or for ending study on the Study Exit Status form. Patients that complete treatment and study for any other reason are considered to have died during "Post-Study Follow Up".
[2] Study Day is relative to the date of the first dose of study medication.
[3] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers

time

date

Programmer notes:

- If patient's death was due to a SAE, provide primary AE number in column 'Cause of Death' If death date is partial, add # follows the study day value in column 'Date of Death / Study Day'
- Footnote [3] is only needed if

appear. In which case, place footnote on the Patient No.


Plexxikon Inc.


Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020


Plexxikon Inc. Protocol PLX121-01

Table 14.3.2.2
Listing of Serious Adverse Events ADAE.AESER=Y
Safety Population ADSL.SAFFL=Y

### DATASETS: ADS, ADAE

| | | | | | | | | - | /<br>Relationshin | Action Taken<br>w/· | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned Patien | MedDRA Patient System Organ Class// | // | | Start Date | | | Severity t<br>(CTCAE | Severity to: PLX9486/ PLX9486/<br>(CTCAE PLX3397/ PLX3397/ | PLX9486/<br>PLX3397/ | Severity to: PLX9486/ PLX9486/ (CTCAE PLX3397/ PLX3397/ Other Action | |
| Study Part | Dose No. | No. Preferred Term | Verbatim Term | AE# | AE# (Study Day) End Date SeriousDLT Grade) | End Date S | erionsDLT | Grade) | Sunitinib- | Sunitinib Taken | Taken | Outcome |
| _ | XXXX | xxxx Respiratory, thoracic ACUTE and mediastinal HYPOX disorders//Acute RESPIR. respiratory failure FAILUR | : ACUTE<br>HYPOXIC<br>RESPIRATORY<br>FAILURE | 27 | (351) | | Yes | Grade 4 | Unlikely\ I<br>Possibly\ F<br>Unlikely\ \ | Drug Permanently Withdrawn/ None/ | Drug Medication, Permanently Hospitalization Withdrawn/ None/ | Medication, Recovered/Resolved<br>Hospitalization |
| | XXXX | xxxx Infections and ALCALIGE infestations//BacterialFAECALIS sepsis SEPSIS | ALCALIGENES<br>alFAECALIS<br>SEPSIS | _ | (8) | | Yes | Grade 3 | Unlikely\ I<br>Possibly\ F<br>Unlikely\ \ | Drug Permanently Withdrawn/ None/ | Drug Medication, Drug Medication, Permanently Hospitalization Withdrawn/None/None | Medication, Recovered/Resolved<br>Hospitalization |
| 2b | XXXX | xxxx Renal and urinary disorders//Renal failure acute | ACUTE<br>KIDNEY<br>INJURY | 6 | (208) | | Yes | Grade 3 | Unlikely\ I<br>Possibly\ 7<br>Unlikely\ \ | Drug<br>Temporarily<br>Withdrawn/<br>None/<br>None | Drug Medication, I<br>Temporarily Hospitalization<br>Withdrawn/<br>None/<br>None | Medication, Recovered/Resolved<br>Hospitalization |
| | XXXX | xxxx Neoplasms benign, malignant and unspecified (incl cysts and polyps)//Renal cell carcinoma | NEW<br>MALIGNANCY<br>- RENAL CELL<br>CARCINOMA | 43 | (1051) | | Yes | Grade 3 | Unlikely\ I Possibly\ Unlikely\ I | Not<br>ed/ | Hospitalization | HospitalizationRecovered/Resolved |

date 

time

Programmer note:

Plexxikon Inc.


<sup>[11]</sup> Study Day is relative to the date of the first dose of study medication.
[22] Not Applicable for Study Parts in study Part 1, relationship to and action take with PLX3397 for Study Parts in study Part 2b, relationship to and action take with sunitinib for Study Parts in study

<sup>(3)</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers AE= Adverse Event; SAE = Serious Adverse Event.

| ethods | |
|--------------|--------|
| tical Mo | |
| f Statis | |
| umentation o | |
| ੁ | , 6 |
| 5.1.9 Do | LX9486 |
| Ť | Ь |

Statistical Analysis Plan 01Jul2020 Clinical Study Report PLX121-01

Remove duplicates from SAE raw dataset. Sort by SAE Case ID within each patient. 5 6 6 6

Plexxikon Inc. PLX121-01

- For column 'Investigator/Reporter...', if one component in the concatenation is missing, display 'Missing' for that component. Footnote [3] is only needed if the listed patient ids appear. In which case, place footnote on the Patient No. Obtain AESTDTC from ADAE by combining raw SAE datset with ADAE by SUBJID and AECASEID

PLX9486

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01


### Summary of Hematology and Coagulation by Cycle and Day Safety Population Table 14.3.4.1.1

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486)

| | | 250 mg OD PLX9486 | PLX9486 | 350 mg OD PLX9486 | PLX9486 | | | Total [1] | 1 [1] |
|---|---|---|---|---|---|---|---|---|---|
| | | $(\mathbf{x} = \mathbf{x})$ $\mathbf{n} (\%)$ | : xx)<br>%) | (N = xx) $n (%)$ | xx)<br>%) | (N = xx) $n (%)$ | (xx) | (N = XX) $n (%)$ | (%) |
| Laboratory Parameter | Time Point | Result | Change from<br>Baseline | Result | Change from<br>Baseline | Result | Change from<br>Baseline | Result | Change from<br>Baseline |
| Hemoglobin (g/dL) | Baseline<br>n<br>Mean (SD)<br>Median<br>Min, Max | n<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | | n<br>XX.X (XX.XX)<br>XX.X<br>XX,X | | n<br>xx.x (xx.xx)<br>xx.x<br>xx,x | | n<br>XX.X (XX.XX)<br>XX.X<br>XX.X | |
| Hematocrit (%) | CxDy n Mean (SD) Median Min, Max Baseline n Mean (SD) | n<br>XX.X (XX.XX)<br>XX.XX<br>XX, XX<br>n<br>XX.X (XX.XX) | n<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | n<br>XX.X (XX.XX)<br>XX.X<br>XX, XX<br>n<br>n<br>XX.X (XX.XX) | n<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | n<br>XX.X (XX.XX<br>XX.X<br>XX, XX<br>n<br>n<br>XX.X (XX.XX) | n<br>xx.x (xx.xx)<br>xx.x<br>xx, xx | n<br>XX.X (XX.XX<br>XX,XX<br>XX,XX<br>n<br>XX,XX | n<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| : | Median<br>Min, Max<br> | XX.X<br>XX, XX | | XX.X<br>XX, XX | | XX.X<br>XX, XX | | XX.X<br>XX, XX | |

WBC (high)[1]

Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug.

[1] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column. The Overall analysis includes the Part 1 or Part 2b result for re-enrolled patients.

Max = Maximum; Min = Minimum; SD = Standard Deviation.


Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

Reference: Listing 16.2.6.1.1

Plexxikon Inc. PLX121-01

date 

#### Programmer notes:

1) Table will continue with hematology parameters including Hematocrit, Hatelets, RBCs, Abs. Neutrophils, Abs. Lymphocytes, Abs. Eosinophils, Abs. Monocytes, Abs. Basophils, etc. (i.e. all the hematology parameters in ADLB), excluding 'Other Tests', followed by coagulation parameters ANC, aPTT, and INR).

time

- Repeat for Parts 2b, 2e and Overall (across all cohorts).
- Include index [1] on column headers 500 mg BID PLX9486 in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column. For the re-enrolled patients, include their initial cohort result (Part 1 or Part 2b) in the Overall summary.
  - 4


PLX9486

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. PLX121-01


Plexxikon Inc. Protocol PLX121-01

Table 14.3.4.1.2
Summary of Hematology and Coagulation – CTCAE Shift from Baseline ADLB.LBCAT=Hematology
Safety Population ADSL.SAFFL=Y

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Grade 0 Grad 0 n (%) n (%) n (%) n (%) n (%) n (%) n (%) | | (XXX) (XXXX) XX (XXXXX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXXX (XXXX) XX (XXXXX (XXXX) XX (XXXXX (XXXXX (XXXXX (XXXXX (XXXXX (XXXX (XXX (XXXX (XXX (XXXX (XXXX (XXXX (XXXX (XXXX (XXX (XX (XXX (XXX (XXX (XX (XXX (XXX (XXX (XXX (XXX (XXX (XX (XXX (XX | XX (XX.X) | | (XXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX) XX (XXXX (XXXX) XX (XXXX) XX (XXXX (XXXX) XX (XXXX (XXXX) XX (XXXX (XXX (XX (XXX (XXX (XX | XX (XX.X) XX (XX | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | $(x \times x) \times (x \times$ | XX (XX.X) XX (XX | (XX.X) XX (XX.X) | | (xx=u) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) vy (vy v) vy (vy v) vy (vy v) vy (vy v) vy (vy v) | $(\lambda\lambda.\lambda) \lambda\lambda (\lambda\lambda.\lambda) \lambda\lambda (\lambda\lambda.$ | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 250 mg QD (N = xx) ADSL.COHORTN Worst Post-Baseline ADI.B.ATOXGR | rade 3 Grade 4<br>1 (%) n (%) | | (n=xx)<br>xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx)<br>xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx)<br>xx (xxx) xx (xxx) xx (xxx) xx (xxx) xx (xxx) | | | XX (XXX) XX (XXXX) XX (XXXXX) XX (XXXXX (XXXXXX (XXXXXXX (XXXXXXX (XXXXXX | | | $(x=x) $ $(x \times x) \times x \times (x \times x) \times (x \times x)$ | (x, x, x) $(x, x, x)$ $(x, x, x)$ | XX (XX.X) XX (XX | $xx \; (xx.x) xx \; (xx.x) xx \; (xx.x) xx \; (xx.x) xx \; (xx.x) \qquad xx \; (xx.x)$ | | XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX | xx (xx.x) xx (xx.x) xx (xx.x) | |
| Lahoratorv Parameter/ | Baseline CTCAE Grade<br>ADLB.BTOXGR | Lahoratory Parameter/ | ANC (10%/L) Grade 0 Grade 1 Grade 2 | Grade 3<br>Grade 4 | Hemoglobin (%) | Grade 0<br>Grade 1 | Grade 2<br>Grade 3 | Grade 4 | WBC (high) <sup>[1]</sup> ADLB.SHIFTI<br>Grade () | Grade 1 | Grade 2<br>Grade 3 | Grade 4 | WBC (low) [1] ADLB.SHIFT2 | Grade 0 | Grade 2 | Grade 3 | A. C. C. |

PLX9486

Plexxikon Inc.

PLX121-01

Statistical Analysis Plan

Clinical Study Report PLX121-01

Note: Lab values are coded using CTCAE v 4.03; Grade 0 indicates normal. CTCAE grading is performed using data values only and does not consider symptomatic criteria.

Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug.

Note: The lower case "n" for a lab parameter is the number of patients in the Study Part who have a baseline and a worst post-baseline CTCAE grade, and it is the denominator for the percentages. [1] High grading is for values increased from normal, low grading is for values decreased from normal.

[2] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column. The Overall analysis includes the Part 1 or Part 2b result for re-enrolled patients. CTCAE = Common Terminology Criteria for Adverse Events.

Reference: Listing 16.2.6.1.1

date 

time

### Programmer note:

Table will continue with hematology parameters given in Section 11.3 of SAP (WBC, hemoglobin, lymphocytes, platelets, ANC, aPTT, and INR).

- Repeat for Parts 2b, 2e and Overall (across all cohorts).
- The following parameters will have a shift table for high and low grading please attach superscript [1] to the parameter name in column 1: WBC, Hemoglobin, and Lymphocytes.
  - Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e, and the Overall column.
    - For the re-enrolled patients, include their initial cohort result (Part 1 or Part 2b) in the Overall summary.


PLX9486

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01


### Table 14.3.4.2.1 Summary of Serum Chemistry by Cycle and Day Safety Population

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486)

| | | 250 mg QD PLX9486 | PLX9486 | 350 mg QD PLX9486 | PLX9486 | | | Total [1] | [1] |
|---|---|---|---|---|---|---|---|---|---|
| | | $(\mathbf{x} = \mathbf{x})$ $\mathbf{n} (\%)$ | (x) | (N = xx) $n (%)$ | xx) %) | (N = xx) $n (%)$ | xx) | (N = xx) $n (%)$ | (xx) |
| Laboratory<br>Parameter | Visit | Result | Change from<br>Baseline | Result | Change from<br>Baseline | Result | Change from<br>Baseline | Result | Change from<br>Baseline |
| Albumin (g/dL) | Baseline | | | | | | | | |
| ) | u | u | | u | | u | | u | |
| | Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | |
| | Median | XX.X | | XX.X | | XX.X | | XX.X | |
| | Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| | CxDy | | | | | | | | |
| | n | п | u | п | п | u | | п | |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | xx.x (xx.xx) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | | XX.X | |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | |
| Alkaline Phosphatase (U/L) Baseline | Baseline | | | | | | | | |
| | u | п | | п | | u | | п | |
| | Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | |
| | Median | XX.X | | XX.X | | XX.X | | XX.X | |
| | Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| | CxDy | | | | | | | | |

Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug.

[1] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column. The Overall analysis includes the Part 1 or Part 2b result for re-enrolled patients.

Max = Maximum; Min = Minimum; SD = Standard Deviation.

Reference: Listing 16.2.6.2.1

date 

time


Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

#### Programmer notes:

- Table will include all serum chemistry parameters -- ALT (SGPT) (U/L), AST (SGOT) (U/L), Blood Urea Nitrogen (BUN), Calcium, Carbon Dioxide, Chloride, Creatinine, Direct Bilirubin, Creatinine Phosphatase, Glucose, LDH, Magnesium, Phosphorus, Potassium, Sodium, Total Bilirubin, Total Protein, Uric Acid, etc. excluding 'Other Tests'. *(*)
  - Repeat for Parts 2b, 2e and Overall (across all cohorts). 36
- Include index [1] on column headers 500 mg BID PLX9486 in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5
  - mg Sunitinib and the Total columns in Part 2e, and the Overall column. For the re-enrolled patients, include their initial cohort result (Part 1 or Part 2b) in the Overall summary. 4


PLX9486

Statistical Analysis Plan


Plexxikon Inc. PLX121-01

Protocol PLX121-01 Plexxikon Inc.

Summary of Serum Chemistry – CTCAE Shift from Baseline ADLB.LBCAT=Chemistry Safety Population ADSL.SAFFL=Y Table 14.3.4.2.2

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.COHORTN

| | | | 250 mg QD | 0 | | | | : | | | | | $Total^{[2]}$ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | (N = XX) | | | | | (N = xx) | | | | | (N = xx) | | |
| | | | n (%) | | | | | n (%) | | | | | n (%) | | |
| Laboratory Parameter/ | Wor | st Post-B | aseline AL | Worst Post-Baseline ADLB.ATOXGR | GR | | Wor | Worst Post-Baseline | eline | | | Wo | Worst Post-Baseline | eline | |
| Baseline CTCAE Grade | Grade 0 Grade 1 Grade 2 | Grade 1 | Grade 2 | | Grade 3 Grade 4 | Grade 0 | Grade 1 | Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 | Grade 3 | Grade 4 | Grade 0 | Grade 1 | Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 | Grade 3 | Grade 4 |
| ADLB.BTOXGR | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| ALT (SGPT) | | | (n=xx) | | | | | (n=xx) | | | | | (n=xx) | | |
| Grade 0 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) | $XX \ (XX.X) \ XX \ (XX.X) \ XX \ (XX.X) \ XX \ (XX.X)$ | (x.xx) xx | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX | xx (xx.x) | XX (XX.X) |
| Grade 1 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) |
| Grade 2 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) |
| Grade 3 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Grade 4 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) |
| AST (SGOT) | | | (n=xx) | | | | | (n=xx) | | | | | (xx=u) | | |
| Grade 0 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | (x.xx) xx | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX | xx (xx.x) | XX (XX.X) |
| Grade 1 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | XX (XX.X) |
| Grade 2 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Grade 3 | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | x (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) | xx (xx.x) | xx (xx.x) | XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) | xx (xx.x) |
| Grade 4 | XX(XX.X) $XX(XX.X)$ $XX(XX.X)$ $XX(XX.X)$ $XX(XX.X)$ | x (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) $xx(xx.x)$ $xx(xx.x)$ $xx(xx.x)$ $xx(xx.x)$ | xx (xx.x) | xx (xx.x) |
| ÷ | | | | | | | | | | | | | | | |

Note: Lab values are coded using CTCAE v 4.03; Grade 0 indicates normal. CTCAE grading is performed using data values only and does not consider symptomatic criteria.

Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug.

Note: The lower case "n" for a lab parameter is the number of patients in the Study Part who have a baseline and a worst post-baseline CTCAE grade, and it is the denominator for the percentages.

[1] High grading is for values increased from normal, low grading is for values decreased from normal.

[2] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2b. These patients are counted in each of the cohorts they enrolled in; however, the patients are only counted once in the Overall column. The Overall analysis includes the Part 1 or Part 2b result for re-enrolled patients.

CTCAE = Common Terminology Criteria for Adverse Events.

Reference: Listing 16.2.6.2.1

date 

time


Statistical Analysis Plan 01Jul2020 Clinical Study Report PLX121-01

#### Programmer notes:

Plexxikon Inc. PLX121-01

- 1) Table will continue with serum chemistry parameters given in Section 11.3 of SAP albumin, ALT, AST, alkaline phosphatase, creatine phosphokinase, creatinine, direct bilirubin, total bilirubin, magnesium, and phosphorus.
  - 36
  - Repeat for Parts 2b, 2e and Overall (across all cohorts).
    Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg
    Sunitinib and the Total columns in Part 2e, and the Overall column.
    For the re-enrolled patients, include their initial cohort result (Part 1 or Part 2b) in the Overall summary.
    - 4


Clinical Study Report PLX121-01

Statistical Analysis Plan


Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01

Summary of PLX9486 Exposure ADEXCOM.PARCAT1=PLX9486 Safety Population ADSL.SAFFL=Y Table 14.3.5.1

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | 250 mg QD | | | | |
|---|---|---|---|---|---|
| | ADSL.COHORTN | 350 mg QD | 500 mg QD | : | $Total^{[3]}$ |
| | (N = xx) | (N = xx) | (N = xx) | (N = xx) | (N = xx) |
| Total Dose Taken ADEXCOM.PARAMN=1 (mg)[1] | | | | | |
| u | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Duration of Treatment (days) ADEACOM: PARAMIN=212 | | | | | |
| u | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X(XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

<sup>[1]</sup> The total dose taken is derived from the duration of treatment (in days) times the assigned dose.

time

date 

### Programmer Note:

- Continue with Study Part 2b, 2e and overall for all parts combined.
- Include index [3] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg

Sunitinib and the Total columns in Part 2e, and the Overall column.

<sup>&</sup>lt;sup>[2]</sup> Duration of treatment is defined as the last dose date of PLX9486 minus the first dose date of PLX9486 plus 1.

<sup>[3]</sup> Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the cohorts they enrolled in; however, the patients are only summarized once in the Overall column with their cumulative exposure across cohorts. Max = Maximum; Min = Minimum; SD = Standard Deviation.

Reference: Listing 16.2.3.3.1

PLX9486

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020


Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01

Table 14.3.5.2 Summary of PLX3397 Exposure ADEXCOM.PARCAT1=PLX3397

Safety Population

Study Part 2b - Dose Extension Study Parts (PLX9486 Combined with PLX3397) PLEASE SEE TABLE 14.3.5.1 ANNOTATIONS

| | mg PLX339/ fasting | mg PLX3397 fasting mg PLX3397 non-fasting | Total |
|---|---|---|---|
| E 4 | (N = xx) | (N = xx) | (N = xx) |
| Total Dose Taken (mg) [1] | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |
| Duration of Treatment (days) <sup>[2]</sup> | | | |
| n | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX |

Programmer Note:

1) Only display Study Part 2b.

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01


### Table 14.3.5.3 Summary of Sunitinib Exposure ADEXCOM.PARCATI=SUNITINIB Safety Population

Study Part 2e - Dose Extension Study Parts (PLX9486 Combined with Sunitinib) PLEASE SEE TABLE 14.3.5.1 ANNOTATIONS

| | 500 mg QD PLX9486+ | 1000 mg QD PLX9486 + | 500 mg QD PLX9486 + 1000 mg QD PLX9486 + 1000 mg QD PLX9486 + | |
|---|---|---|---|---|
| | 25 mg Sunitinib ( $N = xx$ ) | 25 mg Sunitinib $(N = xx)$ | 37.5 mg Sunitinib ( $N = xx$ ) | Total (N = xx) |
| Total Dose Taken (mg) [1] | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |
| Duration of Treatment (days) <sup>[2]</sup> | | | | |
| n | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | XX, XX | XX, XX |

Programmer Note:

1) Only display Study Part 2e.

<sup>&</sup>lt;sup>[1]</sup> The total dose taken is derived from the duration of treatment (in days) times the assigned dose.

<sup>[2]</sup> Duration of treatment is defined as the last dose date of sunitinib minus the first dose date of sunitinib plus 1. Max = Maximum; Min = Minimum; SD = Standard Deviation.

time date
Statistical Analysis Plan 01Jul2020

Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Summary of Vital Signs ADVS.ANL01FL=Y Safety Population ADSL.,SAFFL=Y **Table 14.3.6** 

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | | 250 mg OD ADSL.COHORTN | 3L.COHORTN | 350 mg QD | g QD | : | | Total $(N = xx)^{[1]}$ | $= xx)^{[1]}$ |
|---|---|---|---|---|---|---|---|---|---|
| | | , | (*** | - N- | ( ) ( ) | - 14 | (444 | `` | , (A |
| | | $ \begin{array}{l} \text{(N)} = XX) \\ \text{(N)} \\ \text{(N)} \end{array} $ | (2) | $ \begin{array}{l} \text{(N)} = XX \\ \text{(N)} & \text{(N)} \end{array} $ | (%X) | $ \begin{array}{l} \text{IN} = XX \\ \text{IN} & (\%) \end{array} $ | xx)<br>%) | (%) u | (0) |
| | | Result | Change from Baseline | | Change from | | Change from | | Change from |
| Parameter | Time Point ADVS.AVISIT | ADVS.AVAL | ADVS.CHG | Result | Baseline | Result | Baseline | Result | Baseline |
| Systolic Blood Pressure (mmHg) ADVS.PARAM | | | | | | | | | |
| | u | u | | u | | u | | u | |
| | Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | |
| | Median | XX.X | | XX.X | | XX.X | | XX.X | |
| | Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| | C1D1 – Post-dose | | | | | | | | |
| | u | u | | u | п | u | и | u | |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | |
| | Min, Max | xx, xx | xx, xx | xx, xx | XX, XX | xx, xx | XX, XX | xx, xx | , |
| | : | | | | | | | | |
| Diastolic Blood Pressure (mmHg) | Baseline | | | | | | | | |
| <b>S</b> | n | u | | п | | u | | п | |
| | Mean (SD) | XX.X (XX.XX) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | XX.X | | XX.X | | XX.X | | XX.X | |
| | Min, Max | XX, XX | | XX, XX | | xx, xx | | XX, XX | |

Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug. Some patients enrolled in Part 1 participated in the run in period for the collection of PK samples were treated prior to C1D1 and have a baseline prior to study day 1. These patients have a baseline prior to C1D1 and have change from baseline displayed at C1D1 Pre-Dose.

[1] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the cohorts they enrolled in.

Reference: Listing 16.2.7.1

time

date


## 16.1.9 Documentation of Statistical Methods PLX9486

Statistical Analysis Plan 01Jul2020 Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

- Programmer note:

  I) Table will include the following vital signs: SBP, DBP (mmHg), Heart Rate (bpm), Respiration (breaths/min), Temperature (°C), weight (kg).

  2) Continue with Study Part 2b, and 2e.

  3) Include index [1] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg

  Sunitinib and the Total columns in Part 2e.

16.1.9 Documentation of Statistical Methods

PLX9486

Plexxikon Inc. Protocol PLX121-01 Plexxikon Inc. PLX121-01


Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Table 14.3.7.1
Summary of Electrocardiogram ADEG.ANL01FL=Y
Safety Population ADSL.SAFFL=Y

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486) ADSL.PARTN=1

| | | 250 mg QD AD | QD ADSL.COHORTN | 350 mg QD | g QD | : | | Total [2] | I [2] |
|---|---|---|---|---|---|---|---|---|---|
| | | (N = xx) $n (%)$ | xx)<br>%) | (N = xx) $n (%)$ | xx)<br>%) | (N = xx) $n (%)$ | xx)<br>%) | (N = xx) n (%) | xx)<br>%) |
| ECG Parameter<br>ADEG.PARAM | Time Point ADEG.AVISIT | Result<br>ADEG.AVAL | Change from Baseline ADEG.CHG | Result | Change from<br>Baseline | Result | Change from<br>Baseline | Result | Change from<br>Baseline |
| Ventricular Rate (bpm) | Baseline | | | | | | | | |
| | n | п | | п | | u | | u | |
| | Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | | XX.X (XX.XX) | |
| | Median | XX.X | | XX.X | | XX.X | | XX.X | |
| | Min, Max | XX, XX | | XX, XX | | XX, XX | | XX, XX | |
| | : | | | | | | | | |
| | End of Study | | | | | | | | |
| | d u | ۶ | ۶ | F | £ | = | ۵ | = | £ |
| | M. (CD) | (33, 33) | ("", "") ", "", | (313, 313) | (33, 33) | , | (33, 33) | , | (*** ***) |
| | Median<br>Median | ( | , (, , | (۷۷.۷) | (۷۷.۷) (۷۷.۷) | , (, , | , (, , | (۷۷.۷۷) | (xy.yy)<br>xx x |
| | Min Man | V.V. | V.V. | V.V. | v.v. | V.V. | V.V. | V.V. | V.V. |
| : | иш, иах | үү, үү | XX, XX | үү, үү | xx, xx | үү, үү | νγ, γγ | vy, vy | xx, xx |
| QTcF(msec) | Baseline | | | | | | | | |
| | n | п | | п | | u | | u | |
| | Mean (SD) | XX.X (XX.XX) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | XX.X | | XX.X | | XX.X | | XX.X | |
| | Min, Max | xx, xx | | xx, xx | | xx, xx | | XX, XX | |
| | : | | | | | | | | |
| | End of Study | | | | | | | | |
| | n | п | u | п | u | u | u | u | u |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| : | Upper $95\%~\mathrm{CI}^{[1]}$ | XX.X | | XX.X | | XX.X | | XX.X | |


# 16.1.9 Documentation of Statistical Methods

PLX9486

Plexxikon Inc. PLX121-01

Statistical Analysis Plan

Clinical Study Report PLX121-01

Note: The baseline value is defined as the last non-missing value of the average of the triplicate ECGs prior to the patient's first dose of study drug. Some patients enrolled in Part 1 participated in the run in period for the collection of PK samples were treated prior to CID1 and have a baseline prior to study day 1. These patients have a baseline prior to CID1 and have change from baseline displayed at C1D1 Pre-Dose.

[1] One-sided upper 95% confidence limit.

[2] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2e. These patients are counted in each of the cohorts they enrolled in.

ECG = Electrocardiogram; Max = Maximum; Min = Minimum; SD = Standard Deviation; UCL = Upper Confidence Limit.

Reference: Listing 16.2.7.3.1

date 

## Programmer notes:

Table will continue with the following parameters: PR(msec), QRS(msec), QT(msec), and QTcF(msec) and all scheduled visits in EG/EG1/EG2 datasets. Use derived RR, QTcB, QTcB, QTcF (ADEG.PARAMCD=RRINT, DQTCF, DQTCB) ()

time

- For QTcF an additional row will be added for the one-sided upper 95% confidence interval.
  - Summary statistics for the end of study measurement should be included.
    - For each visit, display all scheduled timepoints in ADEG.
- Continue with Study Part 2b, and 2e.
- Include index [2] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitinib and the Total columns in Part 2e. 25420
- If there are not more than 2 observations in the Total column for a cohort, do not display results for that time point.
  - Record raw values to whole units for min, max, one decimal for mean and median, and 2 decimal places for SD.

16.1.9 Documentation of Statistical Methods PLX9486

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc.

PLX121-01


Summary of Electrocardiogram – Abnormal QTcF Results Safety Population Table 14.3.7.2

# Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486)

| ECG Parameter | 250 mg QD PLX9486<br>(N = xx)<br>n (%) | 350 mg QD PLX9486<br>(N = xx)<br>n (%) | 500 mg QD PLX9486 [3]<br>(N = xx)<br>n (%) | (N = xx) $n (%)$ | Total [3] $(N = xx)$ $n (\%)$ |
|---|---|---|---|---|---|
| QTcF (Fridericia's Method) ≥ 450 msec (for males) [1] ≥ 470 msec (for females) [2] > 500 msec | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| | xx (xx.x) | XX (XX.X) | xx (xx.x) | XX (XX.X) | xx (xx.x) |
| > 30 msec increase from baseline | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| > 60 msec increase from baseline | XX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

Note: Patients experiencing a > 60 msec event are included in the > 30 msec event summary row also.

[1] Denominator is the number of males in Safety Population.

[2] Denominator is the number of females in Safety Population.

[3] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2b. These patients are counted in each of the cohorts they enrolled in.

time

Reference: Listing 16.2.7.3.1 and 16.2.7.3.2

date 

## Programmer notes:

- Continue with Study Part 2b, and 2e.
- Include index [3] on column headers 500 mg BID in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg
  - Sunitinib and the Total columns in Part 2e. Change from baseline incidence is cumulative. That is, a patient who experiences a > 60 msec event is also counted in the > 30 msec event as well.


Plexxikon Inc.


Clinical Study Report PLX121-01


Statistical Analysis Plan

Protocol PLX121-01 Plexxikon Inc.

Plexxikon Inc.

PLX121-01

Summary of ECOG - Shift from Baseline Safety Population **Table 14.3.8** 

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486)

(%) u (%) u n (%) n (%) u (%) n (%) n (%) n n (%) u (%) S (%) u n (%) n n (%) (%) u Baseline ECOG Score n (%) n (%) n (%) n n (%) n (%) n (%) (%) u (%) u n (%) n (%) n u (%) = u) (N = xx)Total [1] (%) u n (%) n (%) n (%) n (%) n (%) n (%) (%) u (%) u n (%) n (%) n n (%) u (%) n (%) n (%) n (%) (%) u n (%) n (%) n n (%) n (%) n n (%) (%) u n (%) С (%) u n (%) n (%) n (%) n (%) n (%) n (%) u (%) u (%) n (%) n u (%) S n (%) n (%) n (%) n (%) n n (%) n (%) n (%) n (%) n (%) n (%) Baseline ECOG Score n (%) n (%) (%) u n (%) n (%) n (%) n (%) n (%) n u (%) n (%) (%) u = u) (N = xx)u (%) n (%) n (%) n (%) n (%) (%) u (%) u n (%) n (%) n n (%) n (%) n (%) n (%) n (%) n (%) (%) u n (%) n n (%) n (%) n (%) n (%) n (%) u (%) n 0 n (%) u (%) u (%) (%) u n (%) n (%) n (%) (%) u n (%) n (%) n n (%) n (%) n (%) 250 mg QD PLX9486 (N = xx)Baseline ECOG Score (%) u n (%) (%) u n (%) n (%) n (%) n (%) (%) u (%) u n (%) n n (%) (%) u (n = n n (%) n (%) (%) u n (%) n (%) (%) u n (%) n (%) n (%) u n (%) (%) u n (%) 10 (%) 10 (%) 10 (%) 10 (%) (%) u n (%) n (%) (%) u (%) u n (%) n n (%) n (%) n (%) n (%) n (%) n (%) n (%) u n (%) n (%) n С Post-Baseline ECOG Score Assessment/ C1D15 C1D8

sedentary nature (e.g., light housework, office work), 2=Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours. 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours, 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair, 5=Dead. Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug. Some patients enrolled in Part 1 participated in the run in period for the collection ECOG Score: 0=Fully active, able to carry on all pre-disease performance without restriction, 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or [1] Two patients who enrolled in Part 2b and one patient who enrolled in Part 1 completed their initial enrolment and subsequently re-enrolled in Part 2c. These patients are counted in each of the of PK samples were treated prior to C1D1 and have a baseline prior to study day 1. These patients have a baseline prior to C1D1 and have change from baseline displayed at C1D1 Pre-Dose. cohorts they enrolled in.

Reference: Listing 16.2.7.4

time

date

Programmer notes:

1) Continue with all study time points and Study Parts 2b, and 2e.


| mentation of Statistical Methods | |
|----------------------------------|---------------------|
| umentation of S | Statistical Methods |
| | umentation of S |

Plexxikon Inc. PLX121-01

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

2) Include index [2] on column headers 500 mg BID PLX9486 in Part 1, 500 mg QD PLX9486 + 600 mg PLX3397 fasting and the Total columns in Part 2b, 1000 mg QD PLX9486 + 37.5 mg Sunitivib and the Total columns in Part 2e.


Statistical Analysis Plan 01Jul2020

Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01

Figure 14.2.1 Progression-Free Survival by Study Part - Study Part 1 (Efficacy Evaluable Population)



Note: PFS is defined as the number of days from the start of therapy (i.e., C1D1) to the date of first documented disease progression / relapse or death, whichever occurs first. If disease progression/relapse or death dose not occur, PFS is censored as of the date of their last evaluable tumor assessment. Reference Table 14.2.3

time

date Programmer notes:

1) Continue with Study Parts 2b, 2e, and Overall.


Plexxikon Inc. PLX121-01

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

Appendix D: Listing Layouts

## Notes to programmer:

# (1) All listings will list Study Parts and planned dose in this order of appearance (for all Study Parts that have data relevant to the listings):

| Study Part | Planned Dose |
|------------|---------------------------------------------------------------|
| 1 | 250 mg QD PLX9486 |
| 1 | 350 mg QD PLX9486 |
| 1 | 500 mg QD PLX9486 |
| 1 | 1000 mg QD PLX9486 |
| 1 | 500 mg BID PLX9486 |
| 2b | 500 mg QD PLX9486 + 600 mg PLX3397 fasting |
| 2b | 500 mg QD PLX9486 + 600 mg PLX3397 non-fasting <sup>[2]</sup> |
| 2e | 500 mg QD PLX9486 + 25 mg Sunitinib |
| 2e | 1000 mg QD PLX9486 + 25 mg Sunitinib |
| 2e | 1000 mg PLX9486 + 37.5 mg Sunitinib |

# (2) For all listings, add following footnotes: (see example in Listing 16.2.1.1 – Patient Disposition)

| (placed on patient number. | |
|-----------------------------------------------------------|-----------|
| led, respectively, as patient numbers | |
| completed Their initial Cohort and subsequently re-enroll | |
| l] Patient numbers | ndicated) |

Number all footnotes first by their order of occurrence from left to right in the table headings, then by their order of occurrence in the body of listing itself

(3) All listings will be ordered by the following (unless otherwise indicated in the mock):

Study Part, Study Part, Patient number, Date, Visit and Time points


Plexxikon Inc.


| 2 |
|---|
| 1 |
| ì |
| 4 |

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

(4) For all listings, the mock shells outline layout for Study Part 1 – Dose Escalation Study Parts (Single-Agent PLX9486). The remainder of the listings will follow the same format for other Study Parts, unless specified otherwise in the mocks. Sponsor, protocol, and footnotes will appear on all pages of all Study Parts.

(5) Display complete and partially missing dates in standard format, with no spaces.

## For example:

15JUN2015
JUN2015 (if day is missing)
2015 (if month and day are missing)

Plexxikon Inc.

PLX121-01

Clinical Study Report PLX121-01


Statistical Analysis Plan 01Jul2020

Plexxikon Inc. Protocol PLX121-01 Listing 16.2.1.1
Patient Disposition

| | | | | | | Date of First | | Date of Last | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Dose/ | | Dose of | | |
| | | | | | | Date of Last | | PLX9486//Date | | |
| | | | | | | Dose/ | | of Last Dose of | f Primary | Pregnancy |
| | | | | | Informed | Duration of | | PLX3397 or | Reason for | during |
| Study Planned Patient | | Safety | EE | PK | Consent | Treatment <sup>[4]</sup> | Date of Reason for Study | Sunitinib [5] | Ending | the |
| Part Dose No. | Site | Population <sup>[1]</sup> P | opulation <sup>[2]</sup> | Population <sup>[3]</sup> Date | Date | (days) | Study Exit Completion/Discontinuation. | | Treatment | study? <sup>[6]</sup> |

Yes Adverse Event: 2\_xxxxx\_14 ■Clincial Progression Yes/No Yes/No Yes/No 250 mg 1 PLX9486

Note: For Study Part column, Px-Cy = Study Part x - Study Part y. For study part 2b, patients in the first Cohort were assigned to fast for at least 8 hours prior to dosing of study drug while patients in the second Cohort were dosed in a non-fasted state. For study part 2e, patients in Cohorts 1 and 2 were dosed with food while patients in Cohort 3 were assigned to fast for at least 8 hours prior to dosing of study drug. As of Amendment 6, patients who were assigned to fasting are no longer required to fast and may take their study medication with food.

[1] All patients who received study medication.

[2] All patients who have taken at least 1 dose of study drug and have had at least 1 post-baseline tumor assessment or discontinue study medication early due to disease progression or death.

[3] All patients who have adequate PK and PD data.

<sup>[4]</sup> Duration of treatment is defined as the last dose date minus the first dose date plus 1. Date of first dose is the earliest dose date of any of the study drugs (PLX3397, and sunitinib), including dose dates from the run-in PK period. Date of last dose is the latest dose date of any of the study drugs (PLX3486, PLX3397, and sunitinib).

[5] Dates of last dose of study drugs are derived.

<sup>[6]</sup> If male, did the patient's partner have a pregnancy during the study?

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [7] Patient numbers

AE = Adverse Event; DLT = Dose Limiting Toxicity.

EE = Efficacy Evaluable; PK = Pharmacokinetic; RECIST = Response Evaluation Criteria In Solid Tumors.

16.1.9 Documentation of Statistical Methods

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020


Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01

Listing 16.2.2.1 Demographics and Baseline Characteristics

| No, Post-<br>Menopausal/Yes,<br>Hormonal<br>Contraception | Dose Pat | tient No. | Study Planned Age Part Dose Patient No. Date of Birth (years) <sup>[1]</sup> Gender | Age<br>(years) <sup>[1]</sup> | Gender | For female, childbearing potential? <sup>[2]</sup> | Ethnicity | Race <sup>[3]</sup> | Weight Height<br>(kg) (cm) | Is paueir to pau | s<br>s<br>(kg/m <sup>2</sup> ) <sup>[4]</sup> | s pauent in<br>ingle dose F<br>PK sub-<br>study? | is patient in Optional Optional single dose Paired Tumor Fresh Tumor PK sub- Biopsy? Biopsy? study? | Optional<br>Fresh Tumor<br>Biopsy? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | xx-xx | DDMMMYYY | , xx | | No, Post-<br>Menopausal/Yes,<br>Hormonal<br>Contraception | Ī | | XXX.X | | xx.x | Yes/No | Yes/No | Yes/No |

date 

time

Programmer note:

1) If there is more than one "Race" separate by "/".

<sup>&</sup>lt;sup>[1]</sup> Age is calculated as of the date the informed consent is signed.
<sup>[2]</sup> If the answer is No, the reason is specified; if the answer is Yes, the method of contraception is specified.

<sup>[3]</sup> Patients could mark more than one race.
[4] BMI is derived as the weight in kilograms divided by the square of the height in meters.
[5] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers BMI = Body mass index.

Clinical Study Report PLX121-01 16.1.9 Documentation of Statistical Methods PLX9486 Statistical Analysis Plan 01Jul2020 Page 1 of x Listing 16.2.2.2 Medical History Plexxikon Inc. Protocol PLX121-01 Plexxikon Inc. PLX121-01

Unknown End Date Ongoing? Yes/No DDMMMYYYY Onset Date Unknown Description Any Past and/or Concomitant Diseases or Past Surgeries? Body System Yes/No Patient No. 250 mg QD PLX9486 Planned Dose Study Part

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers

date 

time

- Programmer notes:

  1) Show body system names vice body system codes.
  2) Sort by body system shown in the CRF then by description within each patient.

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

> Protocol PLX121-01 Plexxikon Inc.


## Listing 16.2.2.3.1 Primary Cancer History – Study Part 1 Part 1 of 2

| | | | Anatomical | At Initia | al Histolog | itial Histologic Diagnosis | | | Anatomical | At Study Entry | Entry |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Patient | Location<br>of Primary | | Tumor | T/N/M | — Histologic Degree of | Date of<br>Metastatic | Location of<br>Metastatic | Tumor | |
| Study Part 1 | study Part Planned Dose No. | No. | Tumor | Date | Stage | Stage | Subtype Differentiation | Diagnosis | Disease | Stage | Stage |
| | 250 mg QD<br>PLX9486 | | | | | Tx/Nx/M0 | | | | | |

Part 2 of 2

| | | Genomi<br>on Tur | Genomic Analysis<br>on Tumor Tissue | | |
|---|---|---|---|---|---|
| | Patient | | Anatomical | KIT Mutation? If yes, | Ö |
| Study Part Planned Dose No. | No. | Performed? Location | Location | specify | If yes, specify |
| | | Yes: lab | | | |
| | | name/No | | Yes: specify / No | Yes: specify / No |
| 1 250 mg QD | | | | | |
| PLX9486 | | | | | |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers

date 

time

## Programmer notes:

- If there is more than one "Anatomical Location of Primary Tumor" separate by "?".
  - Sort by date of initial histologic diagnosis date within each patient.
- If genomic analysis was performed on tumor tissue, specify lab performing analysis in column 'Performed'. 2000
- For column 'T/N/M Diagnosis (under 'At Initial Diagnosis' and 'At Study Entry')) if one of the T, N, or M diagnosis is missing display 'Missing' for that diagnosis (e.g. if T diagnosis is missing and N diagnosis = Nx, and M diagnosis = M, diagnosis = Nx, and M dia
  - For column 'Anatomical Location of Metastatic Disease' combine all applicable locations separated by ";" (locations are variables MH1LOCxx in the raw datasets)


Statistical Analysis Plan 01Jul2020


Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01

Listing 16.2.2.3.2 Primary Cancer History – Study Part 2 Part 1 of 3

| If Germ Cell | E |
|----------------------|---|
| ic Diagnosis I | |
| At Initial Histologi | E |
| V | |
| | • |

| | | | At Initial | Histolog | ic Diagnosis | At Initial Histologic Diagnosis If Germ Cell |
|---|---|---|---|---|---|---|
| | Patient | | | Tumor | Tumor T/N/M | Tumor, |
| Planned Dose No. | No. | Primary Tumor Type | Date | Stage | Date Stage Stage | Specify |
| 250 mg QD<br>PLX9486 | XX-XX | Other: Specify | Date9. | IĀ | Date9. IA Tx/Nx/M0 Non-<br>Seminon<br>Specify | Non-<br>Seminoma:<br>Specify |

### Part 2 of 3

| | T/N/M | tage | |
|---|---|---|---|
| At Study Entry | T/T | Sta | |
| At Stu | Tumor | Stage | |
| Histologic — | Histologic Degree of | Subtype Differentiation | |
| | T/N/M | Stage | Tx/Nx/M0 |
| ologic Diagnosis | Tumor | Stage | |
| At Initial Histologic I | | Date | |
| Anatomical<br>Location — | of Primary | Tumor | |
| | Patient | No. | XX-XX |

Part 3 of 3

| | Specification of | Mutation | Present | XXXXXX | |
|---|---|---|---|---|---|
| | 3, | | Exon Present | ∞ | Other: Specify |
| | | Diagnosis | Timeframe | | |
| Entry | Other non-KIT significant | Mutation? If mutations? Diagnosis | yes, specify If yes, specify Timeframe Exon Present Present | Yes: specify / Yes: specify /<br>No No | |
| issue at Study E | KIT | | yes, specify | Yes: specify<br>No | |
| Genomic Analysis on Tumor Tissue at Study Entry | | Anatomical | Location | XXXXXX | |
| Genomic Ar | | | Performed? | Yes: lab name/No | |
| gnosis | Other non-<br>KIT<br>significant | mutations? | If yes, specify | Yes: specify /<br>No | |
| Genomic Analysis<br>on Tumor Tissue at Initial Diagnosis | KIT | Anatomical Mutation? If | No. Performed? Location yes, specify If yes, specify | Yes: lab xxxxxx Yes: specify / Yes: specify / name/No No | |
| | | Anatomica | 1? Location | XXXXXX | |
| OL | | | Performed | Yes: lab<br>name/No | |
| | | Patient | No. | | |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers


## 16.1.9 Documentation of Statistical Methods PLX9486

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

date 

time

## Programmer notes:

- If there is more than one "Anatomical Location of Primary Tumor" separate by "?".
  - Sort by date of initial histologic diagnosis date within each patient.
- If genomic analysis was performed on tumor tissue, specify lab performing analysis in column 'Performed'.

  For column 'T/N/M Diagnosis (under 'At Initial Diagnosis' and 'At Study Entry')) if one of the T, N, or M diagnosis is missing display 'Missing' for that diagnosis (e.g. if T diagnosis 2284
  - is missing and N diagnosis =Nx, and M diagnosis=M0, display 'Missing/Nx/MO')

    For column 'Anatomical Location of Metastatic Disease' combine all applicable locations separated by ";" (locations are variables MHILOCxx in the raw datasets) 2)


Plexxikon Inc.


Plexxikon Inc. PLX121-01 PLX9486

Plexxikon Inc. Protocol PLX121-01

Statistical Analysis Plan 01Jul2020 Page 1 of x

Clinical Study Report PLX121-01

Listing 16.2.2.4
Prior Treatment for Primary Malignancy

| son<br>ng<br>t | | |
|---|---|---|
| Primary Reason<br>for Stopping<br>Treatment | | |
| Best Response<br>Setting Start Date Stop Date to Treatment | | |
| Stop Date | | |
| Start Date | | |
| Setting | | |
| Description | her: Specify | |
| If Yes, Type of<br>Therapy | Surgery Other: Specify | |
| ecord<br># | 1 | |
| Any previous<br>primary<br>malignancy R<br>treatment? | Yes/No | |
| Patient<br>No. | | |
| Study Patient Patient Part Planned Dose No. | 250 mg QD<br>PLX9486 | 350 mg QD |
| Study<br>Part | - | |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers

time

date 

Programmer note:

1) Sort by Start Date and then record number within each patient.

Clinical Study Report PLX121-01


Statistical Analysis Plan 01Jul2020 Plexxikon Inc. PLX121-01

Prior and Concomitant Medications **Listing 16.2.2.5** 

Protocol PLX121-01

Plexxikon Inc.

| Indication | MH # 21_CONSTIPATION_<br>Primary AE #3_INTERMITTENT DIARRHEA | Additional AE(s): #1_DIARRHEA/ # 2_DIARRHEA/ Other: STABLE BRAIN METASTASES |
|---|---|---|
| Dose Route/<br>Form Frequency Indication | Oral /<br>QD | |
| | 4 (mg) Tablet | |
| Dose<br>(Units) | 4 (mg) | |
| Start Date/<br>Stop Date | Ongoing | |
| Study Planned Patient Any RecordPreferred Name // Part Dose No. Medications # <sup>[1]</sup> Verbatim | NATURAL OPIUM<br>ALKALOIDS//<br>MORPHINE SULFATE//<br>I MS CONTIN | 2 |
| Any<br>Medications | Yes | |
| Patient<br>No. | | |
| Planned<br>Dose | 250 mg QD<br>PLX9486 | |
| Study<br>Part | - | |

Note: Prior medications are those that start prior to the first dose of any study drugs, even if the medications continues after dosing. Concomitant medications are those which are taken at any time between the date of first dose and the date of last dose of any study medication. In cases where it is not possible to determine if a medication is concomitant, the medication is classified as

Note: Only patients who reported taking any non-study medication from 14 days prior to study treatment or during the course of the study (including over-the-counter and prescription drugs) are recorded and listed.

<sup>[1]</sup> Prior medications are denoted by a P, concomitant medications are denoted by a C, prior and concomitant medications are denoted by PC following the CM #.

<sup>[2]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers AE = Adverse Event; ATC = Anatomical Therapeutic Chemical; MH = Medical History.

time date 

## Programmer notes:

- Sort by start date and stop date, and then CM # within each Study Part/patient.
  - Show the unit, dose form, route and frequency, not the codes.
- Use XMED dataset.
- See the footnote regarding flagging of conmeds starting after the first dose of a patient's dose escalation Study Part.
- For column Indiccation', concatenate if there are multiple indications. Use '7' to separate the different indications. 22848

| Occumentation of Statistical Methods | | |
|--------------------------------------|--------------------|----|
| Ğ, | tatistical Methods | |
| | Ť | 98 |

| Plexxikon Inc. PLX121-01 | Statistical Analysis Plan<br>01Jul2020 |
|---|---|
| Plexxikon Inc.<br>Protocol PLX121-01 | Page 1 of x |

Clinical Study Report PLX121-01

| | Medical Monitor Significance | Assessment Significant/ Not significant/More information needed | | |
|---|---|---|---|---|
| Listing 16.2.2.6<br>Major Protocol Deviations | | Verbatim | sts CIDI scan lost | Study drug packages not returned to site |
| | Protocol<br>Deviation | Visit Category | CID1 Procedures/Tests CID1 scan lost | EOS Study Drug |
| | Patient | No. | | |
| | Protocol Study Patient Deviation | Part Planned Dose | 1 250 mg QD<br>PLX9486 | 350 mg QD<br>PLX9486 |

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled.

date 

time

Programmer note:

I) Sort by Start Date, visit, category, and verbatim within each patient.

16.1.9 Documentation of Statistical Methods PLX9486

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020


Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01

Listing 16.2.3.1.1 PLX9486 Dosing Log

| | | XXX; | |
|---|---|---|---|
| Drug Overdose | verdose<br>lated to<br>AE? Related AEs | Primary AE: xxx/<br>Secondary AE(s): xxxxx;<br>xxxxx | |
| Drug | Overdose<br>related to<br>AE? | res/No | |
| | Overdose Overdose<br>Occurred? related to | Yes/No Yes/No | |
| Dose Change due to AE | Overdose Overdose Overdose Dose AE Related to Occurred? related to Change 121 AE? | Yes/No Xxxx xxxx | |
| Dose Cha | Dose<br>Change? | Yes/No | |
| • | Actual Dose Taken Dose Dose AE Related to (mg) <sup>[1]</sup> Reason Change? Dose Change | Starting<br>Dose | PK RUN<br>IN<br>Starting<br>Dose |
| | ribed<br>n by | Yes/No | |
| | Prescribed<br>Total Dail<br>Dose (mg | 250 | 350 |
| Prescribed | Dose (mg) /Prescribed Daily Dose Frequency | ххх/QD | |
| | Stop Date | date9. | |
| | Start Date | date9. | |
| | Study Planned Parient No. Start Date Stop Date Frequency Dose (mg) Patient? | I | |
| | Planned<br>Dose | 250 mg<br>QD<br>PLX9486 | 350 mg<br>QD |
| | Study<br>Part | - | |

time

date 

## Programmer note:

- Sort by start date and stop date within each Study Part/patient.

  For column 'If Yes, AE(s)': concatenate all AEs. Separate primary AE with Secondary AEs by '', separate more than I secondary AEs by ';'
  Continue for all study parts
  If change is due to overdose there may be multiple associated AEs. Append them together with the Primary first, then the Secondary(s).


Plexxikon Inc.


<sup>[1]</sup> If prescribed dose was not taken by the patient.
[2] Patient is considered to have had overdose if Dose Reason is 'Patient Overdose'.
[3] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers

| Methods | |
|---------------|--------|
| Statistical ] | |
| umentation of | |
| .9 Docum | 701011 |
| = | , |
| 16 | ż |

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01


Plexxikon Inc. Protocol PLX121-01

Listing 16.2.3.1.2 PLX3397 Dosing Log

| Overdose<br>occured? <sup>[2]</sup> | |
|---|---|
| as Change<br>Dose due<br>to AE? If Yes, AE(s) | Primary AE:<br>xxx/ Secondary<br>AE(s): xxxxx;<br>xxxxx |
| Was Change<br>in Dose due<br>to AE? | Yes/No |
| Jose<br>Dose<br>Reason | Starting<br>Dose |
| Prescribed Dose (mg) Prescribed Prescribed Actual Dose Daily Dose Total Daily Dose Taken Taken Frequency Prescribed Prescribed Actual Dose Daily Dose (mg) by Patient? (mg) | 250 Yes/No |
| 7 | xxx/QD |
| Date Stop Date | date9. |
| | date9. |
| Study Planned Patient<br>Part Dose No. Start | XX-XXX |
| Planned<br>Dose | |
| Study<br>Part | - |

date 

time

## Programmer note:

- Sort by start date and stop date within each Study Part/patient.
   For column 'If Yes, AE(s)': concatenate all AEs. Separate primary AE with Secondary AEs by '', separate more than I secondary AEs by ';'
   This listing is only relevant for Study Part 2b.

<sup>[1]</sup> If prescribed dose was not taken by the patient.
[2] Patient is considered to have had overdose if Dose Reason is 'Patient Overdose'
[3] Patient Nos completed Study and subsequently re-enrolled, respectively, as Patient Nos

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Listing 16.2.3.1.3 Sunitinib Dosing Log

| | | :xxxx; | |
|---|---|---|---|
| Drug Overdose | verdose<br>lated to<br>AE? Related AEs | Primary AE: xxx/<br>Secondary AE(s): xxxxx;<br>xxxxx | |
| Drug | Overdose<br>related to<br>AE? | Yes/No | |
| | Overdose Overdose<br>Occurred? related to | Yes/No Yes/No | |
| Dose Change due to AE | Overdose Overdose Overdose Dose AE Related to Occurred? related to Change? | Yes/No Xxxxx xxxx | |
| Dose Ch | Dose<br>Change? | Yes/No | |
| | Dose<br>Reason | Starting<br>Dose | PK RUN<br>IN<br>Starting<br>Dose |
| | Actual<br>I Dose<br>Taken<br>(mg) <sup>[1]</sup> | | |
| | Study Planned Study Part Dose Patient No. Start Date Stop Date Frequency Dose (mg) Patient? (mg) <sup>[1]</sup> Reason Change? Dose Change | Yes/No | |
| | Prescribed<br>Total Dail<br>Dose (mg | 250 | 350 |
| Prescribed | Dose (mg)<br>/Prescribed<br>Daily Dose<br>Frequency | ххх/бД | |
| | Stop Date | date9. | |
| | Start Date | date9. | |
| | Patient No. | | I |
| | Planned<br>Dose | 250 mg<br>QD<br>PLX9486 | 350 mg<br>QD |
| | Study<br>Part | - | |

time

date 

## Programmer note:

- Sort by start date and stop date within each Study Part/patient.
   For column 'If Yes, AE(s)': concatenate all AEs. Separate primary AE with Secondary AEs by '', separate more than I secondary AEs by ';'
   This listing is only relevant for Study Part 2e.

<sup>[1]</sup> If prescribed dose was not taken by the patient.
[2] Patient is considered to have had overdose if Dose Reason is 'Patient Overdose'
[3] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers

| ethods | |
|-----------------|---------|
| atistical Me | |
| f Sta | |
| Ocumentation of | |
| Docume | 981 |
| 16.1.9 | PLX9486 |

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01


Plexxikon Inc. Protocol PLX121-01

Listing 16.2.3.2 Study Drug Accountability

| Comments | |
|---|---|
| Amount Returned (Tablets) | |
| Treatment Label<br>ID Returned | |
| Date Returned | date9. |
| Amount Dispensed (Tablets) | |
| Treatment Label<br>ID Dispensed | |
| Study Planned Treatment L. Part Dose Patient No. Date Dispensed ID Dispense | date9. |
| Patient N | |
| Planned<br>Dose | 250 mg QD<br>PLX9486 |
| Study<br>Part | 1 |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers

date 

time

Programmer note:  $I) \quad \textit{Sort by dispensed date and returned date within each Study Part/patient.}$ 


| ethods | |
|-----------------|----------|
| ] Me | |
| tatistica | |
| r | |
| ion of | |
| tatio | |
| umentation of S | |
| Jocui | 20 |
| $\overline{}$ | 7 |
| $\sim$ | 01 VO 10 |
| ∹: | P |
| 9 | 1 |
| $\overline{}$ | _ |

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01


Listing 16.2.3.3.1 PLX9486 Overall Exposure

| Total Dose Taken (mg) <sup>[3]</sup> | XXX |
|------------------------------------------------|----------------------|
| Duration of<br>Treatment (Days) <sup>[2]</sup> | XXX |
| Patient No. | |
| Study Part Planned Dose Patient No. | 250 mg QD<br>PLX9486 |
| Study F | П |

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers <sup>[2]</sup> Duration of treatment of PLX9486, derived as the last dose date of PLX9486 minus the first dose date of PLX9486 plus 1. <sup>[3]</sup> The total dose taken is derived from the duration of treatment (in days) times the assigned dose.

date 

time

Programmer Note:

1) Present all study parts


| s | |
|-----------------|----------|
| Methods | |
| Statistical | |
| umentation of 3 | |
| ocument | 7 |
| 16.1.9 D | DI V0/0/ |

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Listing 16.2.3.3.2 PLX3397 Exposure

| | Total Dose Taken (mg)[3] | | | | | XX |
|---|---|---|---|---|---|---|
| Duration of | Treatment (Days)[2] | | | | | XX |
| | Patient No | | | | | XX-XX |
| | Study Part Planned Dose Patient No | 500 mg QD | PLX9486+ | 600 mg | PLX3397 | fasting |
| | Study Part | | | | | 1 |

time date 

Programmer Note:

1) Present only for Study Part 2b.

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [2] Duration of treatment of PLX3397, derived as the last dose date of PLX3397 minus the first dose date of PLX3397 plus 1.

[3] The total dose taken is derived from the duration of treatment (in days) times the assigned dose.

| thods | |
|-------------------|---|
| 1 Me | |
| tatistic | |
| nentation of S | |
| ocan | ` |
| $\overline{\Box}$ | |
| 5. | |
| $\frac{1}{2}$ | , |
| = | Z |

Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Listing 16.2.3.3.3 Sunitinib Exposure

| | Total Dose Taken (mg) <sup>[3]</sup> | | | xx |
|---|---|---|---|---|
| Duration of | Treatment (Days)[2] | | | XX |
| | Patient No. | | | XXX-XX |
| | Study Part Planned Dose Patient No. | 500 mg QD | PLX9486 + 25 | mg Sunitinib |
| | Study Part | | , | 1 |

time date 

Programmer Note:
1) Present only for Study Part 2e.

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [2] The total dose taken is derived from the duration of treatment (in days) times the assigned dose.
[3] Duration of treatment of PLX9486, derived as the last dose date of PLX9486 minus the first dose date of PLX9486 plus 1.

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020


Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01

Tumor Assessment (Target Lesions) Listing 16.2.4.1

| Percent Change from Any Nadir New (%)[5] Lesions? | Yes/No | Yes/No | Yes/No | Yes/No |
|---|---|---|---|---|
| Percent<br>Change<br>from<br>Nadir<br>(%) <sup>[5]</sup> I | ŕ | , | · | , |
| Change<br>from<br>Nadir<br>(cm) <sup>[5]</sup> | | | | |
| Nadir<br>(cm) | | | | |
| Percent<br>Change<br>from<br>Baseline<br>(%) [3] | | | XX.X | X.X |
| Change<br>from<br>Baseline<br>(cm) <sup>[3]</sup> | | | - 1.9 | - 1.9 |
| Sum of<br>Longest<br>Diameters<br>(cm) | 6.5 | 6.5 | 8.4 | 8.4 |
| Longest Diameter I (cm) [2] | 3.2 | Jnable to<br>Evaluate | 4.60 | 3.80 |
| Sum of Change Longest Longest from Method of Diameter Diameters Baseline Description Location Assessment (cm) <sup>[2]</sup> (cm) (cm) <sup>[3]</sup> | Spiral Computed Tomography | Spiral Computed Tomography | (CT) Spiral Computed Tomography | (CT) Spiral 3.80 Computed Tomography (CT) |
| ocation | Liver | Liver | Liver | Liver |
| Description I | LIVER,<br>SEGMENT<br>II | RIGHT<br>LIVER | LIVER,<br>SEGMENT<br>II | RIGHT<br>LIVER |
| Lesion<br># [1] | * | * | | 7 |
| Radiographic Assessment Evaluation Lesion Date Performed? # [1] | Yes | | Yes | |
| Assessment<br>Date | | | | |
| Visit | SCREEN | | Unscheduled | |
| Patient<br>No. | I | | <u> </u> | |
| Planned Patient<br>Dose No. | 250 mg<br>QD<br>PLX9486 | | | |
| Study Part | - | | | |

Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug.

<sup>[1]</sup> A '\*' indicates baseline. A <sup>A</sup> indicates assessments were collected after last dose date.

time

date

Programmer notes:

1) Sort by visit and lesion number within each patient.


<sup>[2]</sup> If lymph node, short axis is recorded instead.

<sup>&</sup>lt;sup>[3]</sup> Change from baseline, and percent change from baseline of the sum of longest diameters. <sup>[4]</sup> Nadir is the smallest sum of longest diameters recorded since treatment started.

<sup>[5]</sup> Change and percentage change from nadir are shown for the assessment that produces the nadir (equal to zero there by definition) and for each subsequent assessment.

[6] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers UNS = Unscheduled.

16.1.9 Documentation of Statistical Methods PLX9486

Statistical Analysis Plan 01Jul2020 Plexxikon Inc. PLX121-01

Listing 16.2.4.2 Tumor Assessment (Non-Target Lesions) Plexxikon Inc. Protocol PLX121-01


Clinical Study Report PLX121-01

| Non-Target Lesion Status <sup>[2]</sup> | Unable to Evaluate |
|---|---|
| Method | Spiral Computed<br>Tomography (CT) |
| Location | Lung |
| Lesion<br># Description | LEFT UPPER LOBE LUNG |
| Lesion<br># | 1 |
| If No,<br>Reason [2] | |
| Any Non-<br>Target<br>Lesion?/<br>Radiographic<br>Evaluation<br>Performed? | Yes/No |
| Assessment<br>Date | |
| Visit | SCREEN |
| l Patient<br>No. | 9 |
| Study Planned Patient<br>Part Dose No. Visit | 250 mg<br>QD<br>PLX9486 |
| Study<br>Part | 1 |

Note: Baseline is defined as the last value obtained on or before the date and time of the first dose of any study drug.

<sup>[1]</sup> If Baseline records, whether any non-target lesion(s) was identified at baseline. If non-baseline records, whether radiographic evaluation was performed.

<sup>[2]</sup> For non-baseline records.

<sup>[3]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and subsequently re-enrolled.

date 

time

Programmer note:  $I) \quad Sort \, by \, visit, date \, and \, lesion \, number \, within \, each \, patient.$ 

| 70 | |
|----------------|-----------|
| al Method | |
| f Statistica | |
| sumentation of | |
| 1.9 Doc | 781/0X Id |
| 16. | Ы |

Statistical Analysis Plan 01Jul2020 Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Clinical Study Report PLX121-01

| | Method of |
|----------------------------------------------------|---------------------|
| sions | Longest<br>Diameter |
| Listing 16.2.4.3<br>Tumor Assessment - New Lesions | : |
| | Assessment |
| | pə |

Unable to Evaluate? Yes/No Assessment Location completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers (cm) Lesion # Description Date Visit C3D1 Patient No. 250 mg QD PLX9486 Dose Plannec Study Part

[1] Patient numbers UNS = Unscheduled.

date 

time

Programmer note:

1) Sort by time point, date and lesion number within each patient.

16.1.9 Documentation of Statistical Methods

PLX9486

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01 Page 1 of x

Protocol PLX121-01 Plexxikon Inc.

Tumor Response Assessment (Target and Non-Target Lesions) **Listing 16.2.4.4** 

| Study Part Planned Dose Patient No. Visit | Visit | Assessment<br>Date | Days from<br>First Dose <sup>[1]</sup> | Target Lesion<br>Response <sup>[2]</sup> | Days from Target Lesion Non-Target<br>First Dose <sup>[1]</sup> Response <sup>[2]</sup> Lesion Response | New Lesion? | Investigator Assessed Overall New Lesion? Response <sup>[3]</sup> | Investigator Assessed Overall Calculated RECIST Response <sup>[3]</sup> Overall Response <sup>[4]</sup> |
|---|---|---|---|---|---|---|---|---|
| 1 250 mg QD | Screen | | | NE | NE | | NE | NE |
| FLA9400 | Unscheduled | | | Not Done | Non-CR/Non-PD | Yes/No | PD | PD |

Note: A \* after Assessment Date indicates assessments after last dose date.

[1] Days from first dose of study drug is derived as the assessment date - first dose of any study drug + 1.

[2] PD is defined as ≥ 20% relative increase from nadir and absolute increase of at least 5 mm in the sum of diameters of target lesions.

[3] Overall response is determined by Investigator using RECIST v1.1, and recorded in the CRF form Tumor Response Assessment.

[4] Derived programmatically using RECIST v1.1 criteria based on target, non-target responses and new lesion evaluation recorded in the database. [5] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers

CR = Complete Response; NE = Not Evaluable (Inevaluable for Response); PD = Progressive Disease; PR = Partial Response; RECIST = Response Criteria Evaluation in Solid Tumors; SD = Stable

UNS = Unscheduled.

date 

time

## Programmer notes:

- Put 'Not Done' into response columns when response assessment is Not Done (RSND1 or RSDN2 is 1).
- For column 'Reason for PD', fill in if Derived Overall Response is PD. Possible values: New Lesion(s), 20% relative increase [2], New Lesion(s) and 20% relative increase [2] Sort by date, visit and lesion number within each patient.
   Put 'Not Done' into response columns when response ass.
   For column 'Reason for PD', fill in if Derived Overall Re.
   Program for footnote 'Note: A \* after Accomment Details.
  - Program for footnote 'Note: A \* after Assessment Date indicates assessments after last dose date.'

Clinical Study Report PLX121-01

Plexxikon Inc.

Statistical Analysis Plan 01Jul2020

PLX121-01


Protocol PLX121-01 Plexxikon Inc.

Derived Efficacy Endpoints Based on Tumor Response Listing 16.2.4.5

| | | Duration of | uration of Response <sup>[11]</sup> | Progression. | Progression-Free Survival <sup>[2]</sup> | Overall Survival <sup>[3]</sup> | urvival <sup>[3]</sup> | Tumor Response | sponse |
|---|---|---|---|---|---|---|---|---|---|
| Study Planned<br>Part Dose | Planned Patient<br>Dose No. | Days | Censor | Days | Censor | Days | Censor | Clinical Benefit <sup>2[4]</sup> Response <sup>[5]</sup> | Best Overall<br>Response <sup>[5]</sup> |
| 1 250 mg | | | | | | | | Yes/No | |
| G) | | | | | | | | | |
| PI X948 | 5 | | | | | | | | |

<sup>[1]</sup> DOR is calculated for every patient with a response to therapy as the number of days from the date of initial response (PR or CR) to the date of first documented disease progression or death. whichever occurs first. If disease progression or death does not occur, DOR is censored as of the date of their last post-baseline tumor response evaluation.

time date


<sup>&</sup>lt;sup>[2]</sup> PFS is defined as the number of days from the start of therapy (i.e., C1D1) to the date of first documented disease progression or death, whichever occurs first. Patients without a post-baseline tumor response evaluation have their event censored on the first date of study drug If disease progression or death does not occur, PFS is censored as of the date of their last post-baseline tumor

<sup>[3]</sup> OS is defined as the number of days from the start of therapy (i.e., CID1) to the date of death. If a patient is lost to follow-up, OS is censored at the date of last contact. For more details, see SAP

<sup>[4]</sup> A patient is considered to experience Clinical Benefit if they have a Best Overall Response of CR, PR or SD that lasted for at least 16 weeks.

<sup>[5]</sup> Best Overall Tumor Response is the best overall response derived as the best of all Best Responses for each sequential pair of post-treatment time points (and in some cases, triplets of sequential time points). Best Responses for each sequential pair of post-treatment time points follow the rules for determining best response when confirmation of CR, PR, and minimum duration of SD are required. For more details, see SAP Section 8.1.2 and 8.1.3.

Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers Criteria Evaluation in Solid Tumors; SD = Complete Response; DOR = Duration of Response; NE = Not Evaluable; PD = Progressive Disease; PR = Partial Response; RECIST = Response Criteria Evaluation in Solid Tumors; SD =

Reference: Listings 16.2.4.1 and 16.2.4.4

| ethods | |
|----------------|-------|
| ical M | |
| tatisti | |
| n of S | |
| sumentation of | |
| came | |
| .9 Doc | X9486 |
| 16.1 | PLX |

Statistical Analysis Plan 01Jul2020 Plexxikon Inc. PLX121-01

Adverse Events Listing 16.2.5.1 Plexxikon Inc. Protocol PLX121-01

Part 1 of 3


Clinical Study Report PLX121-01

| | | | | Outcome | Recovered /<br>Resolved |
|---|---|---|---|---|---|
| | | Other Actions | | Event | None/xxxx |
| Relationship to PLX3397 or | Sunitinib/ | Action Taken | PLX3397 or | Sunitinib | Not Applicable<br>/ Not<br>Applicable |
| | | Relationship to | Action Taken with | Study Day <sup>[3]</sup> Study Day <sup>[3]</sup> DLT? <sup>[4]</sup> PLX9486 | /Yes/NoPossibly Related/ Not Applicable None/xxxxx Recovered<br>Dose Not Changed / Not Resolved<br>Applicable |
| | | | Start Date/ End Date/ | <sup>1</sup> Study Day <sup>[3]</sup> D | 36 |
| 8 | | | Start Date/ | Study Day <sup>[3</sup> | 2 |
| Initial<br>Severity/Maximum | Severity | | | | Yes/No Grade I/Grade 3 |
| Serious? Initial<br>Severi | | | | | Yes/No |
| System Organ | Class //<br>Preferred Term | Any AE // | Part Planned Dose No. AE? No. <sup>[1]</sup> Verbatim Text <sup>[2]</sup> | Yes/No 1* | |
| | | | Patient | No. | |
| | | | | Planned Dose | 250 mg QD<br>PLX9486 |
| | | | Study | Part | - |

Note: More detailed information about SAE can be found in Part 2, and about subsequent increase in severity can be found in Part 3 of the listing.

 $^{[1]}$  A \* after the adverse event number indicates a treatment emergent adverse event.  $^{[2]}$  AEs are coded using MedDRA v 23.0.

[3] Study Day is relative to the date of the first dose of study medication. Study Day is only displayed for AE dates with complete date information.

[4] DLTs are defined as AEs occurring during the first 28 days of study drug administration (Cycle 1) that are classified as possibly or probably related to the study drug, and meet one of the following Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria listed in SAP Section 3.1

[5] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers composition of the common Terminology Criteria for Adverse Events; DLT = Dose Limiting Toxicity; MedDRA = Medical Dictionary for Drug Activities, NA = Not Applicable

time date

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. PLX121-01

Listing 16.2.5.1 Adverse Events Part 2 of 3

| | s<br>t<br>11 | |
|---|---|---|
| | Other Serious<br>or Important<br>Medical Event | Yes/No |
| | Life-<br>Threatening | Yes/No |
| SAE Criteria | Initial or Prolonged<br>Hospitalization<br>Date of Admission/<br>Date of Discharge | Yes/<br>DDMMMYYYY/<br>DDMMMYYYY |
| | Death | Yes/No |
| | Persistent or<br>significant<br>disability or<br>incapacity | Yes/No |
| | Persistent or significant congenital Anomaly/disability or Birth Defect incapacity | Yes/No |
| | Serious? | Yes/No |
| | System Organ Class // Preferred Term // Verbatim AE No. <sup>[1]</sup> Text <sup>[2]</sup> | <del>*</del> */ |
| | Patient<br>No. | XXXXX |
| | Planned<br>Study Part Dose | 250 mg QD >><br>PLX9486 |
| | Study Part | |

 $<sup>^{[1]}</sup>$  A  $^*$  after the adverse event number indicates a treatment emergent adverse event.  $^{[2]}$  AEs are coded using MedDRA v18.0.

time

date


Plexxikon Inc.


<sup>[3]</sup> Study Day is relative to the date of the first dose of study medication. Study Day is only displayed for AE dates with complete date information.

[4] DLTs are defined as AEs occurring during the first 28 days of study drug administration (Cycle 1) that are classified as possibly or probably related to the study drug, and meet one of the following Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria listed in SAP Section 3.1

[5] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and subsequently re-enrolled.

Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers and subsequently re-enrolled, respectively, as patient numbers and reminology Criteria for Adverse Events; DLT = Dose Limiting Toxicity; MedDRA = Medical Dictionary for Drug Activities.

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan

Adverse Events Listing 16.2.5.1 Part 3 of 3

| 4th Increase in Severity | ity Date | .5 |
|---|---|---|
| Increase | 4th Severity | Yes/No Grade 5<br>(Fatal) |
| 4 <sup>tl</sup> | 4th | Yes/N |
| everity | Date | |
| 3rd Increase in Severity | 3rd Severity | Yes/No Grade 4<br>(Life<br>Threatening) |
| 3rd I | 3rd | Yes/No |
| verity | Date | |
| 2 <sup>nd</sup> Increase in Severity | 2nd Severity | Yes/No Grade 3<br>(Severe) |
| 2 <sup>nd</sup> Ir | 2nd | Yes/No |
| verity | Date | |
| 1st Increase in Severity | Severity | es/No Grade 2<br>(Moderate) |
| 1 <sup>st</sup> In | 1st | Yes/No |
| | System Organ Organ Class // Preferred Preferred Term // Subsequent Study Planned Patient Verbatim Initial increase in Part Dose No. AE No. I <sup>1</sup> Text <sup>[2]</sup> Severity Severity Severity? | Grade 1 Yes/No<br>(Mild) |
| | Initial<br>Severity | Grade 1<br>(Mild) |
| | System Organ Class // Preferred Term // Verbatim | |
| | t<br>AE No. <sup>[7]</sup> | 2* 1* |
| | Patient<br>No. | <b>I</b> |
| | Planned<br>Dose | 250 mg<br>QD<br>PLX9486 |
| | Study<br>Part | - |

 $<sup>^{[1]}</sup>$  A  $^*$  after the adverse event number indicates a treatment emergent adverse event.

time

date 

## Note to Programmer:

- For columns 'Relationship to PLX3397 or Sunitinib/ Action Taken with PLX3397 or Sunitinib[5], in the column body, display 'NA/NA' for data from study part 1, display information of relationship/action taken with PLX3397 for Study Parts in study part 2b, display information of relationship/action taken with Sunitinib for Study Parts in study part 2e.
  - Sort by start date and end date within each patient.
- Note that there may be more than one "other" action taken. List all, separated by "?.
- Leave blanks at column 'End Date/Study Day' for observations which have completely missing AE End Date.
- If AE start date is partial date or missing, display 'DDMMYYY' only in column 'AE Start Date/Study Day'. If AE end date is partial date or missing, display 'DDMMYYY' only in column 'AE End Date/Study Day' 26420
  - Place footnote for re-enrolling patients on the Patient ID number.


<sup>&</sup>lt;sup>[2]</sup> AEs are coded using MedDRA v18.0.

<sup>[3]</sup> Study Day is relative to the date of the first dose of study medication. Study Day is only displayed for AE dates with complete date information.

<sup>&</sup>lt;sup>[4]</sup> DLTs are defined as AEs occurring during the first 28 days of study drug administration (Cycle 1) that are classified as possibly or probably related to the study drug, and meet one of the following Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria listed in SAP Section 3.1

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [5] Patient numbers

AE = Adverse Event; CTCAE = Common Terminology Criteria for Adverse Events; DLT = Dose Limiting Toxicity; MedDRA = Medical Dictionary for Drug Activities.

## 16.1.9 Documentation of Statistical Methods

PLX9486

Statistical Analysis Plan

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01 Page 1 of x

01Jul2020

Protocol PLX121-01 Plexxikon Inc.

Adverse Events Leading Changes in Study Treatment Listing 16.2.5.2

| | Outcome | | |
|---|---|---|---|
| | Severity/Maximum Relationship to Action Taken with A/B/C? Severity A/B/C <sup>[5]</sup> O | | Withdrawl/reduced/modified |
| | Relationship to A/B/C <sup>[5]</sup> | NA/NA/Yes | |
| Initial | Severity/Maximum<br>Severity | | |
| | $ m DLT$ ? $^{[4]}$ | | |
| | Start Date/ End Date/ Severity/Maximu Study Day [3] Study Day [3] Severity | | |
| System Organ<br>Class/ | Planned Patient AE No. Preferred Term/<br>study Part Dose No. [1] Verbatim Text [2] | | |
| | l Patient<br>No. | | 9 |
| | Planned<br>Dose | 250 mg | PLX948( |
| | Study Part | | 1 |

 $<sup>^{[1]}</sup>$  A  $^{*}$  after the adverse event number indicates a treatment emergent adverse event.

AE = Adverse Event; CTCAE = Common Terminology Criteria for Adverse Events; DLT = Dose Limiting Toxicity; MedDRA = Medical Dictionary for Drug Activities, NA = Not Applicable.

## Programmer note:

- Sort by start date and end date within each patient.
- Note that there may be more than one "other" action taken. List all, separated by ".
- Leave blanks at column 'End Date/Study Day' for observations which have completely missing AE End Date.
- If AE start date is partial date or missing, display 'DDMMYYY' only in column 'AE Start Date/Study Day'. If AE end date is partial date or missing, display 'DDMMYYY' only in column 'AE End Date/Study Day'.
- Include AEs if Action is "Drug Withdrawn" or datasets DS/DS2 indicate AE # led to Study Exit/ End of Study Treatmen and has an associated primary AE number.
- For columns 'Relationship to PLX3397 or Sunitinib/ Action Taken with PLX3397 or Sunitinib/5], in the column body, display 'NA/NA' for data from study part 1, display information of relationship/action taken with PLX3397 for Study Parts in study part 2b, display information of relationship/action taken with Sunitinib for Study Parts in study part 2e. 90
  - f a patient has a primary reason for study discontinuation on the study exit status form with an non-missing AE number, append a superscript [7] to the AE verbatim term in the 8
- If patients listed in footnote [8] appear in the listing, append the superscript [8] to the individual patient number in the listing,


Plexxikon Inc.


<sup>&</sup>lt;sup>[2]</sup> AEs are coded using MedDRA v 23.0.

<sup>[3]</sup> Study Day is relative to the date of the first dose of study medication. Study Day is only displayed for AE dates with complete date information.

<sup>[4]</sup> DLTs are defined as AEs occurring during the first 28 days of study drug administration (Cycle 1) that are classified as possibly or probably related to the study drug, and meet one of the following Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria listed in SAP Section 3.1

<sup>[5]</sup> Not Applicable for Study Parts in study part 1, relationship to and action take with PLX3397 for Study Parts in study part 2b, relationship to and action take with sunitinib for Study Parts in study

<sup>[6]</sup> AEs whose actions taken with study drug (PLX9486, PLX3397 or sumitinib) is 'Drug Withdrawn' or if in the CRF form 'End of Treatment', a patient's primary reason for ending treatment from is 'Adverse Event' and a non-missing associated primary AE is recorded.

<sup>[7]</sup> If patient has primary reason for study discontinuation from the CRF from 'Study Exit Status' being 'Adverse Event' and a non-missing associated primary AE. In this study there were no cases completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers which qualify for this footnote. [8] Patient numbers

time date 

16.1.9 Documentation of Statistical Methods PLX9486

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020

Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01


### Dose Limiting Toxicity **Listing 16.2.5.3**

| Other DLT | | | Specify [3] | | XXXX XXXXXX |
|---|---|---|---|---|---|
| DO. | | | Occurred? Type [1] Occurred? [2] Specify [3] | | Yes/No |
| Jose Limiting Hematologic | icities | | Type [1] | Type 1/ | Type 5 |
| Dose Limitin | Toxicities | | Occurred? | | Yes/No |
| Patient on | Study Drug | at Least | 28 Days? | | Yes/No |
| | | Date of | Assessment | | |
| | | AE Associated | with DLT | | |
| | | | DLT# | | |
| | | | Patient No. DLT # | | |
| | | Planned | Dose | 250 mg QD | PLX9486 |
| | | | Study Part | | 1 |

Type 1 = Grade 4 Neutropenia; Type 2 = Grade  $\geq$  3 Neutropenia with fever; Type 3 = Grade 4 Thrombocytopenia, Type 4 = Grade  $\geq$  3 thrombocytopenia with clinically significant bleeding; Type 5 = Grade  $\geq$  3 Anemia.

Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers AE = Adverse Event; DLT = Dose Limiting Toxicity.

date 

Programming note:

I) This can be done using EX3 dataset where the AETERM is populated. Only display the Types found in the data for a DLT, stack Type XType Y for each of the types a patient may have.

time

<sup>[2]</sup> If Yes then any other Grade  $\geq 3$  toxicity (except for those listed on the CRF) for which, either the Principal Investigator or Sponsor deems further dose escalation inappropriate.
Statistical Analysis Plan 01Jul2020

Plexxikon Inc. PLX121-01

Protocol PLX121-01

Plexxikon Inc.


Adverse Events Leading to Death Listing 16.2.5.4

| | 1 | |
|---|---|---|
| | ent Outcome | Recovered /<br>Resolved |
| A model | Taken/ Treatment of Event Outcome | None/xxxxx |
| Relationship to PLX3397 or Sunitinib/ | 480/ Action Taken w PLX3397 or Sunitinib <sup>[5]</sup> | NA/NA |
| Initial Severity/ Maximum Severity / | Serious DLT?! Action Taken with PLX3397 or Taken/ ? 4 PLX9486 Sunitinib <sup>[5]</sup> Treatment of E | Yes/N Grade 1 (Mild)/ o Grade 3 (Severe) Possibly Related/ Yes/No Dose Not Changed |
| | , | 5/<br>2 36 |
| System Organ Class | Patient Any AE Preferred Term // Start Date/ Study No. AE? No. <sup>[1]</sup> Verbatim Text <sup>[2]</sup> Study Day <sup>[3]</sup> Day <sup>[3]</sup> | * |
| | Patient Any<br>No. AE? | Yes/ 1*<br>No 2* |
| | Study Planned Dose | 250 mg QD PLX9486 |
| | Study<br>Part | - |

<sup>[1]</sup> A \* after the adverse event number indicates a treatment emergent adverse event.

date 

time

## Programmer notes:

- Sort by start date and end date within each patient.
- Note that there may be more than one "other" action taken. List all, separated by "!.
- Leave blanks at column 'End Date/Study Day' for observations which have completely missing AE End Date.
- If AE start date is partial date or missing, display 'DDMMYYY' only in column 'AE Start Date/Study Day'. If AE end date is partial date or missing, display 'DDMMYYY' only in column 'AE End Date/Study Day'. 2640
  - Include AEs with Severity, Toxicity Grade = Fatal (Grade 5) or Death Details dataset specified AEs

<sup>&</sup>lt;sup>[2]</sup> AEs are coded using MedDRA v 23.0.

<sup>[3]</sup> Study Day is relative to the date of the first dose of study medication. Study Day is only displayed for AE dates with complete date information.

<sup>&</sup>lt;sup>[4]</sup> DLTs are defined as AEs occurring during the first 28 days of study drug administration (Cycle 1) that are classified as possibly or probably related to the study drug, and meet one of the following Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria listed in SAP Section 3.1 [5] Not Applicable for Study Parts in study part 1, relationship to and action take with PLX3397 for Study Parts in study part 2b, relationship to and action take with sunitinib for Study Parts in study

<sup>&</sup>lt;sup>[6]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers common Terminology Criteria for Adverse Events; DLT = Dose Limiting Toxicity; MedDRA = Medical Dictionary for Drug Activities, NA = Not Applicable.

Plexxikon Inc.

Statistical Analysis Plan 01Jul2020 Page 1 of x

430

430

12.00 L (1)

35.70 L

PLX121-01

Protocol PLX121-01 Plexxikon Inc.

Listing 16.2.6.1.1 Hematology

| WBC | (x10 <sup>9</sup> /L) |
|------------|------------------------|
| RBC | (x10 <sup>12</sup> /L) |
| Platelets | (x10 <sup>9</sup> /L) |
| HCT | (%) |
| HGB | (g/dL) |
| Collection | Date / Time |
| Sampling | Collected? |
| | Visit |
| | Patient No. |
| Planned | Dose |
| | Study Part |

| HGB | (g/dL) | | 12.00 L [1]* | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Collection | Date / Time | ! | 707:57 | | | | | | | |
| Sampling | Collected? | | Yes/No | | | | | | | |
| | Visit | | SCREEN | | CID1 | C1D8 | C1D15 | C2D1 | : | EOS |
| | Patient No. | | | | | | | | | |
| Planned | Dose | 1 | 250 mg QD | PLX9486 | | | | | | |
| | Study Part | | - | | | | | | | |

Part 2 of 2

| Neutrophils Lymphocytes Eosinophils Monocytes |
|---|
| Neutrophils Lyn Planned Sampling Collection (Absolute) (A Dose Patient No. Visit collected? Date / Time (x10%L) (5 |
| Net Planned Sampling Collection (Al Dose Patient No. Visit collected? Date / Time (x |
| Planned Sc<br>Dose Patient No. Visit co |
| Planned Sc<br>Dose Patient No. Visit co |
| Planned<br>Dose Pa |
| Planned<br>Dose Pa |
| PI,<br>I |
| Study Part |

Note: L=Low and H=High with respect to laboratory reference ranges, where applicable. CTCAE v4.03 grades are in parentheses where applicable. \* indicates abnormal, clinically significant, as reported by the investigator. CTCAE grading is performed using data values only and does not consider symptomatic criteria.

[1] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled; CTCAE = Common Terminology Criteria for Adverse Events.

time date 

## Programmer notes:

- Sort by visit and analyte within each patient.
- Note that the same analyte may have different units and ranges for different patients due to test performed at difference among lab and etc.
- Convert lab results to a standard unit for each analyte (use ADLB.AVAL) 2284
- For column 'Result', display the number of decimal places as in ADLB.AVAL

| s | |
|-------------------|-------|
| Method | |
| tistical ] | |
| ta | |
| ocumentation of S | |
| Docum | 90 |
| 6.1.9 | VOV I |

Plexxikon Inc. PLX121-01 PLX9486

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01


## Listing 16.2.6.1.2 Hematology – Other Tests

| ne Other Tests Result Unit Range Low High Significant? 7 HH:MM BANDS xx.x xxxxx xx.x xx.x Yes/No | Visit Date/Time Other Test | Visit |
|---|---|---|
| XXXXX X.XX | | |

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled.

time date 

- Programmer notes:

  1) Sort by visit, date/time and analyte (test name alphabetically) within each patient.
  2) For column 'Result', display the result as original result and in the number of decimal places as in raw data

16.1.9 Documentation of Statistical Methods PLX9486

Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01


Statistical Analysis Plan 01Jul2020

## Listing 16.2.6.1.3 Hematology Laboratory Results: Grade 3 or Higher

| 250 mg QD PLX9486 xx-xx C1D1 date9./time5. 1 Grade 3 date9. 1 date4 date9. 1 date4 date9. 2 date9. date9. 3 | Study Part | Planned Dose | Patient No. | Visit | Collection<br>Visit Date/Time | Lab ID | Lab ID Lab Parameter (Unit) | Result | CTCAE<br>Grade | CTCAE Reference Reference<br>Grade Range Low Range High | Reference<br>Range High |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 1 2 3 3 3 | 1 | 250 mg QD<br>PLX9486 | | CIDI | date9./time5. | 1 | | | Grade 3 | | |
| date9. 2 date9. 3 | | | | | date9.<br>date9.<br>date9. | | | | Grade 4 | | |
| date9. 3 | | | | | date9. | 2 | | | | | |
| | | | | | date9. | 3 | | | | | |

Note: Laboratory parameters are graded according to CTCAE v4.03. CTCAE grading is performed using data values only and does not consider symptomatic criteria.

[11] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and Subsequently re-enrolled, respectively, as patient numbers completed; CTCAE = Common Terminology Criteria for Adverse Events.

date 

time

 Clinical Study Report PLX121-01

Page 1 of x Statistical Analysis Plan 01Jul2020 Phosphokinase Glucose Magnesium (mg/dL) (mg/dL) H 66 Creatine (D/L) 0.66(2)LDH (U/L) Uric Acid (mg/dL) Creatinine (mg/dL) Bilirubin 12.30 H (mg/dL) Direct Blood Urea Nitrogen (BUN) (mg/dL) Phosphorus Carbon Dioxide Bilirubin, (mmol/L) (mg/dL) Total 430 Calcium AST/SGOT 12.00 L [1] (I/I) Chloride (mmol/L) Albumin Listing 16.2.6.2.1 ALT/SGPT Chemistry
Part 1 of 3 35.70 L Protein, Total Potassium (mmol/L) Part 2 of 3 Part 3 of 3 (NT) Phosphatase DDMMYYYYY 12.00 L (1)\* (mmol/L) Sodium Alkaline (MT) Collection Collection Date / Time Date / Time Collection HH:MM Sampling collected? Sampling collected? Sampling collected? Yes/No SCREEN Visit C1D8 C1D1 Visit : Patient No. Dose Patient No. Planned Protocol PLX121-01 250 mg QD PLX9486 Planned Planned Dose Plexxikon Inc. Plexxikon Inc. PLX121-01 Study Study Study

Part

Note: L=Low and H=High with respect to Iaboratory reference ranges, where applicable. CTCAE v4.03 grades are in parentheses where applicable. \* indicates abnormal, clinically significant, as reported by the investigator. CTCAE grading is performed using data values only and does not consider symptomatic criteria.

(mg/dL)

(mg/dL)

(g/dL)

(g/dL)

Date / Time

Visit

Patient No.

Dose

Part

Part

EOS = End of study; UNS = Unscheduled; CTCAE = Common Terminology Criteria for Adverse Events.

time date 

Programmer notes:

Sort by visit, date/time and analyte within each patient.

- Note that the same analyte may have different units and ranges for different patients due to test performed at difference among lab and etc.
- Convert lab results to a standard unit for each analyte (use ADLB.AVAL) 2384
- For column 'Result', display the number of decimal places as in ADLB.AVAL


Plexxikon Inc.


| of Statistical Methods | |
|-------------------------|---------|
| 16.1.9 Documentation or | PLX9486 |

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020 Page 1 of x

Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01

Listing 16.2.6.2.2 Chemistry – Other Tests

| | Planned Patient | Patient | | Collection | | | | Reference | Reference Range | Clinically |
|---|---|---|---|---|---|---|---|---|---|---|
| Part | tudy Part Dose | No. | Visit | Date / Time | Other Tests | Result | Unit | Other Tests Result Unit Range Low | Range Low High Significant? | Significant? |
| 1 25 | 250 mg QD | | SCREEN | SCREEN DDMMMYYYY/HH:MM | XXXXX | XX.X | XXXXX | XX.X | XX.X | Yes/No |
| - | LA9400 | | | | XXXXX | XX.X | XXXXX | XX.X | XX.X | Yes/No |
| | | | : | | | | | | | |

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled.

time date 

- Programmer notes:

  1) Sort by visit, date/time and analyte (test name alphabetically) within each patient.
  2) For column 'Result', display the result and number of decimal places as in raw data

16.1.9 Documentation of Statistical Methods PLX9486

Clinical Study Report PLX121-01

Statistical Analysis Plan 01Jul2020


Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01

Listing 16.2.6.2.3 Chemistry Laboratory Results: Grade 3 or Higher

| Study Dort | Study Dart Dlannad Doca Dationt No Vicit | Dationt No | Vicit | Collection Date/Time | T 4º I | Collaction DetacTime 1 oh ID 1 oh Derematar (Unit) | Daemlt | CTCAE | Reference Reference | Reference<br>Dange High |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Fait | r Idillicu Dosc | r aucili 190. | V ISIL | COLLECTION DAIG TIME | E Lau ID | Lau ralanietei (Unit) | Nesalit | Olauc | Nalige Low | Naligo Iligii |
| | 250 mg QD | | | | | | | | | |
| 1 | PLX9486 | XX-XX | CIDI | date9./time5. | - | | | Grade 3 | | |
| | | | | date9. | _ | | | Grade 4 | | |
| | | | | date9. | - | | | | | |
| | | | | date9. | 1 | | | | | |
| | | | | date9. | 2 | | | | | |
| | | | | date9. | 8 | | | | | |

Note: Laboratory parameters are graded according to CTCAE v4.03. CTCAE grading is performed using data values only and does not consider symptomatic criteria.

[11] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and Subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled; CTCAE = Common Terminology Criteria for Adverse Events.

time date  

Statistical Analysis Plan

01Jul2020


Plexxikon Inc. PLX121-01

Listing 16.2.6.3.1 Urinalysis Plexxikon Inc. Protocol PLX121-01

Part 1 of 2

| udy<br>art | Planned<br>Dose | Patient<br>No. | Study Planned Patient<br>Part Dose No. Visit | Sampling<br>Collected? | Collection<br>Date / Time | Appearance | Color | Hd | Protein/<br>Albumin | Glucose/<br>Sugar | Ketones/<br>Acetones | Hemoglobin/<br>Blood | Nitrite |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 250 mg<br>QD<br>PLX9486 | | SCREEN | Yes/No | DDMMMYYYY/<br>HH:MM | CLEAR | STRAW | 99:0 | Positive,<br>1+* | Positive, Trace | Not Done | Positive, +4 Positive, Trace | sitive, Trace |

| | | | | Microsconic | | |
|---|---|---|---|---|---|---|
| Study | | Sampling | Collection | Exam | WBC | |
| Part Planned Dose Patient No. | Visit | Collected? | Date / Time | Performed? | (cells/hpf) | Casts |
| 1 250 mg QD<br>PLX9486 | SCREEN | Yes/No | DDMMMYYYY/<br>HH:MM | Yes/No | 50-100 | Absent/Present/Not Done |
| | CIDI | | | | | |

Part 2 of 2

Note: L=Low and H=High with respect to laboratory reference ranges for pH; \* indicates abnormal, clinically significant, as reported by the investigator.

[1] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed; WBC = White Blood Cell.

time date 

### Programmer notes:

- Sort by visit, date/time and analyte within each patient.
- Note that the same analyte may have different units and ranges for different patients due to test performed at difference among lab and etc.
  - Convert lab results to a standard unit for each analyte (use ADLB.AVAL)
- For column 'Result', display the number of decimal places as in ADLB.AVAL If test result is positive, Specify will be Trace, 1+, 2+, 3+, 4+ or Unknown. 22848

| tation of Statistical Methods | |
|-------------------------------|--------|
| 5.1.9 Documentation o | 707011 |

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


## Listing 16.2.6.3.2 Urinalysis – Other Tests

| Clinically<br>Significant? | Yes/No | Yes/No |
|---------------------------------------------|------------------|--------|
| Range Low High Significant? | XX.X | XX.X |
| Reference Other Tests Result Unit Range Low | XX.X | xx.x |
| Unit | XXXXX | XXXXX |
| Result | XX.X | XX.X |
| Other Tests | XXXXX | XXXXX |
| Collection<br>Date / Time | DDMMMYYYY/ HH:MM | |
| Visit | SCREEN | |
| Patient<br>No. | | |
| Planned<br>Part Dose | 250 mg QD | LA3400 |
| Study Part | 1 2 | |

[1] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and Subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and N/A = Not applicable; RBC = White Blood Cell; UA = Urinalysis; UNK = Unknown; UNS = Unscheduled.

time

date 

## Programmer notes:

- 1) Sort by visit, time point and analyte (test name alphabetically) within each patient.
  2) For column 'Result', display the result and number of decimal places as in raw data

16.1.9 Documentation of Statistical Methods PLX9486

Plexxikon Inc. PLX121-01


Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01

Listing 16.2.6.4.1 Coagulation

| Other, Specify/<br>Result/<br>Units | |
|------------------------------------------------|----------------------|
| International Oth<br>Normalized Ratio<br>(INR) | 86.0 |
| Partial Thromboplastin I Time (PTT) (sec) | 23.0* |
| Prothrombin Time<br>(PT) (sec) | 9.8 (1) |
| Was Patient<br>Fasting? | Yes/No/Unknown |
| Collection<br>Date / Time | DDMMMYYYY/<br>HH:MM |
| Sampling<br>Collected? | Yes/No |
| Visit | SCREEN |
| Patient No. Visit | |
| / Planned<br>Dose | 250 mg QD<br>PLX9486 |
| Study<br>Part | Н |

Note: L=Low and H=High with respect to laboratory reference ranges, where applicable. CTCAE v4.03 grades are in parentheses where applicable. \* indicates abnormal, clinically significant, as reported by the investigator. CTCAE grading is performed using data values only and does not consider symptomatic criteria.

[1] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and Adverse Events.

EOS = End of study; UNS = Unscheduled; CTCAE = Common Terminology Criteria for Adverse Events.

time date 

Programmer notes:

1) Sort by Visit within each patient.

| ethods | |
|------------------|---------|
| ıl Me | |
| on of Statistica | |
| umentati | |
| 1.9 Doc | 7870X I |
| 16. | 10 |

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01


Plexxikon Inc. Protocol PLX121-01

Listing 16.2.6.4.2 Coagulation – Other Tests

| Reference Reference Range Clinically Range Low High Significant? | Yes/No | Yes/No |
|---|---|---|
| Was patient Reference Reference Range fasting? Other Tests Result Unit Range Low High | XX.X | XX.X |
| Reference<br>Range Low | XX.X | XX.X |
| Unit | XXXXX | XXXXX |
| Result | X.X.X | XX.X |
| Other Tests | XXXXX | XXXXX |
| Was patient fasting? | Yes/No/Unknown xxxxx | |
| Collection<br>Date / Time | DDMMMYYYY/ | IIII:MIM |
| Visit | SCREEN | |
| lanned Patient<br>Dose No. Visit | | |
| Study Planned Patient Part Dose No. | 250 mg QD | FLA9400 |
| Study<br>Part | П | |

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled.

time date 

- Programmer notes:

  1) Sort by visit, time point and analyte (test name alphabetically) within each patient.
  2) For column 'Result', display the result and number of decimal places as in raw data

16.1.9 Documentation of Statistical Methods PLX9486

| Plexxikon Inc.<br>PLX121-01 | Statistical Analysis Plan 01Jul202 <u>0</u> |
|---|---|
| Plexxikon Inc.<br>Protocol PLX121-01 | Page 1 of x |
| | Listing 16.2.7.1 |
| | Vital Signs<br>Part 1 of 2 |

Clinical Study Report PLX121-01

| | | | | | | | | Weight<br>(kg) | | Temperature (°C) | ture | Hea<br>(b | Heart Kate<br>(bpm) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study<br>Part | Planned Dose Patient No. Visit | Patient No. | Visit | Time Point | Vitals Collected? | Measurements Date / Vitals Collected? Measurements Time Result | ate/<br>ime Resu | Change from | | Cha<br>Result B | Change from<br>Baseline | Result | Change from<br>Baseline |
| | 250 mg QD | | SCREEN | | Yes/No | | 09 | | 37 | 9'. | | 09 | |
| | | | CIDI | Pre-Dose | Yes/No | | 61* | | 36. | 36.6* | | 62* | |
| | | | | | | | 62 | 1 | 36 | 4.0 | -0.2 | 70 | ~ |
| | | | | | | | | | | | | 81 | |
| | | : | | | | | | | | | | | |
| | | | | | | Part 2 of 2 | | | | | | | |
| 1 | | | | | | Res | Respiration | | SBP | | DBP | | |
| | | | | | | (brea | (breaths/min) | (L | (mmHg) | | (mmHg) | | |
| | | | | | Measurements | ments | | | | | | | |
| | | | | | Date / | / 6 | | | Change | a) | | | |
| | | | | | Measurements | ments | Change from | m | from | | Cha | Change from Position of | Position of |
| | Part Planned Dose Patient No. Visit | tient No. Visit | | Time Point Vitals Collected? | lected? Time | le Result | Baseline | Result | Baseline | | Result Ba | Baseline | Patient |
| 1 | | | | | | | | | | | | | |

Note: \* Baseline value. ^ indicates decrease from baseline in SBP greater than 20, # indicates decrease from baseline in DBP greater than 10.

[1] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers DBP = Diastolic Blood Pressure; EOS = End of study; SBP = Systolic Blood Pressure; UNS = Unscheduled.

Standing Supine

-15#

-22^

9

15 16\* 22

Yes/No Yes/No

Pre-Dose

SCREEN C1D1

250 mg QD

137H 132H\* 110

83 82\* 67

Prone

Sitting

date Programmer notes:

time

1) Combine data from VS (Vital Signs) & VSI (Pre and Post Dose Vital Signs) 2) Use ADVS.AVAL to get standardized results


| al Methods | |
|---------------|---------|
| of Statistic | |
| sumentation o | |
| 16.1.9 Doc | PLX9486 |

Statistical Analysis Plan 01Jul2020 Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Clinical Study Report PLX121-01

Listing 16.2.7.2 Physical Examination

| Ξ | | |
|---|---|---|
| Any Abnormal Findings? | Yes/No | |
| Examination Date | | |
| Study Part Planned Dose Patient No. Visit Examination Performed? Examination Date Any Abnormal Findings? | Yes/No | |
| Visit | SCREEN | C1D1 |
| Patient No. | | |
| Planned Dose | 250 mg QD<br>PLX9486 | |
| Study<br>Part | - | |

<sup>&</sup>lt;sup>[1]</sup> Abnormal findings prior to treatment are documented in medical history; abnormal findings post treatments are documented as adverse events.

<sup>[2]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled.

date 

time

16.1.9 Documentation of Statistical Methods

PLX9486

Statistical Analysis Plan

Clinical Study Report PLX121-01

01Jul2020


Plexxikon Inc. Protocol PLX121-01

Plexxikon Inc. PLX121-01

12-Lead Electrocardiogram Listing 16.2.7.3.1

| ECG Interpre- HR RR <sup>[2]</sup> PR QRS QT QTcF <sup>[2]</sup> Of | | | Chang |
|---|---|---|---|
| 1 Normal xx xx xx xx xx xx xx 1 4 * xx | Study Planned Patient Performe Date/ Part Dose No. Visit Time Point d? Time | QRS QT nsec) (msec) | Baseli<br>QTcF <sup>[2]</sup> of<br>(msec) QTcF |
| 1 Normal xx xx xx xx xx xx xx | , c | | |
| XX XX XX XX | 10-Day Run-in xxxxx Yes/No | | XX |
| | No | | XX |
| 1 & 4 - 5 & 4 - 5 & 4 - 5 & 6 | SCREEN | | |
| 4 * | | | |
| 3.4.*<br>1.2.2.2.2.2.2.2.2.2.2.2.2.2.2.2.2.2.2.2 | C1D1 Pre-Dose* | | |
| 2 | | | |
| 1.4 m | 1 Hour Post-Dose | | |

Note: \* Baseline value; 4\* = Average of triplicate. L=Low and H=High with respect to reference ranges for PR and QRS.

Note: The baseline value is defined as the last non-missing value of the average of the triplicate ECGs prior to the patient's first dose of study drug.

If If interpretation was abnormal, was the ECG clinically significant?

time date 

## Programmer notes:

1) Combine records from all raw ECG datasets: EG, EGI, EG2, EG3, EG4, EG5, EG7. Display RR, QTcB and QTcF from ADEG.


<sup>[2]</sup> RR and QTcF are derived.

<sup>&</sup>lt;sup>[3]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers CS = [Abnormal] Clinically Significant; BOS = End of study; NCS = [Abnormal] Not Clinically Significant; ND = Not Done; UNS = Unscheduled. [3] Patient numbers

16.1.9 Documentation of Statistical Methods

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020 Clinical Study Report PLX121-01

Plexxikon Inc. Protocol PLX121-01


| om Baseline [1] | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | |
|---|---|---|---|---|
| tual Result <sup>[1]</sup> Change Fr | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X | |
| Baseline Result A | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X | |
| Parameter (msec) | QТсF<br>xxxx | XXXX | XXXX | |
| ECG Time | time5.<br>time5. | time5.<br>time5. | time5.<br>time5. | |
| ECG Date | date9.<br>date9. | date9.<br>date9. | date9. | |
| Visit | Visit 1<br>Visit 2 | Visit 1<br>Visit 2 | Visit 1 | |
| Gender | | | | |
| Patient No. | XXXXXX | XXXXXX | XXXXXX | |
| Planned Dose | 250 mg QD | | XXXXX | |
| Study Part | - | | P1-C2 | |
| | ECG Date | Visit 1 date9. time5. | VisitECG DateECG TimeVisit 1date9.time5.Visit 2date9.time5.Visit 1date9.time5.Visit 2date9.time5. | Part Planned Dose Patient No. Gender Visit ECG Date ECG Time 250 mg QD xxxxxx Visit 1 date9. time5. xxxxxx Visit 2 date9. time5. visit 2 date9. time5. visit 2 date9. time5. xxxxxx Xxxx Xxxxx Visit 1 date9. time5. |

Note: The baseline value is defined as the last non-missing value of the average of the triplicate ECGs prior to the patient's first dose of study drug.

QTcF (Fridericia's method) are derived.

[1] Post-baseline outlier values considered in this listing are as follows: (1) QTcF  $\geq$  450 msec (for males) or  $\geq$  470 msec (for females), or (2) increase from baseline in QTcF > 30 msec. Findings which completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers meet any of these outlier criteria are asterisked. [2] Patient numbers

time 

date

## Programmer Note:

1) Use derived RR, QTcB, QTcF (ADEG.PARAMCD=RRINT, DQTCF, DQTCB)

Plexxikon Inc.

PLX121-01

Plexxikon Inc. Protocol PLX121-01


Statistical Analysis Plan 01Jul2020

## **ECOG Performance Status Assessment Listing 16.2.7.4**

| ECOG[1] | | 0/1/2/3/4/5 | | | | |
|---|---|---|---|---|---|---|
| Assessment Date | | DDMMMYYYY | | | | |
| No. Visit ECOG Performed? | | Yes/No | | | | |
| Visit | C1D1 | | CID8 | C1D15 | C2D1 | <br>TERM |
| Patient No. | | | | | | |
| Planned Dose | 250 mg QD | PLX9486 | | | | |
| Study Part | | _ | | | | |

ECOG: 0 = Fully active, able to carry on all pre-disease performance without restriction, 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours, 3 = Capable of only limited self care, confined to bed or chair more than 50% of waking hours, 4 = Completely disabled. Cannot carry on any self care. Totally confined to bed or chair, 5 = Dead.

[2] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers completed their initial Cohort and subsequently re-enrolled. Eastern Cooperative Oncology Group; EOS = End of study; UNS = Unscheduled.

time date 

Programmer Note:

1) Get ECOG data from releavant parts in CRF form 'Physical Examination' (raw dataset PE)


| Methods | |
|--------------------|-------|
| Statistical N | |
| on of S | |
| Documentation of 3 | |
| 6 | 7 |
| = | ì |
| 6. | 01011 |

Plexxikon Inc. PLX121-01 PLX9486

Plexxikon Inc. Protocol PLX121-01

## Listing 16.2.7.5 Echocardiogram/MUGA Scan

Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01


| -Ser | Patient No. Visit Performed? Assessment Date Assessment Time % LVEF No CIDI 10:15 No | | Associated Primary Description of Interpretation AE <sup>[1]</sup> Abnormality | rmal/Abnormal, |
|---|---|---|---|---|
| Performed? Assessment Date Assessment Time 10:15 | Patient No. Visit Performed? Assessment Date Assessment Time C1D1 10:15 | ose Patient No. Visit | % LVEF | N |
| Performed? Assessment Date | Patient No. Visit Performed? Assessment Date C1D1 | ose Patient No. Visit | Assessment Time | 10:15 |
| Performed? | Patient No. Visit Performed? CID1 | ose Patient No. Visit | Assessment Date | |
| | Patient No. Visit | Part Planned Dose Patient No. Visit 250 mg QD CID1 | Performed? | |

time date 

<sup>[1]</sup> Only recorded if the interpretation is 'Abnormal, CS'.

[2] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers MUGA = Multigatd aequisition; CS = Clinically Significant; NCS = Not Clinically Significant; UNS = Unscheduled.

| of Statistical Methods | |
|-------------------------|----------|
| 16.1.9 Documentation of | 9010V Id |

Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Listing 16.2.7.6 Thyroid Stimulating Hormone (TSH) Level

| Study Par | Study Part Planned Dose Patient No. Visit | Patient No. | Visit | Sample<br>Collected? | Collection Date | Collection Time | TSH Level |
|---|---|---|---|---|---|---|---|
| П | 250 mg QD<br>PLX9486 | XX-XX | C1D1 | Yes/No | DDMMMYYYY | 10:15 | |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers UNS = Unscheduled.

time

| 9 Documentation of Statistical Methods | )486 |
|----------------------------------------|------|
| 16.1. | PLX9 |

| Plexxikon Inc.<br>PLX121-01 | Statistical Analysis Plan<br>01Jul2020 |
|---|---|
| Plexxikon Inc.<br>Protocol PLX121-01 | Page 1 of x |
| Listing 16.2.7.7 Pregnancy Test | |

Clinical Study Report PLX121-01

| | Result | Negative<br>Positive |
|---|---|---|
| | Collection Date | |
| | Test Type | Urine Dipstick<br>Serum |
| If No, Specify | Reason | |
| | Test performed? | Yes/No<br>Yes/No |
| | Visit | SCREEN<br>EOS |
| | Patient No. | I |
| | Study Part Planned Dose Patient No. | 250 mg QD<br>PLX9486 |
| | Study Part | 1 |

<sup>[1]</sup> Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; UNS = Unscheduled.

time

| thods | |
|------------------|-------|
| ical Me | |
| f Statisti | |
| ion of | |
| Documentation or | |
| 9 Docui | X9486 |
| 16.1.9 I | PLX |

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020 Clinical Study Report PLX121-01

Listing 16.2.7.8.1 Circulating DNA Plexxikon Inc. Protocol PLX121-01


| 1 | Time | HH:MM |
|---------------------|--------------|-------------------|
| Assessment | Date | DDMMMYYYY |
| Assessment Obtained | Pre-dose? | Yes/No |
| | Visit | CIDI |
| | Patient No. | I |
| | Planned Dose | 250 mg QD PLX9486 |
| | Study Part | - |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers EOS = End of study; UNS = Unscheduled.

time date 

Programmer notes:
1) Sort by Visit within each patient.


16.1.9 Documentation of Statistical Methods

PLX9486

Clinical Study Report PLX121-01

Plexxikon Inc. PLX121-01

Statistical Analysis Plan 01Jul2020


Plexxikon Inc. Protocol PLX121-01

Listing 16.2.7.8.2 Tumor Markers

| | | | | Sample | Collection | uc | | |
|---|---|---|---|---|---|---|---|---|
| Part | Planned Dose | Patient No. Visit | Visit | Collected? | Date | Time | Test Type | Result (Unit) |
| • • | 250 mg QD PLX9486 | I | CIDI | Yes/No/NA | DDMMMYYYY | нн:мм | Carcinoembryonic Antigen-CEA (Colorectal) CA-125 (Ovarian) Calcitonin (Medullary Thyroid) CA19-9 (Pancreatic) Prostate-Specific Antigen-PSA (Prostate) Other, specify: | 0.5 (ng/mL) |

[1] Patient numbers completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers EOS = End of study; NA = Not Applicable; UNS = Unscheduled.

date 

time

Programmer notes:
1) Sort by Visit within each patient.


| istical Methods | |
|------------------------|---------|
| cumentation of Statist | |
| 16.1.9 Docum | PLX9486 |

Plexxikon Inc. PLX121-01

Plexxikon Inc. Protocol PLX121-01


Statistical Analysis Plan 01Jul2020

Clinical Study Report PLX121-01

Listing 16.2.7.8.3
Archival Tumor Tissue Collection

# Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486)

| | Date Sample Shipped | DDMMMYYYY |
|---------------------|---------------------|----------------------|
| Tracking Number for | Specimen | xxxxxxxx |
| | Anatomical Site | COLON |
| Collection | Time | HH:MM |
| | Collection Date | DDMMMYYYY |
| | Sample Obtained? | Yes/No |
| | Visit | SCREEN |
| | Patient No. | I |
| Study | Planned Dose | 250 mg QD<br>PLX9486 |
| Study | Part | 1 |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers

time

date 

- Programmer notes:

  1) Sort by Visit within each patient.
  2) If tissue specimen collection date is unknown, then put 'Unknown' into collection date column.


Plexxikon Inc.


16.1.9 Documentation of Statistical Methods PLX9486

| Statistical Analysis Plan | 01Jul202 <u>0</u> |
|---------------------------|-------------------|
| Plexxikon Inc. | PLX121-01 |

Clinical Study Report PLX121-01

 Listing 16.2.7.8.4 Optional Paired Tumor Biopsy Plexxikon Inc. Protocol PLX121-01

Study Part 1 - Dose Escalation Study Parts (Single-Agent PLX9486)

| Tracking Number for<br>Specimen | | | |
|---|---|---|---|
| Shipping Date | | | |
| Anatomical Site | | | |
| Type | Core | | |
| Collection<br>Date | I | I | I |
| Sample<br>Collected? | Yes | Yes | Yes |
| | CIDI | CID15 | C2D1 |
| Study Part Planned Dose Patient No. Visit | 1 250 mg QD xx-xxx | | |

completed their initial Cohort and subsequently re-enrolled, respectively, as patient numbers [1] Patient numbers

time

date

Programmer notes:

1) Sort by Visit within each patient.





